

#### 1. RCT Details

This section provides a high-level overview of the RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes (EMPA-REG\_OUTCOME trial)

#### 1.2 Intended aim(s)

To determine the long-term cardiovascular (CV) safety of empagliflozin, as well as investigating potential benefits on macro/microvascular outcomes.

### 1.3 Primary endpoint for replication and RCT finding

Major Adverse Cardiovascular Events, Including CV Death, Nonfatal Myocardial Infarction (MI), and Nonfatal Stroke

### 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

For the test of noninferiority for the primary outcome with a margin of 1.3 at a one-sided level of 0.0249, at least 691 events were required to provide a power of at least 90% on the assumption of a true hazard ratio of 1.0.

### 1.5 Primary trial estimate targeted for replication

HR = 0.86 (95% CI 0.74-0.99) comparing empagliflozin to placebo (Zinman et al., 2015)

#### 2. Person responsible for implementation of replication in Aetion

Ajinkya Pawar, Ph.D. implemented the study design in the Aetion Evidence Platform. S/he is not responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform.

### 3. Data Source(s)

United/Optum, MarketScan, Medicare

#### 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

## Design Diagram - EMPA-REG TRIAL REPLICATION



#### 5. Cohort Identification

#### 5.1 Cohort Summary

This study will involve a new user, parallel group, cohort study design comparing empagliflozin to the DPP-4 inhibitor (DPP4i) antidiabetic class. DPP4is serve as a proxy for placebo, since this class of antidiabetic drugs is not known to have an impact on the outcome of interest. The comparison against DPP4 inhibitors is the **primary comparison**. The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of empagliflozin or a comparator drug (cohort entry date). Follow-up for the outcome (3P-MACE), begins the day after drug initiation. As in the trial, patients are allowed to take other antidiabetic medications during the study.

### 5.2 Important steps for cohort formation

#### 5.2.1 Eligible cohort entry dates

Market availability of empagliflozin in the U.S. started on August 1, 2014.

- For Marketscan and Medicare: Aug 1, 2014-Dec 31, 2017 (end of data availability).
- For Optum: Aug 1, 2014-Mar 31, 2019 (end of data availability).

### 5.2.2 Specify inclusion/exclusion criteria for cohort entry and define the index date

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

### 5.3 Flowchart of the study cohort assembly

| | Optum | | Marketscan | | Medicare* | |
|---|---|---|---|---|---|---|
| | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients |
| All patients | | 74,864,884 | | 191,990,035 | | 23,466,175 |

| Patients who used exposure or a reference between Aug 1, 2014 to Dec 2017 (for Marketscan/Medicare)/March 2019 (for Optum) | -74,294,229 | 570,655 | -191,387,941 | 602,094 | -22,015,231 | 1,450,944 |
|---|---|---|---|---|---|---|
| Patients who have continuous 6 months registration in the database | -77,109 | 493,546 | -41,856 | 560,238 | -387,934 | 1,063,010 |
| Excluded due to prior use of referent | -281,236 | 212,310 | -365,720 | 194,518 | -738,467 | 324,543 |
| Excluded due to prior use of exposure | -45,709 | 166,601 | -35,973 | 158,545 | -25,468 | 299,075 |
| Excluded because patient qualified in >1 exposure category | -716 | 165,885 | -1,192 | 157,353 | -546 | 298,529 |
| Excluded based on missing Age | -6 | 165,879 | 0 | 157,353 | 0 | 298,529 |
| Excluded based on missing Gender | -8 | 165,871 | 0 | 157,353 | 0 | 298,529 |
| Excluded based on Inclusion 1- Age >=18 | -5 | 165,866 | -44 | 157,309 | 0 | 298,529 |
| Excluded based on Inclusion 2- DM Type 2 with ICD-10 codes | -4,270 | 161,596 | -6,031 | 151,278 | -3,158 | 295,371 |
| Excluded based on Inclusion 5- High risk of cardiovascular events | -13,525 | 148,071 | -15,359 | 135,919 | -12,190 | 283,181 |
| Excluded based on Inclusion 6- BMI ≤45 kg/m2 (excluded morbid obese patients) | -4,602 | 143,469 | -3,000 | 132,919 | -6,924 | 276,257 |
| Excluded based on Exclusion 2- Liver disease with ICD-10 and Exclusion 5-<br>Bariatric surgery within the past two years and other gastrointestinal<br>surgeries that induce chronic malabsorption | -458 | 143,011 | -2,049 | 130,870 | -7,325 | 268,932 |
| Excluded based on Exclusion 6- Blood dyscrasias or any disorders causing hemolysis or unstable red blood cells | -9,118 | 133,893 | -5,029 | 125,841 | -29,542 | 239,390 |
| Excluded based on Exclusion 7- History of Malignant Neoplasm past 5 years | -3,550 | 130,343 | -2,870 | 122,971 | -11,850 | 227,540 |
| Excluded based on Exclusion 9- Obesity claim or drug 3 months prior | -466 | 129,877 | -2,810 | 120,161 | -4,053 | 223,487 |
| Excluded based on Exclusion 10- Use of corticosteroids | -1504 | 128,373 | -1147 | 119,014 | -2,798 | 220,689 |
| Excluded based on Exclusion 12- Pregnancy OR Contraceptive | -398 | 127,975 | -627 | 118,387 | -425 | 220,264 |
| Excluded based on Exclusion 13- Alcohol or drug abuse | -67 | 127,908 | -258 | 118,129 | -568 | 219,696 |
| Excluded based on Exclusion 16- Acute coronary syndrome, stroke, or transient ischemic attack within 2 months | -390 | 127,518 | -677 | 117,452 | -2,625 | 217,071 |
| Final cohort | | 127,518 | | 117,452 | | 217,071 |

<sup>\*</sup> Medicare database includes only patients with at least one diagnosis for diabetes, heart failure, or cerebrovascular disease.

<sup>\*\*</sup>Exclusion 2 and 5 collapsed to adhere to CMS cell suppression guidelines.

Effectiveness research with Real World Data to support FDA's regulatory decision making

#### 6. Variables

#### 6.1 Exposure-related variables:

### Study drug:

The study exposure of interest is initiation of empagliflozin. Initiation will be defined by no use of empagliflozin or a comparator in the prior 6 months before treatment initiation (washout period).

#### Comparator agents-

- · Initiators of empagliflozin will be compared to initiators of
  - o DPP4i

Because empagliflozin and comparators are frequently used as second or third line treatments of T2DM, we expect it to be unlikely that empagliflozin and comparators are initiated in patients with substantially different baseline risk for proposed outcomes.

#### 6.2 Covariates:

- Age
- Sex
- Combined Comorbidity Index (CCI), measured over the baseline covariate assessment period, defined as 180 days prior to and including index date

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (Appendix B). These covariates are based on those used by Patorno et al. (2019).

## 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcomes of interest (definitions provided in Appendix A):

- <u>Primary outcome</u>: 3-point major adverse cardiovascular events (MACE), i.e., non-fatal myocardial infarction, non-fatal stroke, or CV mortality
- · Secondary outcomes: Individual components:
  - Hospital admission for MI (for purposes of this individual component, fatal MI is included)
  - Hospital admission for stroke (for purposes of this individual component, fatal stroke is included)
  - All-cause mortality/CV mortality:
    - All-cause inpatient mortality identified using discharge status codes will be used as a proxy for "CV mortality" in commercial databases

Information on CV mortality through data linkage with the National Death Index (NDI) will only become available at a later date for Medicare and will be used in secondary analyses.

Control outcomes of interest (control outcomes only serve to assess aspects of study validity but are not further interpreted):

- 1. Diabetes Ketoacidosis (we expect to see a positive association; Neal et al., 2017)
- 2. Heart failure (we expect to see a protective effect; Neal et al., 2017)

#### Control outcome definitions

| Outcome | Definition | Comments |
|---|---|---|
| Control Outcomes | | |
| Diabetic Ketoacidosis | Inpatient ICD-9 diagnosis: 250.1x | Note- The corresponding ICD-10 codes will also be used |
| Heart Failure | Inpatient ICD-9 diagnosis (primary diagnosis): 428.x, 398.91, 402.01, 402.11, 402.91, 404.01, 404.11, 404.91, 404.03, 404.13, 404.93 | Note- The corresponding ICD-10 codes will also be used |

#### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real world databases is expected to be much worse than in the trial, the AT analysis is the **primary** analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analyses, the follow-up will start the day after initiation of empagliflozin and comparator and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (empagliflozin and comparator) plus a defined grace period (i.e., 30 days after the end of the last prescription's days' supply in main analyses).
- The date of augmentation or switching from an exposure to a comparator or any other agent in the comparator class and vice versa (e.g. switching from saxagliptin to linagliptin would be a censoring event);
  - o A dosage change on the index treatment does not fulfill this criterion
  - An added treatment that is not part of the exposure or comparator group does not fulfill this criterion (e.g. if a empagliflozin user adds insulin, he or she does not get censored at the time of insulin augmentation)

For the ITT analyses, the censoring based on the augmentation/switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

### 7. Initial Feasibility Analysis

### Aetion report name:

For empagliflozin vs. DPP4i

Optum-https://bwh-dope.aetion.com/projects/details/654/results/43641/result/0

Marketscan- https://bwh-dope.aetion.com/projects/details/655/results/43642/result/0

Medicare- https://bwh-dope.aetion.com/projects/details/653/results/43643/result/0

Date conducted: 10/29/2019

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

- Report patient characteristics by treatment group
- Report summary parameters of the overall study population
- · Report median follow-up time by treatment group
- · Report reasons for censoring in the overall study population

#### 8. Initial Power Assessment

#### Aetion report name:

For empagliflozin vs. DPP4i

Optum- https://bwh-dope.aetion.com/projects/details/654/results/43644/result/0

Marketscan- <a href="https://bwh-dope.aetion.com/projects/details/655/results/43645/result/0">https://bwh-dope.aetion.com/projects/details/655/results/43645/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/projects/details/653/results/43646/result/0">https://bwh-dope.aetion.com/projects/details/655/results/43645/result/0</a>

#### Date conducted: 10/29/2019

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 11/4/2019 |
|-------------------------|------------------|----------------|-----------|
| Reviewed by FDA: | | Date reviewed: | |
| Reasons for stopping | | | |
| analysis (if required): | | | |

### 9. Balance Assessment after PS matching

#### Aetion report name:

Optum- https://bwh-dope.aetion.com/projects/details/654/results/45417/result/0

Marketscan- https://bwh-dope.aetion.com/projects/details/655/results/45418/result/0

Medicare- https://bwh-dope.aetion.com/projects/details/653/results/45419/result/0

Date conducted: 11/30/2019

After review of initial feasibility and power analyses, complete creation of the remaining covariates (see Table 1 below for list of covariates). Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates (excluding laboratory values, which are missing in some patients).

· Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

Report covariate balance after matching.

Note- For Table 1, please refer to Appendix B.

· Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy Outcome | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
| Death | 228 (0.22%) | 142 (0.27%) | 86 (0.17%) |
| Start of an additional exposure | 3,474 (3.35%) | 1,357 (2.62%) | 2,117 (4.08%) |
| End of index exposure | 50,368 (48.55%) | 26,107 (50.33%) | 24,261 (46.77%) |
| Specified date reached (Dec 16/Sep 17) | 35,687 (34.40%) | 17,006 (32.78%) | 18,681 (36.01%) |
| End of patient enrollment | 11,469 (11.05%) | 5,415 (10.44%) | 6,054 (11.67%) |
| Switch to other DPP4i (for censoring) + nursing home admission | 2,526 (2.43%) | 1,849 (3.56%) | 677 (1.31%) |

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

· Report follow-up time by treatment group.

| | Median Follow-Up Time (Days) [IQR] | | |
|---|---|---|---|
| Patient Group | Optum | Marketscan | Medicare |
| Overall Patient Population | 118 [58-243] | 118 [58-268] | 118 [58-215] |
| Referent | 118 [58-228] | 118 [58-218] | 118 [58-218] |
| Exposure | 118 [58-262] | 118 [58-211] | 118 [58-211] |

Report overall risk of the primary outcome.

| | Optum | Marketscan | Medicare |
|-------------------------|-------|------------|----------|
| Risk per 1,000 patients | 12.51 | 7.31 | 23.78 |

#### 10. Final Power Assessment

Date conducted: 12/1/2019

- Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9.
   All other parameters in the table should be the same as in Section 8. If the study is to be implemented in more than one database, copy and paste excel sheet to report power for each database separately and for the pooled analysis that uses data from all databases together. Power calculations are based on the formulas from Chow et al. (2008).
  - o Pooled

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 51,876 | Reference | 51,876 |
| Exposed | 51,876 | Exposed | 51,876 |
| Risk per 1,000 patients | 14.53 | Risk per 1,000 patients | 14.53 |
| Desired HR from RCT | 0.86 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 1507.51656 | Number of events expected | 1507.51656 |
| Power | 0.833482663 | Power | 0.999136066 |

## o Optum

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 23,348 | Reference | 23,348 |
| Exposed | 23,348 | Exposed | 23,348 |
| Risk per 1,000 patients | 12.51 | Risk per 1,000 patients | 12.51 |
| Desired HR from RCT | 0.86 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 584.16696 | Number of events expected | 584.16696 |
| Power | 0.445473008 | Power | 0.886984947 |

## o Marketscan

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 16,256 | Reference | 16,256 |
| Exposed | 16,256 | Exposed | 16,256 |
| Risk per 1,000 patients | 7.31 | Risk per 1,000 patients | 7.31 |
| Desired HR from RCT | 0.86 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 237.66272 | Number of events expected | 237.66272 |
| Power | 0.213506619 | Power | 0.524870241 |

## o Medicare

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 12,272 | Reference | 12,272 |
| Exposed | 12,272 | Exposed | 12,272 |
| Risk per 1,000 patients | 23.78 | Risk per 1,000 patients | 23.78 |
| Desired HR from RCT | 0.86 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 583.65632 | Number of events expected | 583.65632 |
| Power | 0.44515838 | Power | 0.886719001 |

Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of
advisory board. Reviewers evaluate the results of the analyses described above in Sections 9 and 10, including numbers of
patients, balance in patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates
of outcomes and study power.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 12/5/19 |
|-------------------------|------------------|----------------|------------|
| Reviewed by FDA: | David Martin | Date reviewed: | 12/20/2019 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

### 11. Study Confidence and Concerns

Deadline for voting on study confidence and listing concerns: 12/20/19

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the
  success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may
  contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study
  variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the
  individual respondent.

### 12. Register study protocol on clinicalTrials.gov

### Date conducted:

Register the study on <u>clinicalTrials.gov</u> and upload this document.

### 13. Comparative Analyses

Aetion report name:

Date conducted:

#### 13.1 For primary analysis:

 In the PS-matched cohort from Section 9, calculate the HR for each outcome for empagliflozin versus referent patients using a Cox proportional hazards model.

### 13.2 For secondary analyses:

• In the pre-matched cohort, perform asymmetrical trimming to remove patients with PS values below the 2.5<sup>th</sup> percentile of treated patients and above the 97.5<sup>th</sup> percentile of untreated patients. In the trimmed cohort, calculate the HR for empagliflozin versus referent patients using a Cox proportional hazards model, adjusting for deciles of the PS.

### 14. Requested Results

#### 14.1 Results from primary and secondary analyses:

Separately for each endpoint:

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Primary analysis | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

#### 15. References

American Diabetes Association. 8. Pharmacologic Approaches to Glycemic Treatment: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018;41(Suppl 1):S73-S85. doi:10.2337/dc18-S008.

Effectiveness research with Real World Data to support FDA's regulatory decision making

Chow S, Shao J, Wang H. 2008. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177

Patorno E, Pawar A, Franklin JM, et al. Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study. Circulation. 2019;139:2822-30.

Zinman B, Wanner C, Lachin JM, et al. Empagliflozin, cardiovascular outcomes, and mortality in type 2 diabetes. New England Journal of Medicine. 2015;373(22):2117-28.

| # | | Empa-Reg trial definitions | Implementation in routine care | References/Rationale | Color coding |
|---|---|---|---|---|---|
| | | Trial details- Secondary Indication; 4s- Unit | tended 5 with label change | Please see the following-Google Drive for further details or any relating informations:<br>https://drive.annels.com/sees/7d=1W0618 www/filetch/cold/Vcnblobe/V | Citaria |
| | | EXPOSURE vs. COMP | arison | ED-10 codes are not listed in this document because of eacel call dis limitations and exceedes number of<br>ED-10 codes. Full ICD-10 code lists will be excluded in the above Google Order Folder (fish above), ED-10 codes. Full ICD-10 code conservious were completed using a SAS reacre that implements forward/ backward reapplay based on the CMS ICD-10 reapplay; three If however the constitution for each consensation.<br>Amount and above constitution from | Adequatemapping in claims |
| | _ | empagiffosin 10 mg, empagiffosin 25 mg, or placebo | Empaglificoln vs. Individual non-glificath antidiabetic class (is, a DPP-41, a GLP-31A, and a sulfomplures) | Patonno, Blabbetta et al. "Cardiovascular outcomes associated with canaglificatin versus other non-glificatin<br>varidiabettic druger population based cohort study." BMI 2018;360:k119<br>http://dx.doi.org/10.1136/pmi.k119 | intermediate mapping in claims |
| Н | 4 | PRIMARY OUTCO | ME | | Poor mapping or cannot be measured in claims |
| | | | Measured 1 days after drug tritisation in diagnosis position specified below and investent care setting inpatient nortality/MaySevals — For Mil Any diagnosis position in inpatient care setting KD-9 diagnosis position in inpatient care setting KD-9 diagnosis (0.0.1) journe myocardial inferction) excluding 410.12 (subsequent splands of care) For stools. Primary diagnosis position in inpatient care setting KD-9 discharge diagnosis. KD-9 dischar | For Mill: | Can't be measured in claims but not important for the analysis |
| Н | - | INCLUSION CRITE | RIA | | |
| 1 | | Ageistifi years (For Japan: Ageistif) years); (For India: Ageistifi years and 665 years) | Age it it 8 years at drug initiation | | |
| 2 | 1 | | Measured 180 days prior to drug initiation in any diagnosis position and the inpatient or outgatient care setting<br>Tree 2 Disbetts (CD-9 diagnosis 250.x0, 250.x2 | Patorno, Blashetta et al. "Cardiovacular outcomes associated with caragificion versus other non-gifficoin articlabetic drugs population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Blashetta et al. "Engagificion and the Risk of Heart Fallure Hospitalization in Boutine Clinical Care: A First Avalytic from the Engagificion Comparative Effectiveness and Safety (BMPRES) Study." Circulation. 2018 Agrid. doi: 10.1161/CRECUATIONMA.118.01916. | |
| , | - | On a diet and exercise netimen | N/A | | |
| 4. | 1 | roufficient decemic control, defined as either: - Drug-nalve(no arti-diabetes agents for >=6.2 weeks prior to randomization) + HbA5c a7.0% (653 mmol/mol) and 48.0% (475 mmol/mol) at creating | (Covered below in 4b) | Patomo, Blashetta et al. "Cardiovaccular outcomes associated with canaglificoln versus other non-glifficoln<br>antidiabetic drugs: population hased cohort study." BMJ 2018;360:k119<br>http://dx.doi.org/10.1186/brigis119<br>Patomo, Blashetta et al. "Ringagifficoln and the Not of Heart Fallure Hospitalization in Routine Clinical Care:<br>A Rint Analysis than the Empagifficoln Comparative (Shoctiveness and Safety (SMPRSS) Study." Circulation.<br>2018 April. doi: 10.1161/SIDEUINDEMPALIA 10.0161 | |
| | 1 | • Taking any background anti-diabetes therapy (except pinglitzzone in Japan) + HbA1c 27.0% (x53 mmol/mol) and x50.0% (x66 mmol/mol) at screening | During the cohort creation, depending on the comparison group, we will require new-use/defined as no use 180 days<br>prior to index date) of empagificoin and a comparator drug | | |
| ľ | | -Background wit-dishers therapy had to be unchanged for it? I weeks prior to prodomization -If background with dishers therapy included insulin, insulin dose had to be unchanged by >10% from the dose at randomization in the previous 12 weeks. | | | |
| 5 | | iligh risk of cardiovascular events, defined by ≫i of the following: | Measured 61 days prior to drug initiation to 3650 days prior to drug hilldation in any diagnosis position and the impatient or outputient care setting Colde system ICD-9 diagnosis: 413.xx OR Measured 365 days prior to drug initiation as a dispensing of one of the following medications ACE inhibitor Bensseyst, cartopril, wralapril, flosinopril, Binopril, monetyril, perindopril, quimapril, ramigril, translolapril ACB | | |

| Sa | ■ History of myocardial infarction >2 months prior to informed consent — History of myocardial infarction >2 months prior to informed consent. | Measured 61 days prior to drug initiation to 3650 days prior to drug initiation in any diagnosis position and the Inquitient or outpatient care setting - <u>Acute M</u> KD-9 diagnosis: 610.m., <u>Old M</u> KD-9 diagnosis: 612.m. | Patono, Blashetts et al. "Cardiovaccular outcomes associated with caragificatin versus other non-gliffocis and disbatic druger population based cohort mody." BMJ 2018;360:h119 http://dx.doi.org/10.118/phnj.h119 Patono, Blashetts et al. "Empagificatin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Avaignit from the Empagificatin Comparative Effectiveness and Safety (BMP985I) Study." Circulation. 2019 April. 40: 10.1161/CIRCULANDWANL 18.0.0316. |
|---|---|---|---|
| $\vdash$ | + Evidence of multi-vessel CAD La. In a 2 major coronary arteries or the left main coronary artery, documented by any of the following: | | |
| | -Presence of significant stenosis: 250% luminal narrowing during angiography (soronary or multi-dice computed tomography) | Measured 1 days prior to drug initiation to 3650 days prior to drug initiation in any diagnosis position and the inputient<br>or outpatient care setting<br>Coronary atheroadeosis and other forms of chronic ischemic heart disease | |
| 1 | - Previous revascularization (percutaneous transluminal coronary angioplasty estent or coronary artery bypass graft >2 months prior to consent | Coronary respects a restriction: | |
| | | Measured 61 days prior to drug initiation to 3650 days prior to drug initiation in any procedure position and inpatient<br>care setting—CPT-4: 33510—33536, 33546, 33573. CRI. Measured 61 days prior to drug initiation to 3650 days prior to drug initiation in any procedure position and inpatient or outpellent care setting—CPD procedure 36.1s, 36.2x | |
| | | PTG: Measured 61 days prior to drug initiation to 3650 days prior to drug initiation in any procedure position and inpatient care setting - CP14-19371, 92802, 92864, 92895, 92996, 92920-92921, 92924 - 92925, 92937, 92936, 92941, 92943, 92944 OR- Measured 61 days prior to drug initiation to 3650 days prior to drug initiation in any procedure position and inpatient or outputient are setting - (CP2-9 procedure OC.66, 86.01, 36.02, 36.03, 36.05, 86.05, 86.05). | Petorno, Bisabetta et al. "Cardiovascular outcomer associated with canagificoin versus other non-gifficoin articlishetic drugs population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmjk119 |
| ſ | - The combination of revacularization in one-major coronary artery and significant stenosis | Starting: Measured 61 days prior to drug initiation to 3650 days prior to drug initiation in any procedure position and Inpatient care setting-CPT-4: 92980, 92981, 92928-92929, 93933-92934 OR- | Petrono, Disabetta et al. "Engagificorio and the Risk of Heart Failure Hospitalization in Routine Clinical Care:<br>A First Analysis Com the Engagificorio Comparative Michitemeses and Safety (IMMPRSS) Study," Circulation.<br>2019 Apr S. doi: 10.1161/CIRCULATIONANA.118.039177 |
| | | Measured 61 days prior to drug initiation to 3650 days prior to drug initiation in any procedure position and inpatient<br>or outpatient care setting-ICD-9 procedure: 36.06, 36.07 | |
| | | Transproper file reasoning tration: Measured 61 days prior to drug initiation to 3650 days prior to drug initiation in any procedure position and impatient care setting-CFT-4: 33140, 33141 CR - | |
| - | | Measured 61 days prior to drug initiation to 3650 days prior to drug initiation in any procedure position and inpatient<br>or outpatient care setting-ICD-9 procedure: 36.33-36.34 | |
| | <ul> <li>Folderce of single-vessel CAD, 250% furnised narrowing during angiography (coronary or multi-size computed tomography) not<br/>subsequently successfully researcherized, with at least 1 of the following:</li> </ul> | - | |
| - | - A positive non-invadive-threst test for ischemia | Measured 365 days prior to drug initiation in any diagnosis position and the inpatient care setting | |
| L | Hiospital discharge for unstable angina si 2 months prior to consent | ACS/unctable angine ICD-9 diagnosis: 411.ux | |
| se | Unitable angina >2 months prior to consent with evidence of single-or multi-vessel CAD | Measured 61 days prior to drug infiltration to 3650 days prior to drug initiation in any diagnosis position and the<br>outputted care setting<br>ACSUMEDIA and any NO-9 diagnosis: 611.xx | |
| sa | + lifettory of stroke (such emic or hemorrhagic) >2 months prior to consent | Measured 61 days prior to drug initiation to 3650 days prior to drug initiation in any diagnosis position and the Inpatient<br>or outpatient care witing | Patorno, Blazhetta et al. "Cardiovascular outcomes sacciated with canagificoin versus other non-gifficoin artificial-etic drugs population based cohort study," 884) 2018;360:s119 http://dx.doi.org/10.1196/bmjk119 |
| L | | <u>Aevetroke</u> ICO-9 diagnosis: 430.xx, 431.xx, 433.xx, 434.xx, 436.xx | Patonso, Blabbetta et al. "Ropagificion and the Risk of Heart Failure Hospitalization in Routine Clinical Care:<br>A First Analysis from the Empagificain Comparative Effectiveness and Safety (EMPRES) Study." Circulation.<br>2019 Apr B. doi: 10.1161/CIRCULATIONAVA.118.019177 |
| Г | Circlustve partipheral artery disease documented by any of the following: | Measured 180 days prior to drug infiliation in any procedure position and the impatient or outpatient care setting | Patomo, Bisabeta et al. "Cardiovascular outcomes associated with canagificoin versus other non-glificoin sertifishetic drugs population based cohort study," 884) 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 |
| | | Peripheral arterial stentingor surgical revocularization ICD-9 procedure 39.25, 39.50, 39.99 | Patomo, Blaubetta et al. "Impaglificoin and the Rick of Heart Failure Hospitalization in Routine Clinical Care:<br>A Rick Avaigist from the Impaglificoin Comparative Effectiveness and Safety (IMPRES) Study." Circulation.<br>2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| Se | —Umb angloplashy, steerling, or bignass surgery | Measured 180 days prior to drug initiation in any procedure position and the impatient or outpatient care setting<br>Lover-uniteditic broads: (CPP synchronic 1812, 9-19) (CPP synchronic 1812, 9-19) (CPP synchronic 1812, 9-19) (CPP synchronic 1812, 9-19) (CPP synchronic 1812, 9-19) (CPP synchronic 1815), 18565, 18566, | Petono, Blashetta et al. "Cardiovaccular outconse succiated with canagilifotin venus other non-glifotin articlated: drugs: population based cohort muly," BMJ 2018;360:bi19 http://dx.doi.org/10.1136/bmj.ki19 Petono, Blashetta et al. "Singagificoin and the Risk of Heart Failure Hospitalisation in Routine Clinical Care: A First Area (verying to ton the Engagificoin Congar ative Effectiveness and Safety (RMPRES) Study." Circulation. 2019 Apr S. doi: 10.1161/CRCULATIONAVIA.118.039177 |
| | -Unit or foot amountation due to circulatory insufficiency | Measured 180 days prior to drug initiation in any diagnosis/procedure position and the inpatient or outpatient care acting the inpatient procedure in the inpatient or outpatient care acting the international procedure is 4.10-4.18 [CD-9 procedure is 4.10-4.18 [Chypatien cold/CT-6: 27590, 27591, 27592, 27880, 27881, 27882, 27884, 27886, 27888, 27889, 28800, 28805, 28810, 28820, 288200, 2882000, 2882000, 2882000, 2882000, 28820000000000 | Patomo, Blashetta et al. "Cardiovascular outcomes sacciated with canagificoin versus other non-gifficoin artifiabatic drugs population based cohort mudy." 8849 2018;360:4:19 http://dx.doi.org/10.1136/dmi.kl/10.1136/d |

| | -Gridence of significant peripheral artery stenods (>50% on angiography, or >50% or hemodynamically significant via non-invasive methods)<br>in 1 limb | Measured 180 days prior to drug initiation in any diagnosis position and the inpatient or outpatient care setting<br><u>Parishwal vacuular diames</u> ICD+ diagnosis e40.20 –440.24, 440.29 –440.32, 440.3, 640.4, 643.9 | Patomo, Blashetta et al. "Cardiovacoular outcomes associated with caragifición versus other non-giffición<br>artifidabetic drugo: population based cohort study." BASI 2018;36(2):119.06(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2):119.07(2): |
|---|---|---|---|
| | - Anklebrachkil Index-40.9 in at ankle | Measured 180 days prior to drug initiation in any diagnosis position and the impatient or outpatient care setting<br>hold-bitachial index 40.9 ICD-9 diagnosis: 440.31 | |
| 6 | BMI 645 kg/m2 at baseline | Measured 180 days prior to drug initiation in any diagnosis position and the inpatient or outpatient care setting | |
| 7 | An estimated glomerular filtration rate (eGFR) of at least 30 ml per minute per 1.73 m2 of body-surface area | Morbid Chestry ICD-9 diagnosis: 278.01<br>N/A | |
| | Signed and dated written informed consent prior to screening in accordance with Good Clinical Practice and local legislation | N/A | |
| $\vdash$ | EXCLUSION CRITI | ERIA | |
| 1 | Uncontrolled hypergiv, emis with glucose >240 mg/dl, (>43.3 mmol/L) after an overnight fast during placebo nun-in and confirmed by a second measurement (not on the same day) | N/A | we disclided not to apply this criteria because we can captured hypergipt availabut can't captures everity of it<br>and we may end up looling many patients at this step. In case we disclide to apply it, the codes would be ICD-9<br>790.21 and ICD-90 973.01 |
| 2 | Indication of liver disease, defined by serum levels of slavine amininotrandersse, aspartate aminotrandersse, or sikaline phosphatase above<br>3 x upper limit of normal (VLN) during screening or run-in phase | Measured 590 days prior to and including day of drug initiation in any diagnosis/procedure position and the inpatient or outputient care setting <a associated="" canagifición="" cardiovascular="" href="https://diagnosis.org/lines/states-setting-lines/states-setting-states-setting-setti&lt;/th&gt;&lt;th&gt;Patomo, Bisabetta et al. " non-gifición<br="" other="" outcomes="" versus="" with="">artificiabett drugs population based cohort study." BMJ 2018;360:k119<br/>http://dx.doi.org/10.1136/phmj.k119<br/>ptomo, Bisabetta et al. "Enpagifición and the Ridu of Heart Fallure Hospitalization in Routine Clinical Care:<br/>A Rice Analysis from the Enpagifición Comparative (Biscotvenes and Safety (BMPRES) Study." Circulation.<br/>2019 Apr 8. doi: 10.1161/CIRCULATIONAVIA.118.039177</a> | |
| 3 | Planned cardiac surgery or angioplasty within 3 months | N/A | |
| 4 | Estimated glomerular filtration rate-30 mi/min/1.73m2 (according to the Modification of Diet in Renal Disease equation) at screening or during run-in phase | N/A. | N/A |
| 5 | Barlatric surgery within the past two years and other gestroint estinal surgeries that induce chronic malabsorption | Measured 780 days prior to drug finitiation in any procedure position and inputient or outpatient care setting CPT-6. CPT-6. 43644 - 1896 - Lapanoscopic Roux-en-Y gestric bepass (Roux limit 150 cm or less) 43645 - 189680- Lapanoscopic getric bypass with small intestine-ecconstruction to Brist absorption 43770 - 4469- Lapanoscopic adjustable gestric band 43770 - 4469- Lapanoscopic adjustable gestric band 43847 - 0469- Lapanoscopic adjustable gestric band 43847 - 0476- Lapanoscopic adjustable gestric band 43847 - 0476- 1049- Roux-en-Y gestric bypass (Roux limit 150 cm or less) 43847 - 0476- 1049- Roux-en-Y gestric bypass with untall intestine reconstruction to limit 43847 - 0476- 1049- 1 | Natours, ids 1, et al. "Clinical Factors Associated With Remission of Obedby-Related Consorbidities After Barlatric Surgery." JAMA Surg. 2016;151(2):180-137. doi:10.1001/Jamasurg.2015.3221 |
| 6 | Blood dyscrailas or any disorders causing hemolysis or unstable red blood cells e.g. malaria, babesiosis, hemolysis anemia) | Measured 190 days prior to and including day of drug initiation in any diagnosis position and inquitient or outpatient care setting. Greenest of the blood and blood-forming organs (ICD+0 diagnosis: 180.xx-189.xx, ICD-10 diagnosis: D50.xx-097.xx Malignost monitoris of the production of the setting of the blood of the product 100.xx-100.xx, ICD-10 diagnosis: C51.xx-C62.xx Hermochromatosis (ICD+0 diagnosis: 275.0x, ICD-10 diagnosis: C53.1.1x | |
| 7 | Medical history of cancer (suc apt for basal cell carcinoma) and/or trestment for cancer within the last 5 years | Measured 1825 days prior to drug initiation in any diagnosis position and inpatient or outpatient case setting<br>History of malignant necessary ICD-9 diagnosis: 140. so-206. so (escapt 173. so, non-melanoma skin cancer) | Patomo, Blashetta et al. "Cardiovascular outcomes associated with canagificion versus other non-gifficion<br>articlabellic druge population based cohort study." BMI 2018;3603119<br>http://dx.doi.org/10.1186/phis.1019<br>Patomo, Blashetta et al. "Engagificion and the Risk of Heart Fallure Hospitalization in Routine Clinical Care:<br>A Rick Analysis from the Engagificion and the Risk of Heart Fallure Hospitalization in Routine Clinical Care:<br>A Rick Analysis from the Engagificion Comparative Effectiveness and Safety (EMPRES) Study." Circulation.<br>2019 April. doi: 10.1161/ciRCULANDEWAL 118.0091777 |
| • | Contraindications to background therapy according to the local label | N/A | |
| , | Treatment with anti-obesity drugs 3 months prior to informed consent or any other treatment at time of screening feeding to unstable body weight (e.g. surgery, aggressive dist regimen, etc.) | Measured 90 days prior to drug infritation as a dispensing of one of the following medications: Use of criticat, forceserin, phentermine/bopksmate/(faed combo), bupropion/platesmone@tad combo), phentermine, destrujaropion, phendimetratine, beruphetamine, disutramine, destrutamine, for fluramine OR Measured 90 days prior to drug infritation in any diagnosis/procedure position and inpatient or outpatient care setting ICD=8 diagnosis 27% 0, 77% 00, 77% 01, 77% 03, 59% ou, 68% 15, 64% 12% VSC 5.14, VSC 5.45 CD=9 procedure 4312, 412, 413, 413, 413, 413, 414, 414, 414, 415, 415, 415, 415, 415 | Patomo, Blashetta et al. "Cardionacular outcomer saccclated with canagifiction versus other non-gifficein articlahetic drugs population based cohort mady." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patomo, Blashetta et al. "Snpagfificein and the Risk of Heart Fallure Hospitalization in Routine Clinical Care: A Rick Analysis from the Empagfificein comparative Effectiveness and Safety (SAPRES) Study." Circulation. 2019 Apr 8. doi: 10.1161/CRCULATIONAVIA.118.039177 |
| 10 | Treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent | Measured 42 days prior to drug initiation as a dispending of one of the following medications<br>Certicotesistic Continues, by decorrisons, predissons, predissons, methylpredissolons, triamcinolons,<br>desamethacons, betamethacone | Petonon, Blashets et al. "Cardiovescolar outcomes associated with canagificatin versus other non-glifficatin<br>writidatives drugs population based colour early." BMI 2018;190:b119<br>https://doi.org/10.1136/pnij.1119<br>Petrono, Blashets et al. "Engaglificatin and the Bok of Heart Fellure Hospitalization in Routine Clinical Care:<br>A Pirot Availables from the Engaglification Comparative (Bhot Versus and Salley (BMPHSI) Study." Circulation.<br>2019 April. doi: 10.1161/CRCULATIONNIA.118.039177 |
| 11 | Any uncontrolled endocrine disorder except T2DM | • | Weareunable to capture "uncontrolled" endoorine disorders. |

| _ | | | |
|---|---|---|---|
| 12 | Pre-menopausal women (last menstruation 61 year prior to informed consent) who were running, pregnant, or of child-bearing potential and we went practions as copylable method of birth control, or 66 not plan to continue using this method throughout the study, or 66 not agree to submit to periodic pregnancy testing during the trial. | Measured 180 days prior to and including day of drug initiation in any diagnosts position and inputient or outputient care setting. Broconter for contraceptivemanagement ICD-9 diagnosts VSS R Presency—See "Pregnancy" for ICD-9 diagnosts and procedure codes. CR Measured 180 days prior to and including day of drug initiation as a dispensing of one of the following medications Non-oral contraceptives (brand names)- Deposalid. Provers 104 Depo-Trovers, generic Mirrors Crtho Iora Narvaling Implanon Collacontraceptives (generic names)- See "oral contraceptives—generic" theet. Cral contraceptives (generic names)- See "oral contraceptives—brand" dheet. | Krumme, Alexie A, et. al. "Study protocol for the dabigatran, aploaban, rivarousban, edocaban, warhrin comparative effectiveness research study." J. Comp. Eff. Rec. (2018):7(1), 57-66. doi: 10.2217/ce-2017-0053. We excluded patients using contract aptives because this trial includes non-pregnant women, patients without childhesing potential, and patients who have-childhesing potential but are taking precardions such as oral contraceptive incomparany other weep/10 avoid pregnancy during theretial pariod. It is impossible to implement such inclusion in real-world data, as childhesing potential in oral recording in claims. In this trials used to the following: [jillack on incomplement as an inclusion criteria is due to the following: [jillack of nexcoding of contraceptive and other precardions to avoid pregnancy and lighatients with disbets and baseline-CYteed to be older and a en or likely to be act following on Three whose, we assumed that patients stating coal contraceptive have childhesing potential, on if they were to stop contraceptive use excludes very few patients (hypically) see than 0.1% of patients). |
| | -Acceptable methods of birth control include tubal ligation, transfermal patch, intrauserine devices/systems, oral, implantable or<br>injectable contraceptives, sessal abstinence, double barrier method, vasectomy of partner | | |
| 13 | Alcohol or drug abuse within 3 months of informed consent that would interfere with trial participation or any ongoing condition leading to decreased compliance with study procedures or study drug intake | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inspatient or outpatient core setting. Alcohol abserts dependence ICD-9 diagnosis: 291.w., 203.w., 205.bs, 571.bs, 571.bs, 571.bs, 571.bs, 357.bs, 425.5s, 586.0s, V11.bs Days abset or dependence ICD-9 diagnosis: 292.xs, 204.xs, 205.2x-305.9s, 648.bs | Patons, Blashetta et al. "Cardiovascular outcomes associated with canagifición versus other non-gifición<br>artificiás-leic druges population based cohort study." BMI 2018;360:k119<br>http://dx.doi.org/10.1136/bmi.jk119<br>Patorno, Blashetta et al. "Enpagifición and the-Rick of Heart Failure Hospitalization in Routine Clinical Care:<br>A Rick Analysis from the Enpagifición Comparative Bibicultureus and Safety (BMPRES) Study." Circulation.<br>2018 April. doi: 10.1161/c/BRCUROWWA 118.0.00177 |
| 34 | intake of an investigational drug in another trial within 30 days prior to intake of study medication in this trial or participating in another trial involving an investigational drug and/or fallow-up | N/A | |
| 15 | Any clinical condition that would jeopardize patient sufety while participating in this clinical trial (in Canada, this included current genito-<br>urinal infection or genito-urinal infection within 2 weeks prior to informed consent) | N/A | |
| 36 | Acute-coronary syndrome, stroke, or translent ischemic attack within 2 months prior to informed consent | Measured 50 days prior to day of drug hithation in any diagnosis position and inpatient or outpatient care setting- ACG annuals augins CV-8 diagnosis et 81.x s. 20x1a; CD-8 diagnosis: 40.0x siderarchosis in monthage (240) 40.0x siderarchosis in benonthage (240) 40.0x siderarchos | Patomo, Bisabetta et al. "Cardiovascular outcomes associated with canagifician versus other non-giffician artificial-sets population based cohort suby." BMI 2018;3603119 https://dx.doi.org/10.1136/pmi.2011.136/pmi |
| 17 | In South Africa: blood pressure >1.60/100 mmHg at screening | N/A | |

| Trial ID | sNDA21 |
|---|---|
| Trial Name (with web links) | EMPA-REG OUTCOME |
| Trial Name (with pdf links) | EMPA-REG OUTCOME |
| NCT | NCT01131676 |
| Trial category | Secondary indication |
| Therapeutic Area | Endocrinology |
| RCT Category | 4a- Unintended S with label change |
| Brand Name | Synjardy |
| Generic Name | Empagliflozin; metformin hydrochloride |
| <u>Sponsor</u> | Boehringer Ingelheim |
| <u>Year</u> | 2016 |
| Measurable endpoint | Primary composite endpoint of CV death, non-fatal MI, non-fatal stroke |
| <u>Exposure</u> | Empagliflozin |
| <u>Comparator</u> | Placebo |
| <u>Population</u> | 95% on Anti-hypertensive therapy, 80% on Lipid-lowering therapy & 89% on Anti-coagulants |
| Trial finding | HR = 0.86 (95% CI 0.74–0.99) |
| No. of Patients | 7,064 |
| Non-inferiority margin | HR=1.3 |
| Assay Sens. Endpoint | |
| Assav Sens. Finding | |
| | 0.90. For the test of noninferiority for the primary outcome with a margin of 1.3 at a one-sided level of 0.0249, at least 691 events were |
| <u>Power</u> | required to provide a power of at least 90% on the assumption of a true hazard ratio of 1.0. |
| Blinding | Double-blinded |
| | Accidental superiority, the non-inferiority margin was chosen as 1.3 based on Food and Drug Administration (FDA) Guidance for Industry – |
| Statistical Method | Diabetes Mellitus – Evaluating Cardiovascular Risk in New Antidiabetic Therapies to Treat Type 2 Diabetes |
| Approval indication | Proposes a new indication for Synjardy based on results of the cardiovascular safety study 1245.25, the EMPA-REG OUTCOME trial. |

## Mortality-Dependent on data source. 1. All-cause mortality / inpatient mortality Identified using the vital status file-Medicare Identified using the discharge status codes-Optum-20 = EXPIRED • 21 = EXPIRED TO BE DEFINED AT STATE LEVEL 22 = EXPIRED TO BE DEFINED AT STATE LEVEL 23 = EXPIRED TO BE DEFINED AT STATE LEVEL 24 = EXPIRED TO BE DEFINED AT STATE LEVEL 25 = EXPIRED TO BE DEFINED AT STATE LEVEL 26 = EXPIRED TO BE DEFINED AT STATE LEVEL 27 = EXPIRED TO BE DEFINED AT STATE LEVEL • 28 = EXPIRED TO BE DEFINED AT STATE LEVEL • 29 = EXPIRED TO BE DEFINED AT STATE LEVEL 40 = EXPIRED AT HOME (HOSPICE) 41 = EXPIRED IN A MEDICAL FACILITY (HOSPICE) 42 = EXPIRED - PLACE UNKNOWN (HOSPICE) Truven- 20 - Died 22 - Died • 23 - Died • 24 - Died 25 - Died 26 - Died 27 - Died 28 - Died 29 - Died

• 40 - Other died status or Expired at home (Hospice claims only) (depends on year)

- 41 Other died status or Expired in medical facility (Hospice claims only) (depends on year)
- 42 Other died status or Expired place unknown (Hospice claims only) (depends on year)
- 21 Died or Disch./Transf. to court/law enforcement (depends on year)

### 2. CV mortality

Information on CV mortality through data linkage with the National Death Index (NDI) will be available for Medicare at a later date. We will conduct secondary analyses using CV mortality at that time.

| Antidiabetic class | Specific agent | Notes |
|---|---|---|
| | Canagliflozin | Approved 3/29/2013 |
| SGLT2-inhibitors | Dapagliflozin | |
| SGL12-minonors | Empagliflozin | |
| | Ertugliflozin | Approved Dec 21, 2017 |
| | Glimepiride | |
| 2 <sup>nd</sup> generation sulfonylureas | Glipizide | |
| | Glyburide | |
| | Alogliptin | |
| DPP-4 inhibitors | Linagliptin | |
| DPP-4 inhibitors | Saxagliptin | |
| | Sitagliptin | |
| | Exenatide | |
| | Liraglutide | |
| GLP-1 receptor agonist (GLP1-RA) | Albiglutide | Approved April 15, 2014 and discontinued July 26, 2017 |
| | Dulaglutide | Approved Sep 18, 2014 |
| | Lixisenatide | Approved July 28, 2016 |
| | Semaglutide | Approved Dec 5, 2017 |
| | Insulin Aspart | |
| | Insulin Aspart/Insulin Aspart Protamine | |
| | Insulin Degludec | |
| | Insulin Detemir | |
| | Insulin Glargine | |
| | Insulin Glulisine | |
| Insulin | Insulin human isophane (NPH) | |
| | Insulin human regular (search with NPH, | |
| | don't want bf-pk) | |
| | Insulin human regular/ Insulin human isophane (NPH) | |
| | Insulin Lispro | |
| | Insulin Lispro/Insulin Lispro Protamine | |
| Glitzzones | Pioglitazone | |

| Опидонея | Rosiglitazone |
|------------------------------------------|----------------|
| Meglitinides | Nateglinide |
| Megnimides | Repaglinide |
| Alaba alaaasidaa inkikisaa | Acarbose |
| Alpha-glucosidase inhibitors | Miglitol |
| Pramlintide | Pramlintide |
| 45 10 1 | Acetohexamide |
| | Chlorpropamide |
| 1 <sup>st</sup> generation sulfonylureas | Tolazamide |
| | Tolbutamide |

| drug_class | Brand Name |
|--------------------|---------------|
| oral contraceptive | Apri; |
| oral contraceptive | Desogen; |
| oral contraceptive | Ortho-Cept; |
| oral contraceptive | Reclipsen |
| oral contraceptive | Kariva; |
| oral contraceptive | Mircette |
| oral contraceptive | Cyclessa; |
| oral contraceptive | Velivet |
| oral contraceptive | Yasmin |
| oral contraceptive | Yaz |
| oral contraceptive | Demulen 1/35; |
| oral contraceptive | Kelnor; |
| oral contraceptive | Zovia 1/25 |
| oral contraceptive | Demulen 1/50; |
| oral contraceptive | Zovia 1/50 |
| oral contraceptive | Alesse; |
| oral contraceptive | Aviane; |
| oral contraceptive | Lessina; |
| oral contraceptive | Lutera |
| oral contraceptive | Nordette; |
| oral contraceptive | Portia; |
| oral contraceptive | Levora |
| oral contraceptive | Lybrel |
| oral contraceptive | Seasonale; |
| oral contraceptive | Quasense; |
| oral contraceptive | Jolessa |
| oral contraceptive | Seasonique |
| oral contraceptive | Empresse; |
| oral contraceptive | Triphasil; |
| oral contraceptive | Trivora |
| oral contraceptive | Ovcon 35 |
| oral contraceptive | Balziva; |

| oral contraceptive | Femcon Fe |
|--------------------|----------------------|
| oral contraceptive | Brevicon; |
| oral contraceptive | Nortrel 0.5/35; |
| oral contraceptive | Modicon; |
| oral contraceptive | Necon 0.5/35 |
| oral contraceptive | Norinyl 1/35; |
| oral contraceptive | Nortrel 1/35; |
| oral contraceptive | Ortho-Novum 1/35; |
| oral contraceptive | Necon 1/35 |
| oral contraceptive | Ovcon 50; |
| oral contraceptive | Necon 1/50 |
| oral contraceptive | Ortho-Novum 10/11 |
| oral contraceptive | Aranelle; |
| oral contraceptive | Tri-Norinyl |
| oral contraceptive | Ortho-Novum 7/7/7; |
| oral contraceptive | Necon |
| oral contraceptive | Micronor; |
| oral contraceptive | Nor-QD; |
| oral contraceptive | Camila; |
| oral contraceptive | Emin; |
| oral contraceptive | Jolivette |
| oral contraceptive | Junel 21 1/20; |
| oral contraceptive | Junel 21 Fe 1/20; |
| oral contraceptive | Loestrin 21 1/20; |
| oral contraceptive | Loestrin 21 Fe 1/20; |
| oral contraceptive | Loestrin 24 Fe; |
| oral contraceptive | Microgestin 1/20 |
| oral contraceptive | Microgestin Fe 1/20 |
| oral contraceptive | Junel 21 1.5/30; |
| oral contraceptive | Junel 21 Fe 1.5/30; |
| oral contraceptive | Loestrin 1.5/30; |
| oral contraceptive | Loestrin Fe 1.5/30 |
| oral contraceptive | Microgestin 1.5/30 |

| oral contraceptive | Microgestin Fe 1.5/30 |
|--------------------|-----------------------|
| oral contraceptive | Estrostep Fe; |
| oral contraceptive | Tilia Fe; |
| oral contraceptive | TriLegest Fe |
| oral contraceptive | Ortho-Cyclen; |
| oral contraceptive | Sprintec; |
| oral contraceptive | MonoNessa; |
| oral contraceptive | Previfem |
| oral contraceptive | Ortho Tri-Cyclen Lo; |
| oral contraceptive | Tri-Previfem; |
| oral contraceptive | TriNessa |
| oral contraceptive | Ortho Tri-Cyclen; |
| oral contraceptive | Tri-Sprintec |
| oral contraceptive | Cryselle; |
| oral contraceptive | Lo/Ovral; |
| oral contraceptive | Low-Ogestrel |
| oral contraceptive | Ovral; |
| oral contraceptive | Ogestrel |
| oral contraceptive | Zovia 1/50 |
| oral contraceptive | Alesse; |
| oral contraceptive | Aviane; |
| oral contraceptive | Lessina; |
| oral contraceptive | Lutera |
| oral contraceptive | Nordette; |
| oral contraceptive | Portia; |
| oral contraceptive | Levora |
| oral contraceptive | Lybrel |
| oral contraceptive | Seasonale; |
| oral contraceptive | Quasense; |
| oral contraceptive | Jolessa |
| oral contraceptive | Seasonique |
| oral contraceptive | Empresse; |
| oral contraceptive | Triphasil; |

| oral contraceptive | Trivora |
|--------------------|----------------------|
| oral contraceptive | Ovcon 35 |
| oral contraceptive | Balziva: |
| oral contraceptive | Femcon Fe |
| oral contraceptive | Brevicon; |
| oral contraceptive | Nortrel 0.5/35; |
| oral contraceptive | Modicon; |
| oral contraceptive | Necon 0.5/35 |
| oral contraceptive | Norinyl 1/35; |
| oral contraceptive | Nortrel 1/35: |
| oral contraceptive | Ortho-Novum 1/35; |
| oral contraceptive | Necon 1/35 |
| oral contraceptive | Ovcon 50; |
| oral contraceptive | Necon 1/50 |
| oral contraceptive | Ortho-Novum 10/11 |
| oral contraceptive | Aranelle; |
| oral contraceptive | Tri-Norinyl |
| oral contraceptive | Ortho-Novum 7/7/7; |
| oral contraceptive | Necon |
| oral contraceptive | Micronor; |
| oral contraceptive | Nor-QD; |
| oral contraceptive | Camila: |
| oral contraceptive | Emin: |
| oral contraceptive | Jolivette |
| oral contraceptive | Junel 21 1/20; |
| oral contraceptive | Junel 21 Fe 1/20; |
| oral contraceptive | Loestrin 21 1/20; |
| oral contraceptive | Loestrin 21 Fe 1/20; |
| oral contraceptive | Loestrin 24 Fe; |
| oral contraceptive | Microgestin 1/20 |
| oral contraceptive | Microgestin Fe 1/20 |
| oral contraceptive | Junel 21 1.5/30; |
| oral contraceptive | Junel 21 Fe 1.5/30; |

| oral contraceptive | Loestrin 1.5/30; |
|--------------------|-----------------------|
| oral contraceptive | Loestrin Fe 1.5/30 |
| oral contraceptive | Microgestin 1.5/30 |
| oral contraceptive | Microgestin Fe 1.5/30 |
| oral contraceptive | Estrostep Fe; |
| oral contraceptive | Tilia Fe; |
| oral contraceptive | TriLegest Fe |
| oral contraceptive | Ortho-Cyclen; |
| oral contraceptive | Sprintec; |
| oral contraceptive | MonoNessa; |
| oral contraceptive | Previfem |
| oral contraceptive | Ortho Tri-Cyclen Lo; |
| oral contraceptive | Tri-Previfem; |
| oral contraceptive | TriNessa |
| oral contraceptive | Ortho Tri-Cyclen; |
| oral contraceptive | Tri-Sprintec |
| oral contraceptive | Cryselle; |
| oral contraceptive | Lo/Ovral; |
| oral contraceptive | Low-Ogestrel |
| oral contraceptive | Ovral; |
| oral contraceptive | Ogestrel |

| drug_class | generic | generic_ndc |
|---|---|---|
| oral contraceptive | estradiol | desogestrel-ethinyl estradiol |
| oral contraceptive | estradiol | desogestrel-ethinyl estradiol/ethinyl estradiol |
| oral contraceptive | estradiol | drospirenone/estradiol |
| oral contraceptive | estradiol | drospirenone/ethinyl estradiol/levomefolate calcium |
| oral contraceptive | estradiol | estradiol |
| oral contraceptive | estradiol | estradiol acetate |
| oral contraceptive | estradiol | estradiol benzoate |
| oral contraceptive | estradiol | estradiol cypionate |
| oral contraceptive | estradiol | estradiol cypionate/medroxyprogesterone acet |
| oral contraceptive | estradiol | estradiol hemihydrate, micronized |
| oral contraceptive | estradiol | estradiol micronized |
| oral contraceptive | estradiol | estradiol valerate |
| oral contraceptive | estradiol | estradiol valerate/dienogest |
| oral contraceptive | estradiol | estradiol valerate/sesame oil |
| oral contraceptive | estradiol | estradiol/estrone |
| oral contraceptive | estradiol | estradiol/estrone/vit b12 |
| oral contraceptive | estradiol | estradiol/levonorgestrel |
| oral contraceptive | estradiol | estradiol/norethindrone acetate |
| oral contraceptive | estradiol | estradiol/norgestimate |
| oral contraceptive | estradiol | estradiol/progesterone |
| oral contraceptive | estradiol | ethinyl estradiol |
| oral contraceptive | estradiol | ethinyl estradiol/drospirenone |
| oral contraceptive | estradiol | ethinyl estradiol/norethindrone acetate |
| oral contraceptive | estradiol | ethynodiol d-ethinyl estradiol |
| oral contraceptive | estradiol | ethynodiol diacetate-ethinyl estradiol |
| oral contraceptive | estradiol | etonogestrel/ethinyl estradiol |
| oral contraceptive | estradiol | levonorgestrel-ethinyl estradiol |
| oral contraceptive | estradiol | levonorgestrel/ethinyl estradiol and ethinyl estradiol |
| oral contraceptive | estradiol | me-testosterone/eth estradiol |
| oral contraceptive | estradiol | metttm/estradiol/multivits |
| oral contraceptive | estradiol | norelgestromin/ethinyl estradiol |
| oral contraceptive | estradiol | norethindrone a-e estradiol |

| oral contraceptive | estradiol | norethindrone a-e estradiol/fe |
|---|---|---|
| oral contraceptive | estradiol | norethindrone a-e estradiol/ferrous fumarate |
| oral contraceptive | estradiol | norethindrone acetate-ethinyl estradiol |
| oral contraceptive | estradiol | norethindrone acetate-ethinyl estradiol/ferrous fumarate |
| oral contraceptive | estradiol | norethindrone-ethin estradiol |
| oral contraceptive | estradiol | norethindrone-ethinyl estradiol |
| oral contraceptive | estradiol | norethindrone-ethinyl estradiol/ferrous fumarate |
| oral contraceptive | estradiol | norgestimate-ethinyl estradiol |
| oral contraceptive | estradiol | norgestrel-ethinyl estradiol |
| oral contraceptive | estradiol | testosterone cypionate/estradiol cypionate |
| oral contraceptive | estradiol | testosterone enanthate/estradiol valerate |
| oral contraceptive | estradiol | testosterone/estradiol |
| oral contraceptive | levonorgestrel | estradiol/levonorgestrel |
| oral contraceptive | levonorgestrel | levonorgestrel |
| oral contraceptive | levonorgestrel | levonorgestrel-eth estra |
| oral contraceptive | levonorgestrel | levonorgestrel-eth estra/pregnancy test kit |
| oral contraceptive | levonorgestrel | levonorgestrel-ethinyl estradiol |
| oral contraceptive | levonorgestrel | levonorgestrel/ethinyl estradiol and ethinyl estradiol |
| oral contraceptive | norethindrone | estradiol/norethindrone acetate |
| oral contraceptive | norethindrone | ethinyl estradiol/norethindrone acetate |
| oral contraceptive | norethindrone | leuprolide acetate/norethindrone acetate |
| oral contraceptive | norethindrone | norethindrone |
| oral contraceptive | norethindrone | norethindrone a-e estradiol |
| oral contraceptive | norethindrone | norethindrone a-e estradiol/fe |
| oral contraceptive | norethindrone | norethindrone a-e estradiol/ferrous fumarate |
| oral contraceptive | norethindrone | norethindrone acetate |
| oral contraceptive | norethindrone | norethindrone acetate-ethinyl estradiol |
| oral contraceptive | norethindrone | norethindrone acetate-ethinyl estradiol/ferrous fumarate |
| oral contraceptive | norethindrone | norethindrone-ethin estradiol |
| oral contraceptive | norethindrone | norethindrone-ethinyl estrad |
| oral contraceptive | norethindrone | norethindrone-ethinyl estradiol |
| oral contraceptive | norethindrone | norethindrone-ethinyl estradiol/ferrous fumarate |

| oral contraceptive | norethindrone | norethindrone-mestranol |
|--------------------|-------------------------|------------------------------|
| oral contraceptive | norgestrel | norgestrel |
| oral contraceptive | norgestrel | norgestrel-ethinyl estradiol |
| oral contraceptive | polyestradiol phosphate | polyestradiol phosphate |

## Pregnancy Dx codes 650 NORMAL DELIVERY 660 OBSTRUCTED LABOR 661 ABNORMALITY OF FORCES OF LABOR 662 LONG LABOR 663 UMBILICAL CORD COMPLICATIONS DURING LABOR AND DELIVERY 664 TRAUMA TO PERINEUM AND VULVA DURING DELIVERY 665 OTHER OBSTETRICAL TRAUMA 667 RETAINED PLACENTA OR MEMBRANES WITHOUT HEMORRHAGE 668 COMPLICATIONS OF THE ADMINISTRATION OF ANESTHETIC OR OTHER SEDATION IN LABOR AND DELIVERY 669.94 UNSPECIFIED COMPLICATION OF LABOR AND DELIVERY POSTPARTUM CONDITION OR COMPLICATION V24 POSTPARTUM CARE AND EXAMINATION V24.0 POSTPARTUM CARE AND EXAMINATION IMMEDIATELY AFTER DELIVERY V24.1 POSTPARTUM CARE AND EXAMINATION OF LACTATING MOTHER V24.2 ROUTINE POSTPARTUM FOLLOW V27 OUTCOME OF DELIVERY V27.0 MOTHER WITH SINGLE LIVEBORN V27.1 MOTHER WITH SINGLE STILLBORN V27.2 MOTHER WITH TWINS BOTH LIVEBORN V27.3 MOTHER WITH TWINS ONE LIVEBORN AND ONE STILLBORN V27.4 MOTHER WITH TWINS BOTH STILLBORN V27.5 MOTHER WITH OTHER MULTIPLE BIRTH ALL LIVEBORN V27.6 MOTHER WITH OTHER MULTIPLE BIRTH SOME LIVEBORN V27.7 MOTHER WITH OTHER MULTIPLE BIRTH ALL STILLBORN V27.9 MOTHER WITH UNSPECIFIED OUTCOME OF DELIVERY Procedure codes 72.0 LOW FORCEPS OPERATION 72.1 LOW FORCEPS OPERATION WITH EPISIOTOMY 72.2 MID FORCEPS OPERATION 72.21 MID FORCEPS OPERATION WITH EPISIOTOMY 72.29 OTHER MID FORCEPS OPERATION 72.3 HIGH FORCEPS OPERATION 72.31 HIGH FORCEPS OPERATION WITH EPISIOTOMY 72.39 OTHER HIGH FORCEPS OPERATION

| 72.4 FORCEPS ROTATION OF FETAL HEAD |
|------------------------------------------------------------------|
| 72.5 BREECH EXTRACTION |
| 72.51 PARTIAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD |
| 72.52 OTHER PARTIAL BREECH EXTRACTION |
| 72.53 TOTAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD |
| 72.54 OTHER TOTAL BREECH EXTRACTION |
| 72.6 FORCEPS APPLICATION TO AFTERCOMING HEAD |
| 72.7 VACUUM EXTRACTION |
| 72.71 VACUUM EXTRACTION WITH EPISIOTOMY |
| 72.79 OTHER VACUUM EXTRACTION |
| 72.8 OTHER SPECIFIED INSTRUMENTAL DELIVERY |
| 72.9 UNSPECIFIED INSTRUMENTAL DELIVERY |
| 73.0 ARTIFICIAL RUPTURE OF MEMBRANES |
| 73.01 INDUCTION OF LABOR BY ARTIFICIAL RUPTURE OF MEMBRANES |
| 73.09 OTHER ARTIFICIAL RUPTURE OF MEMBRANES |
| 73.1 OTHER SURGICAL INDUCTION OF LABOR |
| 73.2 INTERNAL AND COMBINED VERSION AND EXTRACTION |
| 73.21 INTERNAL AND COMBINED VERSION WITHOUT EXTRACTION |
| 73.22 INTERNAL AND COMBINED VERSION WITH EXTRACTION |
| 73.3 FAILED FORCEPS |
| 73.4 MEDICAL INDUCTION OF LABOR |
| 73.5 MANUALLY ASSISTED DELIVERY |
| 73.51 MANUAL ROTATION OF FETAL HEAD |
| 73.59 OTHER MANUALLY ASSISTED DELIVERY |
| 73.6 EPISIOTOMY |
| 73.8 OPERATIONS ON FETUS TO FACILITATE DELIVERY |

73.9 OTHER OPERATIONS ASSISTING DELIVERY
73.91 EXTERNAL VERSION ASSISTING DELIVERY

73.93 INCISION OF CERVIX TO ASSIST DELIVERY

73.99 OTHER OPERATIONS ASSISTING DELIVERY

73.94 PUBIOTOMY TO ASSIST DELIVERY

74.0 CLASSICAL CESAREAN SECTION
74.1 LOW CERVICAL CESAREAN SECTION
74.2 EXTRAPERITONEAL CESAREAN SECTION

73.92 REPLACEMENT OF PROLAPSED UMBILICAL CORD

- 74.3 REMOVAL OF EXTRATUBAL ECTOPIC PREGNANCY
- 74.4 CESAREAN SECTION OF OTHER SPECIFIED TYPE
- 74.9 CESAREAN SECTION OF UNSPECIFIED TYPE
- 74.91 HYSTEROTOMY TO TERMINATE PREGNANCY
- 74.99 OTHER CESAREAN SECTION OF UNSPECIFIED TYPE
- 75.4 MANUAL REMOVAL OF RETAINED PLACENTA
- 75.5 REPAIR OF CURRENT OBSTETRIC LACERATION OF UTERUS
- 75.6 REPAIR OF OTHER CURRENT OBSTETRIC LACERATION
- 75.7 MANUAL EXPLORATION OF UTERINE CAVITY, POSTPARTUM
- 75.9 OTHER OBSTETRIC OPERATIONS
#### Appendix B



| | Unmatched | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| · · | Optu | m | Market | ican | Medicare | | | POOLED | |
| • | Орго | Exposure - Empaginican | | Exposure - Empagimozin | THE GIVE | Exposure - | | Exposure - Empaginiozin | |
| Variable | Reference-DPP4i v2 | v3 | Reference-DPP4iv2 | v3 | Reference-DPP4i v2 | | Reference-DPP4iv2 | v3 | St. Diff. |
| Number of patients | 99,903 | 27,394 | 98,345 | 18,912 | 203,294 | 13,156 | 401,542 | 59,462 | |
| Age | | | | | | | | | |
| mean (sd) | 64.93 (11.69) | 60.53 (10.62) | 58.66 (11.12) | 55.47 (8.77) | 74.08 (6.94) | 71.46 (5.19) | 68.03 (9.42) | 61.34 (9.08) | 0.72 |
| median [IQR] | 66.00 [37.00, 73.00] | 61.00 [53.00, 68.00] | 58.00 [52.00, 64.00] | 56.00 [50.00, 61.00] | 73.00 [68.00, 78.00] 0 | .00 [68.00, 74.00] | 67.58 (9.42) | 61.40 (9.08) | 0.67 |
| Age categories without zero category | | | | | | | | | |
| 18 - 54; n (%) | 19,490 (19.5%) | 7,748 (28.3%) | 33,966 (34.5%) | 7,944 (42.0%) | 0 (0.0%) | 0 (0.0%) | 53,456 (13.3%) | 15,692 (26.4%) | -0.33 |
| 55 -64; n (%) | 23,551 (23.6%) | 8,844 (32.3%) | 41,612 (42.3%) | 9,123 (48.2%) | 1,132 (0.6%) | 43 (0.3%) | 66,295 (16.5%) | 18,010 (30.3%) | -0.33<br>0.18 |
| 65 - 74; n (%)<br>>=75; n (%) | 36,281 (36.3%)<br>20,581 (20.6%) | 8,539 (31.2%)<br>2,263 (8.3%) | 13,769 (14.0%)<br>8,998 (9.1%) | 1,483 (7.8%)<br>362 (1.9%) | 119,235 (58.7%)<br>82,927 (40.8%) | 9,986 (75.9%)<br>3,127 (23.8%) | 169,285 (42.2%)<br>112,506 (28.0%) | 20,008 (33.6%)<br>5,752 (9.7%) | 0.18 |
| Gender without zero category-United | 20,361 (20.6/6) | 2,203 (0.3/9) | 0,330 [3.1/6] | 302 (1.3/6) | 02,327 [40.070] | 3,127 (23.0/9) | 112,300 (20.0/6) | 3,732 (3.770) | 0.46 |
| Males; n (%) | 53,340 (53.4%) | 16,618 (60.7%) | 57,603 (58.6%) | 11,785 (62.3%) | 92,595 (45.5%) | 7,494 (57.0%) | 203,538 (50.7%) | 35,897 (60.4%) | -0.20 |
| Females; n (%) | 46,563 (46.6%) | 10,776 (39.3%) | 40,742 (41.4%) | 7,127 (37.7%) | 110,699 (54.5%) | 5,662 (43.0%) | 198,004 (49.3%) | 23,565 (39.6%) | 0.20 |
| Race | | | | | | | | | |
| White; n (%) | N/A | N/A | N/A | N/A | 151,073 (74.3%) | 10,799 (82.1%) | 151,073 (74.3%) | 10,799 (82.1%) | -0.19 |
| Black; n (%) | N/A | N/A | N/A | N/A | 22,905 (11.3%) | 916 (7.0%) | 22,905 (11.3%) | 916 (7.0%) | 0.15 |
| Asian; n (%) | N/A | N/A | N/A | N/A | 9,749 (4.8%) | 387 (2.9%) | 9,749 (4.8%) | 387 (2.9%) | 0.10 |
| Hispanic; n (%) | N/A | N/A | N/A | N/A | 9,554 (4.7%) | 333 (2.5%) | 9,554 (4.7%) | 333 (2.5%) | 0.12 |
| North American Native; n (%) | N/A | N/A | N/A | N/A | 1,385 (0.7%) | 58 (0.4%) | 1,385 (0.7%) | 58 (0.4%) | 0.04 |
| Other/Unknown; n (%) | N/A | N/A | N/A | N/A | 8,628 (4.2%) | 663 (5.0%) | 8,628 (4.2%) | 663 (5.0%) | -0.04 |
| Region without zero category-United v3 (lumping missing | &other category with West) | | | | | | | | |
| Northeast; n (%) | 10,960 (11.0%) | 2,334 (8.5%) | 17,603 (17.9%) | 2,575 (13.6%) | 38,218 (18.8%) | 2,505 (19.0%) | 66,781 (16.6%) | 7,414 (12.5%) | 0.12 |
| South; n (%) | 52,164 (52.2%) | 15,303 (55.9%) | 20,254 (20.6%) | 3,296 (17.4%) | 86,895 (42.7%) | 5,524 (42.0%) | 159,313 (39.7%) | 24,123 (40.6%) | -0.02 |
| Midwest; n (%) | 18,103 (18.1%) | 5,373 (19.6%) | 50,370 (51.2%) | 11,006 (38.2%) | 42,468 (20.9%) | 2,506 (19.0%) | 110,941 (27.6%) | 18,885 (31.8%) | -0.09 |
| West; n (%) | 18,676 (18.7%) | 4,384 (16.0%) | 9,489 (9.6%) | 1,978 (10.5%) | 35,713 (17.6%) | 2,621 (19.9%) | 63,878 (15.9%) | 8,983 (15.1%) | 0.02 |
| Unknown+missing; n (%) | N/A | N/A | 629 (0.6%) | 57 (0.3%) | N/A | N/A | 629 (0.6%) | 57 (0.3%) | 0.04 |
| CV Covariates | | | | | | | | | |
| Ischemicheart disease; n (%)<br>Acute MI; n (%) | 18,990 (19.0%)<br>931 (0.9%) | 5,885 (21.5%)<br>344 (1.3%) | 12,693 (12.9%)<br>372 (0.4%) | 2,535 (13.4%)<br>104 (0.5%) | 54,534 (26.8%)<br>1,288 (0.6%) | 4,200 (31.9%)<br>89 (0.7%) | 86,217 (21.5%)<br>2,591 (0.6%) | 12,620 (21.2%)<br>537 (0.9%) | 0.01<br>-0.03 |
| ACS/unstable angina; n (%) | 702 (0.7%) | 231 (0.8%) | 300 (0.5%) | 107 (0.6%) | 1,499 (0.7%) | 118 (0.9%) | 2,701 (0.7%) | 456 (0.8%) | -0.01 |
| Old MI; n (%) | 2,549 (2.6%) | 819 (3.0%) | 906 (0.9%) | 191 (1.0%) | 5,824 (2.9%) | 466 (3.5%) | 9,279 (2.3%) | 1,476 (2.5%) | -0.01 |
| Stable angina; n (%) | 3,164 (3.2%) | 1,100 (4.0%) | 1,545 (1.6%) | 382 (2.0%) | 6,343 (3.1%) | 626 (4.8%) | 11,052 (2.8%) | 2,108 (3.5%) | -0.04 |
| Coronary atherosclerosis and other forms of chronic ischer | 17,701 (17.7%) | 5,558 (20.3%) | 11,987 (12.2%) | 2,406 (12.7%) | 52,219 (25.7%) | 4,074 (31.0%) | 81,907 (20.4%) | 12,038 (20.2%) | 0.00 |
| Other atherosclerosis with ICD10 v2 Copy; n (%) | 501 (0.5%) | 106 (0.4%) | 451 (0.5%) | 57 (0.3%) | 2,443 (1.2%) | 86 (0.7%) | 3,395 (0.8%) | 249 (0.4%) | 0.05 |
| Previous cardiac procedure (CABG or PTCA or Stent) v4; n (5 | 407 (0.4%) | 189 (0.7%) | 212 (0.2%) | 52 (0.3%) | 461 (0.2%) | 55 (0.4%) | 1,080 (0.3%) | 296 (0.5%) | -0.03 |
| History of CABG or PTCA; n (%) | 4,493 (4.5%) | 1,679 (6.1%) | 1,629 (1.7%) | 369 (2.0%) | 13,342 (6.6%) | 1,156 (8.8%) | 19,464 (4.8%) | 3,204 (5.4%) | -0.03 |
| Anystroke; n (%) | 4,963 (5.0%) | 1,153 (4.2%) | 2,035 (2.1%) | 273 (1.4%) | 10,123 (5.0%) | 391 (4.3%) | 17,121 (4.3%) | 2,017 (3.4%) | 0.05 |
| | 4,000 (0.0.4) | 2,222(1.2.4) | 2,000 [2.2.4] | 2.0 (2) | 20,223 (3.0.4) | 552() | | 4,444 | |
| Ischemic stroke (wand w/o mention of cerebral infarction) | 4,899 (4.9%) | 1,140 (4.2%) | 2,000 (2.0%) | 271 (1.4%) | 9,999 (4.9%) | 385 (4.4%) | 16,898 (4.2%) | 1,996 (3.4%) | 0.04 |
| Hemorrhagic stroke; n (%) | 163 (0.2%) | 23 (0.1%) | 48 (0.0%) | 4 (0.0%) | | | | | |
| TIA; n (%) | 1,176 (1.2%) | 266 (1.0%) | 465 (0.5%) | 68 (0.4%) | 1,913 (0.9%) | 98 (0.7%) | 3,554 (0.9%) | 432 (0.7%) | 0.02 |
| Other cerebrovascular disease; n (%) | 1,704 (1.7%) | 322 (1.2%) | 670 (0.7%) | 86 (0.5%) | 3,962 (1.9%) | 236 (1.8%) | 6,336 (1.6%) | 644 (1.1%) | 0.04 |
| Late effects of cerebrovascular disease; n (%) | 1,554 (1.6%) | 233 (0.9%) | 423 (0.4%) | 34 (0.2%) | 3,186 (1.6%) | 107 (0.8%) | 5,163 (1.3%) | 374 (0.6%) | 0.07 |
| Cerebrovascular procedure; n (%)<br>Heart failure (CHF); n (%) | 70 (0.1%)<br>6,419 (6.4%) | 28 (0.1%)<br>1,435 (5.2%) | 15 (0.0%)<br>2,935 (3.0%) | 4 (0.0%)<br>399 (2.1%) | 18,631 (9.2%) | 951 (7.2%) | 27 005 /7 0%) | 2,785 (4.7%) | 0.10 |
| Heart failure (CHF); ft (76) | 6,419 (6.4%) | 1,453 (3.2%) | 2,933 (3.0%) | 399 (2.176) | 18,631 (9.276) | 931 (7.2%) | 27,985 (7.0%) | 2,783 [4.776] | 0.10 |
| Peripheral Vascular Disease (PVD) or PVD Surgery v2; n (%) | 6,638 (6.6%) | 1,465 (5.3%) | 3,369 (3.4%) | 497 (2.6%) | 20,972 (10.3%) | 1,195 (9.1%) | 30,979 (7.7%) | 3,157 (5.3%) | 0.10 |
| Atrial fibrillation; n (%) | 5,807 (5.8%) | 1,313 (4.8%) | 3,583 (3.6%) | 474 (2.5%) | 20,723 (10.2%) | 1,268 (9.6%) | 30,113 (7.5%) | 3,055 (5.1%) | 0.10 |
| Other cardiac dysrhythmia; n (%) | 8,278 (8.3%) | 2,142 (7.8%) | 4,579 (4.7%) | 793 (4.2%) | 24,622 (12.1%) | 1,806 (13.7%) | 37,479 (9.3%) | 4,741 (8.0%) | 0.05 |
| Cardiac conduction disorders; n (%) | 2,246 (2.2%) | 580 (2.1%) | 1,171 (1.2%) | 192 (1.0%) | 6,903 (3.4%) | 459 (3.5%) | 10,320 (2.6%) | 1,231 (2.1%) | 0.03 |
| Other CVD; n (%) | 8,797 (8.8%) | 2,259 (8.2%) | 5,483 (5.6%) | 817 (4.3%) | 25,637 (12.6%) | 1,671 (12.7%) | 39,917 (9.9%) | 4,747 (8.0%) | 0.07 |
| Diabetes-related complications | p to -== | | | | | | | !* ' | |
| Diabetic retinopathy; n (%) | 6,367 (6.4%) | 2,196 (8.0%) | 3,371 (3.4%) | 764 (4.0%) | 14,304 (7.0%) | 1,298 (9.9%) | 24,042 (6.0%) | 4,258 (7.2%) | -0.05 |
| Diabetes with other ophthalmic manifestations; n (%) | 904 (0.9%) | 230 (0.8%) | 1,868 (1.9%) | 305 (1.6%) | 4,906 (2.4%) | 267 (2.0%) | 7,678 (1.9%) | 802 (1.3%) | 0.05 |
| Retinal detachment, vitreous hemorrhage, vitrectomy; n (7 | 415 (0.4%) | 135 (0.5%) | 328 (0.3%) | 76 (0.4%) | 780 (0.4%) | 80 (0.6%) | 1,523 (0.4%) | 291 (0.5%) | -0.01 |
| Retinal laser coagulation therapy; n (%) | 560 (0.6%) | 158 (0.6%) | 504 (0.5%) | 115 (0.6%) | 1,220 (0.6%) | 74 (0.6%) | 2,284 (0.6%) | 347 (0.6%) | 0.00 |
| Occurrence of Diabetic Neuropathy v2 Copy; n (%) | 19,198 (19.2%) | 5,771 (21.1%) | 10,496 (10.7%) | 2,631 (13.9%) | 39,771 (19.6%) | 3,284 (25.0%) | 69,465 (17.3%) | 11,686 (19.7%) | -0.06 |

| Occurrence of diabetic nephropathy V3 with ICD10 Copy; r | 15,429 (15.4%) | 3,259 (11.9%) | 6,218 (6.3%) | 1,309 (6.9%) | 22,695 (11.2%) | 1,478 (11.2%) | 44,342 (11.0%) | 6,046 (10.2%) | 0.03 |
|---|---|---|---|---|---|---|---|---|---|
| Hypoglycemia v2; n (%) | 1,757 (1.8%) | 141 (0.5%) | 1,705 (1.7%) | 183 (1.0%) | 4,423 (2.2%) | 107 (0.8%) | 7,885 (2.0%) | 431 (0.7%) | 0.11 |
| Hyperglycemia; n (%) | 4,186 (4.2%) | 1,098 (4.0%) | 3,136 (3.2%) | 518 (2.7%) | 8,064 (4.0%) | 466 (3.5%) | 15,386 (3.8%) | 2,082 (3.5%) | 0.02 |
| 11 01 - 17 | | | | | | | | | |
| Disorders of fluid electrolyte and acid-base balance; n (%) | 6,080 (6.1%) | 1,099 (4.0%) | 3,203 (3.3%) | 434 (2.3%) | 12,731 (6.3%) | 479 (3.6%) | 22,014 (5.5%) | 2,012 (3.4%) | 0.10 |
| Diabetic ketoacidosis: n (%) | 385 (0.4%) | 76 (0.3%) | 309 (0.3%) | 47 (0.2%) | 668 (0.3%) | 22 (0.2%) | 1,362 (0.3%) | 145 (0.2%) | 0.02 |
| | | | | | | | 4 | | |
| Hyperosmolar hyperglycemic nonketotic syndrome (HONK | 589 (0.6%) | 166 (0.6%) | 468 (0.5%) | 92 (0.5%) | 1,077 (0.5%) | 80 (0.6%) | 2,134 (0.5%) | 338 (0.6%) | -0.01 |
| · | () | | 100 | 55 (5.5.4) | 2,011 (0.014) | | -,, | | |
| Diabetes with peripheral circulatory disorders with ICD-10 | 7,150 (7.2%) | 1,909 (7.0%) | 2,798 (2.8%) | 630 (3.3%) | 15,464 (7.6%) | 1,122 (8.5%) | 25,412 (6.3%) | 3,661 (6.2%) | 0.00 |
| Diabetic Foot; n (%) | 1,967 (2.0%) | 591 (2.2%) | 1,422 (1.4%) | 320 (1.7%) | 4,932 (2.4%) | 286 (2.2%) | 8,321 (2.1%) | 1,197 (2.0%) | 0.01 |
| | | | - 1 | · · · | | | | | 0.00 |
| Gangrenev2; n (%) | 235 (0.2%) | 63 (0.2%) | 144 (0.1%) | 28 (0.1%) | 380 (0.2%) | 33 (0.3%) | 759 (0.2%) | 124 (0.2%) | |
| Lower extremity amputation; n (%) | 644 (0.6%) | 207 (0.8%) | 256 (0.3%) | 66 (0.3%) | 1,155 (0.6%) | 81 (0.6%) | 2,055 (0.5%) | 354 (0.6%) | -0.01 |
| Osteomyelitis; n (%) | 491 (0.5%) | 155 (0.6%) | 361 (0.4%) | 78 (0.4%) | 936 (0.5%) | 34 (0.4%) | 1,788 (0.4%) | 287 (0.5%) | -0.01 |
| Skin infections v2; n (%) | 4,914 (4.9%) | 1,384 (5.1%) | 4,428 (4.5%) | 886 (4.7%) | 11,729 (5.8%) | 781 (5.9%) | 21,071 (5.2%) | 3,051 (5.1%) | 0.00 |
| Erectile dysfunction; n (%) | 2,938 (2.9%) | 1,188 (4.3%) | 2,680 (2.7%) | 585 (3.1%) | 4,367 (2.1%) | 501 (3.8%) | 9,985 (2.5%) | 2,274 (3.8%) | -0.07 |
| Diabetes with unspecified complication; n (%) | 5,922 (5.9%) | 1,946 (7.1%) | 4,818 (4.9%) | 1,306 (6.9%) | 11,396 (5.6%) | 953 (7.2%) | 22,136 (5.5%) | 4,205 (7.1%) | -0.07 |
| Diabetes mellitus without mention of complications; n (%) | 82,871 (83.0%) | 21,178 (77.3%) | 86,660 (88.1%) | 15,269 (80.7%) | 184,478 (90.7%) | 11,109 (84.4%) | 354,009 (88.2%) | 47,556 (80.0%) | 0.23 |
| Hypertension: 1 inpatient or 2 outpatient claims within 36 | 84,740 (84.8%) | 23,304 (85.1%) | 75,314 (76.6%) | 14,637 (77.4%) | 185,875 (91.4%) | 11,981 (91.1%) | 345,929 (86.2%) | 49,922 (84.0%) | 0.06 |
| Hyperlipidemia v2; n (%) | 70,468 (70.5%) | 19,569 (71.4%) | 65,929 (67.0%) | 13,478 (71.3%) | 154,166 (75.8%) | 10,169 (77.3%) | 290,563 (72.4%) | 43,216 (72.7%) | -0.01 |
| Edema; n (%) | 5,273 (5.3%) | 1,202 (4.4%) | 2,878 (2.9%) | 467 (2.5%) | 16,056 (7.9%) | 876 (6.7%) | 24,207 (6.0%) | 2,545 (4.3%) | 0.08 |
| Renal Dysfunction (non-diabetic) v2; n (%) | 19,382 (19.6%) | 3,179 (11.6%) | 8,494 (8.6%) | 958 (5.1%) | 42,497 (20.9%) | 1,822 (13.8%) | 70,573 (17.6%) | 5,959 (10.0%) | 0.22 |
| Occurrence of acute renal disease v2; n (%) | 2,581 (2.6%) | 332 (1.2%) | 1,243 (1.3%) | 80 (0.4%) | 5.423 (2.7%) | 130 (1.0%) | 9.247 (2.3%) | 542 (0.9%) | 0.11 |
| | | | | | -, | | -, | | |
| Occurrence of chronic renal insufficiency; n (%) | 16,369 (16.4%) | 2,354 (8.6%) | 6,265 (6.4%) | 657 (3.5%) | 36,061 (17.7%) | 1,453 (11.0%) | 58,695 (14.6%) | 4,464 (7.5%) | 0.23 |
| Chronic kidney disease v2; n (%) | 15,864 (15.9%) | 2,270 (8.3%) | 5,871 (6.0%) | 615 (3.3%) | 34,532 (17.0%) | 1,391 (10.6%) | 56,267 (14.0%) | 4,276 (7.2%) | 0.22 |
| CKD Stage 3-4; n (%) | 10,687 (10.7%) | 1,245 (4.5%) | 3,761 (3.8%) | 303 (1.6%) | 24,060 (11.8%) | 839 (6.4%) | 38,508 (9.6%) | 2,387 (4.0%) | 0.22 |
| Occurrence of hypertensive nephropathy; n (%) | 6,766 (6.8%) | 968 (3.5%) | 2,293 (2.3%) | 229 (1.2%) | 13,584 (6.7%) | 526 (4.0%) | 22,643 (5.6%) | 1,723 (2.9%) | 0.13 |
| Occurrence of miscellaneous renal insufficiency v2; n (%) | 4,400 (4.4%) | 874 (3.2%) | 2,417 (2.5%) | 271 (1.4%) | 11,162 (5.5%) | 523 (4.0%) | 17,979 (4.5%) | 1,668 (2.8%) | 0.09 |
| Glaucoma or cataracts v2; n (%) | 18,320 (18.3%) | 4,419 (16.1%) | 12,973 (13.2%) | 2,270 (12.0%) | 54,403 (26.8%) | 3,639 (27.7%) | 85,696 (21.3%) | 10,328 (17.4%) | 0.10 |
| Cellulitis or abscess of toe; n (%) | 1,284 (1.3%) | 391 (1.4%) | 849 (0.9%) | 225 (1.2%) | 2,592 (1.3%) | 237 (1.8%) | 4,725 (1.2%) | 853 (1.4%) | -0.02 |
| Footuicer; n (%) | 1,877 (1.9%) | 539 (2.0%) | 1,377 (1.4%) | 296 (1.6%) | 4.802 (2.4%) | 270 (2.1%) | 8.056 (2.0%) | 1,105 (1.9%) | 0.01 |
| Bladder stones; n (%) | 125 (0.1%) | 27 (0.1%) | 71 (0.1%) | 11 (0.1%) | 307 (0.2%) | 17 (0.1%) | 503 (0.1%) | 55 (0.1%) | 0.00 |
| Kidneystones; n (%) | 1,974 (2.0%) | 533 (1.9%) | 1,775 (1.8%) | 310 (1.6%) | 4,540 (2.2%) | 294 (2.2%) | 8,289 (2.1%) | 1,137 (1.9%) | 0.01 |
| 1 | | | | | | | | | |
| Urinary tract infections (UTIs); n (%) | 7,752 (7.8%) | 1,339 (4.9%) | 4,684 (4.8%) | 565 (3.0%) | 23,016 (11.3%) | 885 (6.7%) | 35,452 (8.8%) | 2,789 (4.7%) | 0.16 |
| Dipstick urinelysis; n (%) | 34,548 (34.6%) | 8,269 (30.2%) | 29,300 (29.8%) | 5,259 (27.8%) | 76,034 (37.4%) | 4,496 (34.2%) | 139,882 (34.8%) | 18,024 (30.3%) | 0.10 |
| Non-dipstick urinalysis; n (%) | 43,363 (43.4%) | 12,648 (46.2%) | 36,411 (37.0%) | 8,432 (44.6%) | 84,136 (41.4%) | 6,319 (48.0%) | 163,910 (40.8%) | 27,399 (46.1%) | -0.11 |
| Urine function test; n (%) | 1,897 (1.9%) | 418 (1.5%) | 1,625 (1.7%) | 200 (1.1%) | 6,250 (3.1%) | 434 (3.3%) | 9,772 (2.4%) | 1,052 (1.8%) | 0.04 |
| Cytology; n (%) | 360 (0.6%) | 117 (0.4%) | 522 (0.5%) | 60 (0.3%) | 1,497 (0.7%) | 67 (0.5%) | 2,579 (0.6%) | 244 (0.4%) | 0.03 |
| Cystoscopy; n (%) | 843 (0.8%) | 204 (0.7%) | 726 (0.7%) | 103 (0.5%) | 2,199 (1.1%) | 129 (1.0%) | 3,768 (0.9%) | 436 (0.7%) | 0.02 |
| Other Covariates | 1 | 1 | 1 | 1 | | | | ( ) | |
| Liver disease; n (%) | 3,416 (3.4%) | 1,355 (4.9%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 3,416 (0.9%) | 1,355 (2.3%) | -0.11 |
| Osteoarthritis; n (%) | 14,159 (14.2%) | 3,503 (12.8%) | 8,944 (9.1%) | 1,459 (7.7%) | 41,716 (20.5%) | 2,523 (19.2%) | 64,819 (16.1%) | 7,485 (12.6%) | 0.10 |
| Carcara tra rea, in proj | 24,255 (24.274) | 3,505 (12.074) | 0,544 (5.254) | 2,455 (1.114) | 42,720 (20.579) | 2,23(23,23) | 04,025 (20.254) | 7,405 (12.074) | 0.20 |
| Other arthritis, arthropathies and musculoskeletal pain; n | 33,077 (33.1%) | 8,620 (31.5%) | 26,598 (27.0%) | 4,912 (26.0%) | 82,377 (40.5%) | 4,956 (37.7%) | 142,052 (35.4%) | 18,488 (31.1%) | 0.09 |
| Dorsopathies; n (%) | 20,631 (20.7%) | 3,739 (21.0%) | 15,907 (16.2%) | 3,084 (16.3%) | 48,687 (23.9%) | 3,203 (24.3%) | 85,225 (21.2%) | 12,046 (20.3%) | 0.02 |
| Fractures; n (%) | 2,412 (2.4%) | 501 (1.8%) | 1,716 (1.7%) | 279 (1.5%) | 6,339 (3.1%) | 342 (2.6%) | 10,467 (2.6%) | 1,122 (1.9%) | 0.05 |
| Fallsv2; n (%) | 3,187 (3.2%) | 522 (1.9%) | 965 (1.0%) | 123 (0.7%) | 7,872 (3.9%) | 346 (2.6%) | 12,024 (3.0%) | 991 (1.7%) | 0.09 |
| Osteoporosis; n (%) | 4,316 (4.3%) | 634 (2.3%) | 1,543 (1.6%) | 149 (0.8%) | 15,070 (7.4%) | 631 (4.8%) | 20,929 (5.2%) | 1,414 (2.4%) | 0.15 |
| Hyperthyroidism; n (%) | 588 (0.6%) | 179 (0.7%) | 466 (0.5%) | 85 (0.4%) | 1,690 (0.8%) | 99 (0.8%) | 2,744 (0.7%) | 363 (0.6%) | 0.01 |
| Hypothyroidism v2; n (%) | 13,829 (13.8%) | 3,532 (12.9%) | 10,304 (10.5%) | 2,178 (11.5%) | 21,523 (10.6%) | 946 (7.2%) | 45,656 (11.4%) | 6,636 (11.2%) | 0.01 |
| Other disorders of thyroid gland V2; n (%) | 3,455 (3.5%) | 1,215 (4.4%) | 2,934 (3.0%) | 902 (4.8%) | 7,712 (3.8%) | 667 (5.1%) | 14,101 (3.5%) | 2,784 (4.7%) | -0.06 |
| Depression; n (%) | 7,320 (7.3%) | 1,821 (6.6%) | 5,335 (5.4%) | 914 (4.8%) | 17,919 (8.8%) | 902 (6.9%) | 30,574 (7.6%) | 3,637 (6.1%) | 0.06 |
| Anxiety; n (%) | 7,953 (8.0%) | 2,396 (8.7%) | 5,309 (5.4%) | 1,125 (5.9%) | 15,687 (7.7%) | 995 (7.6%) | 28,949 (7.2%) | 4,516 (7.6%) | -0.02 |
| Sleep Disorder; n (%) | 3,987 (4.0%) | 673 (2.5%) | 5,785 (5.9%) | 766 (4.1%) | 11,002 (5.4%) | 418 (3.2%) | 20,774 (5.2%) | 1,857 (3.1%) | 0.11 |
| Dementia: n (%) | 3,796 (3.8%) | 361 (1.3%) | 1,343 (1.4%) | 91 (0.5%) | 14,445 (7.1%) | 369 (2.8%) | 19,584 (4.9%) | 821 (1.4%) | 0.11 |
| - 17 | | | | | | ١ ، | | \ \ / | 0.20 |
| Delirium; n (%) | 1,038 (1.0%) | 110 (0.4%) | 410 (0.4%) | 31 (0.2%) | 2,997 (1.5%) | 80 (0.6%) | 4,445 (1.1%) | 221 (0.4%) | |
| Psychosis; n (%) | 1,115 (1.1%) | 171 (0.6%) | 403 (0.4%) | 36 (0.2%) | 3,561 (1.8%) | 67 (0.5%) | 5,079 (1.3%) | 274 (0.5%) | 0.08 |
| Obesity; n (%) | 17,344 (17.6%) | 7,711 (28.1%) | 6,568 (6.7%) | 1,684 (8.9%) | 10,068 (5.0%) | 806 (6.1%) | 34,180 (8.5%) | 10,201 (17.2%) | -0.26 |
| Overweight; n (%) | 7,117 (7.1%) | 2,123 (7.7%) | 3,068 (3.1%) | 700 (3.7%) | 8,443 (4.2%) | 650 (4.9%) | 18,628 (4.6%) | 3,473 (5.8%) | -0.05 |
| Smoking; n (%) | 10,562 (10.6%) | 3,243 (11.8%) | 4,864 (4.9%) | 882 (4.7%) | 21,088 (10.4%) | 1,434 (10.9%) | 36,514 (9.1%) | 5,559 (9.3%) | -0.01 |
| Alcohol abuse or dependence; n (%) | 683 (0.7%) | 199 (0.7%) | o (o.a%) | 0 (0.0%) | ò (0.0%) | ò (0.0%) | #VALUE! | 199 (0.3%) | #VALUE! |
| Drug abuse or dependence; n (%) | 1,133 (1.1%) | 359 (1.3%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 1,133 (0.3%) | 359 (0.6%) | -0.04 |
| COPD; n (%) | 6,952 (7.0%) | 1,485 (5.4%) | 3,056 (3.1%) | 386 (2.0%) | 17,808 (8.8%) | 895 (6.8%) | 27,816 (6.9%) | 2,766 (4.7%) | 0.09 |
| | -,(-,) | -, () | -,() | | | | | | |

| Asthma; n (%) | 4,622 (4.6%) | 1,225 (4.5%) | 3,363 (3.4%) | 592 (3.1%) | 9,980 (4.9%) | 656 (5.0%) | 17,965 (4.5%) | 2,473 (4.2%) | 0.01 |
|---|---|---|---|---|---|---|---|---|---|
| Obstructive sleep apnes; n (%) | 7,880 (7.9%) | 3,326 (12.1%) | 7,903 (8.0%) | 2,046 (10.8%) | 10,766 (5.3%) | 1,274 (9.7%) | 26,549 (6.6%) | 6,646 (11.2%) | -0.16 |
| Pneumonia; n (%) | 1,745 (1.7%) | 319 (1.2%) | 1,136 (1.2%) | 158 (0.8%) | 4,422 (2.2%) | 214 (1.6%) | 7,303 (1.8%) | 691 (1.2%) | 0.05 |
| Imaging; n (%) | 73 (0.1%) | 17 (0.1%) | 17 (0.0%) | 4 (0.0%) | | ** | | | •• |
| Diabetes Medications | | | | | | | | | |
| DM Medications - AGIs; n (%) | 499 (0.5%) | 97 (0.4%) | 310 (0.3%) | 64 (0.3%) | 1,243 (0.6%) | 58 (0.4%) | 2,052 (0.5%) | 219 (0.4%) | 0.01 |
| DM Medications - Glitazones; n (%) | 7,594 (7.6%) | 2,318 (8.5%) | 6,881 (7.0%) | 1,520 (8.0%) | 14,722 (7.2%) | 1,253 (9.5%) | 29,197 (7.3%) | 5,091 (8.6%) | -0.05 |
| DM Medications - GLP-1 RA; n (%) | 4,184 (4.2%) | 5,850 (21.4%) | 4,354 (4.4%) | 4,829 (25.5%) | 5,290 (2.6%) | 2,529 (19.2%) | 13,828 (3.4%) | 13,208 (22.2%) | -0.59 |
| DM Medications - Insulin; n (%) | 17,835 (17.9%) | 7,838 (28.6%) | 14,817 (15.1%) | 5,867 (31.0%) | 39,115 (19.2%) | 4,548 (34.6%) | 71,767 (17.9%) | 18,253 (30.7%) | -0.30 |
| DM Medications - Meglitinides; n (%) | 1,041 (1.0%) | 212 (0.8%) | 1,089 (1.1%) | 171 (0.9%) | 3,580 (1.8%) | 247 (1.9%) | 5,710 (1.4%) | 630 (1.1%) | 0.03 |
| DM Medications - Metformin; n (%) | 74,681 (74.8%) | 20,362 (74.3%) | 79,574 (80.9%) | 14,355 (75.9%) | 142,034 (69.9%) | 9,591 (72.9%) | 296,289 (73.8%) | 44,308 (74.5%) | -0.02 |
| Concomitant initiation or current use of 2nd Generation S | 33,222 (33.3%) | 7,632 (27.9%) | 29,037 (29.5%) | 4,720 (25.0%) | 73,210 (36.0%) | 4,236 (32.2%) | 135,469 (33.7%) | 16,588 (27.9%) | 0.13 |
| Concomitant initiation or current use of AGIs; n (%) | 359 (0.4%) | 65 (0.2%) | 216 (0.2%) | 39 (0.2%) | 888 (0.4%) | 35 (0.3%) | 1,463 (0.4%) | 139 (0.2%) | 0.04 |
| Concomitant initiation or current use of Glitazones; n (%) | 6,052 (6.1%) | 1,790 (6.5%) | 5,547 (5.6%) | 1,221 (6.5%) | 11,634 (5.7%) | 990 (7.5%) | 23,233 (5.8%) | 4,001 (6.7%) | -0.04 |
| Concomitant initiation or current use of GLP-1 RA; n (%) | 2,392 (2.4%) | 4,382 (16.0%) | 2,527 (2.6%) | 3,730 (19.7%) | 2,849 (1.4%) | 1,906 (14.5%) | 7,768 (1.9%) | 10,018 (16.8%) | -0.53 |
| Concomitant initiation or current use of Insulin; n (%) | 13,381 (13.4%) | 5,986 (21.9%) | 11,021 (11.2%) | 4,466 (23.6%) | 29,957 (14.7%) | 3,603 (27.4%) | 54,359 (13.5%) | 14,055 (23.6%) | -0.26 |
| Concomitant initiation or current use of Meglitinides; n (% | 773 (0.8%) | 145 (0.5%) | 768 (0.8%) | 117 (0.6%) | 2,607 (1.3%) | 170 (1.3%) | 4,148 (1.0%) | 432 (0.7%) | 0.03 |
| Concomitant initiation or current use of Metformin; n (%) | 64,669 (64.7%) | 16,361 (60.3%) | 70,407 (71.6%) | 11,825 (62.5%) | 122,594 (60.3%) | 8,039 (61.1%) | 257,670 (64.2%) | 36,425 (61.3%) | 0.06 |
| Past use of 2nd Generation SUs Copy; n (%) | 7,266 (7.3%) | 2,028 (7.4%) | 6,956 (7.1%) | 1,253 (6.6%) | 14,813 (7.3%) | 902 (6.9%) | 29,035 (7.2%) | 4,183 (7.0%) | 0.01 |
| Past use of AGIs Copy; n (%) | 140 (0.1%) | 32 (0.1%) | 94 (0.1%) | 25 (0.1%) | 355 (0.2%) | 23 (0.2%) | 589 (0.1%) | 80 (0.1%) | 0.00 |
| Past use of Glitazones Copy; n (%) | 1,542 (1.5%) | 528 (1.9%) | 1,334 (1.4%) | 299 (1.6%) | 3,088 (1.5%) | 263 (2.0%) | 5,964 (1.5%) | 1,090 (1.8%) | -0.02 |
| Past use of GLP-1 RA Copy; n (%) | 1,977 (2.0%) | 1,701 (6.2%) | 2,007 (2.0%) | 1,253 (6.6%) | 2,441 (1.2%) | 623 (4.7%) | 6,425 (1.6%) | 3,577 (6.0%) | -0.23 |
| | | | | | | | | | -0.12 |
| Past use of Insulin Copy; n (%) | 4,434 (4.5%) | 1,852 (6.8%) | 3,797 (3.9%) | 1,401 (7.4%) | 9,160 (4.5%) | 945 (7.2%) | 17,411 (4.3%) | 4,198 (7.1%) | |
| Past use of Meglitinides Copy; n (%) | 268 (0.3%) | 67 (0.2%) | 321 (0.3%) | 54 (0.3%) | 973 (0.5%) | 77 (0.6%) | 1,562 (0.4%) | 198 (0.3%) | 0.02 |
| Past use of metformin (final) Copy; n (%) | 10,012 (10.0%) | 3,801 (13.9%) | 9,167 (9.3%) | 2,530 (13.4%) | 19,440 (9.6%) | 1,552 (11.8%) | 38,619 (9.6%) | 7,883 (13.3%) | -0.12 |
| Other Medications | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 52,616 (52.7%) | 14,800 (54.0%) | 52,849 (53.7%) | 10,492 (55.5%) | 96,076 (47.3%) | 6,205 (47.2%) | 201,541 (50.2%) | 31,497 (53.0%) | -0.06 |
| Use of ARBs; n (%) | 33,459 (33.5%) | 9,268 (33.8%) | 32,714 (33.3%) | 6,489 (34.3%) | 69,748 (34.3%) | 4,833 (36.7%) | 135,921 (33.8%) | 20,590 (34.6%) | -0.02 |
| Use of Loop Diuretics - United; n (%) | 10,502 (10.5%) | 2,316 (8.5%) | 6,912 (7.0%) | 1,075 (5.7%) | 33,131 (16.3%) | 1,744 (13.3%) | 30,343 (12.6%) | 5,135 (8.6%) | 0.13 |
| Use of other diuretics- United; n (%) | 2,623 (2.6%) | 833 (3.0%) | 2,133 (2.2%) | 453 (2.4%) | 6,785 (3.3%) | 483 (3.7%) | 11,541 (2.9%) | 1,769 (3.0%) | -0.01 |
| Use of nitrates-United; n (%) | 4,760 (4.8%) | 1,425 (5.2%) | 3,232 (3.3%) | 624 (3.3%) | 14,468 (7.1%) | 976 (7.4%) | 22,460 (5.6%) | 3,025 (5.1%) | 0.02 |
| Use of other hypertension drugs; n (%) | 6,251 (6.3%) | 1,267 (4.6%) | 4,430 (4.5%) | 643 (3.4%) | 15,746 (7.7%) | 809 (6.1%) | 26,447 (6.6%) | 2,719 (4.6%) | 0.09 |
| Use of digoxin-United; n (%) | 1,351 (1.4%) | 278 (1.0%) | 1,001 (1.0%) | 112 (0.6%) | 5,685 (2.8%) | 306 (2.3%) | 8,037 (2.0%) | 696 (1.2%) | 0.06 |
| | 1,058 (1.1%) | 283 (1.0%) | 807 (0.8%) | 143 (0.8%) | 3,770 (1.9%) | 218 (1.7%) | 5,635 (1.4%) | 644 (1.1%) | 0.03 |
| Use of Anti-errhythmics; n (%) | | , , | | , , | | | | , , | |
| Use of COPD/asthma meds- United; n (%) | 14,067 (14.1%) | 3,637 (13.3%) | 12,756 (13.0%) | 2,412 (12.8%) | 32,384 (15.9%) | 2,112 (16.1%) | 59,207 (14.7%) | 8,161 (13.7%) | 0.03 |
| Use of statins; n (%) | 71,183 (71.3%) | 20,272 (74.0%) | 65,053 (66.1%) | 13,377 (70.7%) | 148,529 (73.1%) | 10,331 (78.5%) | 284,765 (70.9%) | 43,980 (74.0%) | -0.07 |
| Use of other lipid-lowering drugs; n (%) | 11,144 (11.2%) | 3,351 (12.2%) | 12,301 (12.5%) | 2,743 (14.5%) | 24,891 (12.2%) | 1,915 (14.6%) | 48,336 (12.0%) | 8,009 (13.5%) | -0.04 |
| Use of antiplatelet agents; n (%) | 12,026 (12.0%) | 3,756 (13.7%) | 10,435 (10.6%) | 2,047 (10.8%) | 30,403 (15.0%) | 2,275 (17.3%) | 52,864 (13.2%) | 8,078 (13.6%) | -0.01 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban, Apixal | 5,155 (5.2%) | 1,283 (4.7%) | 3,619 (3.7%) | 581 (3.1%) | 17,505 (8.6%) | 1,132 (8.6%) | 26,279 (6.5%) | 2,996 (5.0%) | 0.06 |
| Use of heparin and other low-molecular weight heparins; n | 198 (0.2%) | 43 (0.2%) | 9 (0.0%) | 1 (0.0%) | 420 (0.2%) | 21 (0.2%) | 627 (0.2%) | 065 (0.1%) | 0.03 |
| Use of NSAIDs; n (%) | 16,220 (16.2%) | 4,317 (16.5%) | 16,087 (16.4%) | 3,178 (16.8%) | 32,311 (15.9%) | 1,975 (15.0%) | 64,618 (16.1%) | 9,670 (16.3%) | -0.01 |
| Use of oral corticosteroids; n (%) | 10,445 (10.5%) | 2,832 (10.3%) | 9,420 (9.6%) | 1,722 (9.1%) | 23,684 (11.7%) | 1,501 (11.4%) | 43,549 (10.8%) | 6,055 (10.2%) | 0.02 |
| Use of bisphosphonate (United); n (%) | 2,212 (2.2%) | 322 (1.2%) | 803 (0.8%) | 70 (0.4%) | 6,829 (3.4%) | 252 (1.9%) | 9,844 (2.5%) | 644 (1.1%) | 0.11 |
| Use of opioids-United; n (%) | 20,346 (20.4%) | 5,472 (20.0%) | 18,620 (18.9%) | 3,581 (18.9%) | 42,529 (20.9%) | 2,588 (19.7%) | 81,495 (20.3%) | 11,641 (19.6%) | 0.02 |
| Use of antidepressants; n (%) | 22,602 (22.6%) | 6,573 (24.0%) | 19,480 (19.8%) | 4,303 (22.8%) | 48,867 (24.0%) | 3,160 (24.0%) | 90,949 (22.6%) | 14,036 (23.6%) | -0.02 |
| Use of antipsychotics; n (%) | 2,384 (2.6%) | 556 (2.0%) | 1,381 (1.4%) | 263 (1.4%) | 6,338 (3.1%) | 258 (2.0%) | 10,303 (2.6%) | 1,077 (1.8%) | 0.05 |
| Use of anticonvulsants; n (%) | 16,330 (16.3%) | 4,552 (16.6%) | 10,690 (10.9%) | 2,193 (11.6%) | 34,272 (16.9%) | 2,157 (16.4%) | 61,292 (15.3%) | 8,902 (15.0%) | 0.01 |
| | | | | | 34,272 (10.376) | 2,137 (10.4/6) | 01,252 (13.3/6) | 0,502 (15.076) | 0.01 |
| Use of lithium-United; n (%) | 147 (0.1%) | 39 (0.1%) | 115 (0.1%) | 29 (0.2%) | | 4 222 (2 25) | an entre de afri | | |
| Use of Benzos-United; n (%) | 9,376 (9.4%) | 2,472 (9.0%) | 7,846 (8.0%) | 1,587 (8.4%) | 21,369 (10.5%) | 1,277 (9.7%) | 38,591 (9.6%) | 5,336 (9.0%) | 0.02 |
| Use of anxiolytics/hypnotics-United; n (%) | 4,899 (4.9%) | 1,421 (5.2%) | 5,117 (5.2%) | 1,058 (5.6%) | 10,049 (4.9%) | 683 (5.2%) | 20,065 (5.0%) | 3,162 (5.3%) | -0.01 |
| Use of dementia meds-United; n (%) | 2,332 (2.3%) | 208 (0.8%) | 1,003 (1.0%) | 51 (0.3%) | 10,424 (5.1%) | 272 (2.1%) | 13,759 (3.4%) | 531 (0.9%) | 0.17 |
| Use of antiparkinsonian meds- United; n (%) | 2,112 (2.1%) | 562 (2.1%) | 1,514 (1.5%) | 265 (1.4%) | 6,081 (3.0%) | 335 (2.5%) | 9,707 (2.4%) | 1,162 (2.0%) | 0.03 |
| Any use of pramtintide; n (%) | 2 (0.0%) | 9 (0.0%) | 9 (0.0%) | 23 (0.1%) | | | | | ** |
| Any use of 1st generation sulfonyluress; n (%) | 2 (0.0%) | 1 (0.0%) | 10 (0.0%) | 1 (0.0%) | | | | | ** |
| Entresto (sacubitril/valsartan); n (%) | 158 (0.2%) | 122 (0.4%) | 52 (0.1%) | 22 (0.1%) | 158 (0.1%) | 43 (0.3%) | 368 (0.1%) | 187 (0.3%) | 0.00 |
| Initiation as monotherapy v4 Copy; n (%) | 85,916 (86.0%) | 25,773 (94.1%) | 84,176 (85.6%) | 17,936 (94.8%) | 184,924 (91.0%) | 12,565 (95.5%) | 355,016 (88.4%) | 36,274 (94.6%) | -0.22 |
| Labs | | | | | ( | | 198,248 | 46,306 | |
| Lab values- HbA1c (%) v3; n (%) | 43,141 (43.2%) | 11,298 (41.2%) | 6,423 (6.5%) | 1,049 (5.5%) | N/A | N/A | 49,564 (25.0%) | 12,347 (26.7%) | -0.04 |
| Lab values- HbA1c (%) (within 3 months) v3; n (%) | 34,616 (34.6%) | 9,068 (33.1%) | 5,174 (5.3%) | 858 (4.5%) | N/A | N/A | 39,790 (20.1%) | 9,926 (21.4%) | -0.03 |
| | 21,020 (34.079) | 2,000 (23.279) | 2,2.4 (3.3%) | 536 [4.576] | II/A | Total Control | 25,150 [20.270] | 2,220 (22.470) | 0.03 |

| Lab values- HbA1c (%) (within 6 months) v3; n (%) | 43,141 (43.2%) | 11,298 (41.2%) | 6,423 (6.5%) | 1,049 (5.5%) | N/A | N/A | 49,564 (25.0%) | 12,347 (26.7%) | -0.04 |
|---|---|---|---|---|---|---|---|---|---|
| Lab values- BNP; n (%) | 749 (0.7%) | 156 (0.6%) | 74 (0.1%) | 5 (0.0%) | N/A | N/A | 823 (0.4%) | 161 (0.3%) | 0.02 |
| | | | | | N/A | N/A | | | 0.02 |
| Lab values- BNP (within 3 months); n (%) | 463 (0.5%) | 98 (0.4%) | 53 (0.1%) | 1 (0.0%) | | | 516 (0.3%) | 099 (0.2%) | |
| Lab values- BNP (within 6 months); n (%) | 749 (0.7%) | 156 (0.6%) | 74 (0.1%) | 5 (0.0%) | N/A | N/A | 823 (0.4%) | 161 (0.3%) | 0.02 |
| Lab values- BUN (mg/di); n (%) | 42,226 (42.3%) | 10,947 (40.0%) | 6,201 (6.3%) | 967 (5.1%) | N/A | N/A | 48,427 (24.4%) | 11,914 (25.7%) | -0.03 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 33,174 (33.2%) | 8,603 (31.4%) | 4,838 (4.9%) | 783 (4.1%) | N/A | N/A | 38,012 (19.2%) | 9,386 (20.3%) | -0.03 |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 42,226 (42.3%) | 10,947 (40.0%) | 6,201 (6.3%) | 967 (5.1%) | N/A | N/A | 48,427 (24.4%) | 11,914 (25.7%) | -0.03 |
| Lab values- Creatinine (mg/dl) v2; n (%) | 43,684 (43.7%) | 11,561 (42.2%) | 6,653 (6.8%) | 1,095 (5.8%) | N/A | N/A | 50,337 (25.4%) | 12,656 (27.3%) | -0.04 |
| cab values ci dacinine (ing/ui) vz, ii (xi) | 43,004 (43.776) | 11,361 (42.276) | 0,033 (0.8/6) | 1,050 (5.6.4) | N/A | IV. | 30,337 (23.4/6) | 12,030 (27.376) | 0.04 |
| Lab values- Creatinine (mg/dl) (within 3 months) v2; n (%) | 34,353 (34.4%) | 9,066 (33.1%) | 5,215 (5.3%) | 882 (4.7%) | N/A | N/A | 39,568 (20.0%) | 9,948 (21.5%) | -0.04 |
| cab values a cacinine (ingrai) (waliin s monais) vz., n (x) | 34,333 (34.4/8) | 3,000 (33.1/0) | اورو دا درود | 002 (4.770) | nya. | IVA | 35,366 (20.0/9) | 3,340 [21.3/9] | 0.04 |
| to the second se | 42 424 (42 28) | 44 864 (45 881) | a con la obil | 4 000 (0 00) | | *** | | 42 525 (22.25) | |
| Lab values- Creatinine (mg/dl) (within 6 months) v2; n (%) | 43,684 (43.7%) | 11,561 (42.2%) | 6,653 (6.8%) | 1,095 (5.8%) | N/A | N/A | 50,337 (25.4%) | 12,656 (27.3%) | -0.04 |
| Lab values- HDL level (mg/dl); n (%) | 36,599 (36.6%) | 9,688 (35.4%) | 5,867 (6.0%) | 1,004 (5.3%) | N/A | N/A | 42,466 (21.4%) | 10,692 (23.1%) | -0.04 |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 27,311 (27.3%) | 7,215 (26.3%) | 4,458 (4.5%) | 768 (4.1%) | N/A | N/A | 31,769 (16.0%) | 7,983 (17.2%) | -0.03 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 36,599 (36.6%) | 9,688 (35.4%) | 5,867 (6.0%) | 1,004 (5.3%) | N/A | N/A | 42,466 (21.4%) | 10,692 (23.1%) | -0.04 |
| Lab values-LDL level (mg/dl) v2; n (%) | 37,864 (37.9%) | 10,005 (36.5%) | 6,037 (6.1%) | 991 (5.2%) | N/A | N/A | 43,901 (22.1%) | 10,996 (23.7%) | -0.04 |
| 107-17 | | | | | | | | | |
| Lab values- LDL level (mg/dl) (within 3 months) v2; n (%) | 28,216 (28.2%) | 7,452 (27.2%) | 4,563 (4.6%) | 765 (4.0%) | N/A | N/A | 32,779 (16.5%) | 8,217 (17.7%) | -0.03 |
| | ,, | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | 3,555 (3,554) | | - | | | -, () | |
| Lab values-LDL level (mg/dl) (within 6 months) v2; n (%) | 37,864 (37.9%) | 10,005 (36.5%) | 6,037 (6.1%) | 991 (5.2%) | N/A | N/A | 43,901 (22.1%) | 10,996 (23.7%) | -0.04 |
| | | | | | N/A | | | | 0.00 |
| Lab values- NT-proBNP; n (%) | 114 (0.1%) | 43 (0.2%) | 17 (0.0%) | 2 (0.0%) | | N/A | 131 (0.1%) | 45 (0.1%) | 0.00 |
| Lab values- NT-proBNP (within 3 months); n (%) | 66 (0.1%) | 27 (0.1%) | 12 (0.0%) | 2 (0.0%) | N/A | N/A | 78 (0.0%) | 29 (0.1%) | - |
| Lab values- NT-proBNP (within 6 months); n (%) | 114 (0.1%) | 43 (0.2%) | 17 (0.0%) | 2 (0.0%) | N/A | N/A | 131 (0.1%) | 45 (0.1%) | - |
| Lab values-Total cholesterol (mg/dl) v2; n (%) | 37,177 (37.2%) | 9,915 (36.2%) | 5,903 (6.0%) | 1,018 (5.4%) | N/A | N/A | 43,080 (21.7%) | 10,933 (23.6%) | -0.05 |
| (0) | | | | | | | | | |
| Lab values-Total cholesterol (mg/dl) (within 3 months) v2; | 27,768 (27.8%) | 7,384 (27.0%) | 4,489 (4.6%) | 783 (4.1%) | N/A | N/A | 32,257 (16.3%) | 8,167 (17.6%) | -0.03 |
| and the state of t | 27,700 (27.0.4) | ,,201,21101 | 4,100 [1.0.4] | 100 (1.004) | - | 141 | 32,237 (20.374) | 0,207 (27.074) | |
| Lab values-Total cholesterol (mg/dl) (within 6 months) v2; | 37,177 (37.2%) | 9,915 (36.2%) | 5,903 (6.0%) | 1,018 (5.4%) | N/A | N/A | 43,080 (21.7%) | 10,933 (23.6%) | -0.05 |
| | | | | | | - | | | -0.05 |
| Lab values-Triglyceride level (mg/dl); n (%) | 36,829 (36.9%) | 9,848 (35.9%) | 5,814 (5.9%) | 1,000 (5.3%) | N/A | N/A | 42,643 (21.5%) | 10,848 (23.4%) | -0.05 |
| Lab values-Triglyceride level (mg/dl) (within 3 months); n (: | 27,527 (27.6%) | 7,338 (26.8%) | 4,418 (4.5%) | 771 (4.1%) | N/A | N/A | 31,945 (16.1%) | 8,109 (17.5%) | -0.04 |
| Lab values-Triglyceride level (mg/dl) (within 6 months); n (: | 36,829 (36.9%) | 9,848 (35.9%) | 5,814 (5.9%) | 1,000 (5.3%) | N/A | N/A | 42,643 (21.5%) | 10,848 (23.4%) | -0.05 |
| Lab result number- HbA1c (%) mean (only 2 to 20 included) | 42,905 | 11,242 | 6,311 | 1,018 | N/A | N/A | 49,216 | 12,260 | |
| mean (sd) | 8.36 (1.78) | 8.55 (1.75) | 8.53 (1.88) | 8.32 (1.79) | N/A | N/A | 8.38 (1.79) | 8.53(1.75) | -0.08 |
| median (IQR) | 8.00 [7.15, 9.25] | 8.20 [7.30, 9.55] | 8.05 [7.15, 9.50] | 8.00 [7.00, 9.00] | N/A | N/A | 8.01 (1.79) | 8.18(1.75) | -0.10 |
| | | | | | N/A | N/A | | | 0.10 |
| Missing n (%) | 56,998 (57.1%) | 16,152 (59.0%) | 92,034 (93.6%) | 17,894 (94.6%) | | | 149,032 (75.2%) | 34,046 (73.5%) | 0.04 |
| Lab result number- BNP mean v2 | 749 | 156 | 74 | 3 | N/A | N/A | 823 | 161 | |
| mean (sd) | 154.93 (290.29) | 146.64 (514.40) | 3,931.76 (32,532.43) | 32.60 (34.74) | N/A | N/A | 494.52 (9710.65) | 143.10 (509.52) | 0.05 |
| median [IQR] | 65.20 [25.55, 167.50] | 34.45 [14.55, 89.70] | 76.50 [29.75, 193.00] | 18.00 [13.50, 59.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 99,154 (99.3%) | 27,238 (99.4%) | 98,271 (99.9%) | 18,907 (100.0%) | N/A | N/A | 197,425 (99.6%) | 46,145 (99.7%) | -0.02 |
| Lab result number- BUN (mg/di) mean v2 | 42,226 | 10.947 | 6.201 | 967 | N/A | N/A | 48.427 | 11 914 | |
| meen (sd) | 17.98 (7.45) | 16.64 (5.62) | 1,795.05 (17,168.60) | 2,184.17 (18,571.33) | N/A | N/A | 245.53 (6143.29) | 192.57 (5288.81) | 0.01 |
| | 16.50 [13.00, 21.00] | 16.00 [13.00, 19.50] | 16.00 [13.00, 20.00] | 15.50 [13.00, 19.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| median [IQR] | | | | | | | | | #VALUE: |
| Missing n (%) | 57,677 (57.7%) | 16,447 (60.0%) | 92,144 (93.7%) | 17,945 (94.9%) | N/A | N/A | 149,821 (75.6%) | 34,392 (74.3%) | 0.03 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 to 15 | 43,333 | 11,484 | 5,645 | 711 | N/A | N/A | 48,978 | 12,195 | |
| mean (sd) | 1.01 (0.39) | 0.92 (0.24) | 0.98 (0.33) | 0.94 (0.20) | N/A | N/A | 1.01 (0.38) | 0.92 (0.24) | 0.28 |
| median [IQR] | 0.93 [0.78, 1.15] | 0.89 [0.75, 1.05] | 0.95 [0.79, 1.08] | 0.95 [0.81, 1.00] | N/A | N/A | 0.93 (0.38) | 0.89 (0.24) | 0.13 |
| Missing; n (%) | 56,570 (56.6%) | 15,910 (58.1%) | 92,700 (94.3%) | 18,201 (96.2%) | N/A | N/A | 149,270 (75.3%) | 34,111 (73.7%) | 0.04 |
| <del></del> | | ,,, | | | - | | | | |
| Lab result number- HDL level (mg/dl) mean (only =5000 in | 36,599 | 9.688 | 5,805 | 994 | N/A | N/A | 42.404 | 10,682 | |
| | 45.86 (13.58) | 44.26 (12.89) | 44.94 (13.83) | 47.81 (132.54) | N/A | N/A | 45.73 (13.61) | 44.59 (42.24) | 0.04 |
| mean (sd) | , , | , , | , , | , , | | | , , | , , | |
| median [IQR] | 44.00 [37.00, 53.00] | 42.00 [36.00, 51.00] | 43.00 [36.00, 52.00] | 42.00 [35.00, 50.00] | N/A | N/A | 43.86 (13.61) | 42.00 (42.24) | 0.06 |
| Missing: n (%) | 63,304 (63.4%) | 17,706 (64.6%) | 92,540 (94.1%) | 17,918 (94.7%) | N/A | N/A | 155,844 (78.6%) | 35,624 (76.9%) | 0.04 |
| Lab result number-LDL level (mg/dl) mean (only =:5000 in | 36,994 | 9,856 | 5,343 | 919 | N/A | N/A | 42,337 | 10,775 | |
| mean (sd) | 85.89 (39.91) | 81.77 (40.57) | 90.89 (42.17) | 84.41 (40.86) | N/A | N/A | 86.52 (40.20) | 82.00 (40.60) | 0.11 |
| median (IQR) | 83.50 [62.00, 108.75] | 80.50 [58.00, 105.00] | 89.00 [67.00, 116.00] | 84.00 [61.00, 109.00] | N/A | N/A | 84.19 (40.20) | 80.80 (40.60) | 0.08 |
| Missing: n (%) | 62,909 (63.0%) | 17,538 (64.0%) | 93,002 (94.6%) | 17,993 (95.1%) | N/A | N/A | 155,911 (78.6%) | 35,531 (76.7%) | 0.05 |
| | UZ,303 (03.076) | 27,330 04,070 | 23,002 (34.0/0) | 27,333 [33.170] | N/A | N/A | 222,311 (70.0/6) | 22,331 [10.770] | 0.03 |
| International Principles of the International Control of the International | | | | | and a | *** | 42 982 | | |
| Lab result number-Total cholesterol (mg/dl) mean (only =< | 37,141 | 9,912 | 5,841 | 1,005 | N/A | N/A | | 10,917 | |
| mean (sd) | 173.84 (47.32) | 170.49 (47.05) | 179.36 (49.26) | 171.92 (49.48) | N/A | N/A | 174.59 (47.59) | 170.62 (47.28) | 0.08 |
| median (IQR) | 167.50 [143.00, 198.00] | 165.00 [139.00, 195.00] | 174.00 [148.00, 205.00] | 165.50 [140.25, 196.00] | N/A | N/A | 168.38 (47.59) | 165.05 (47.28) | 0.07 |
| Missing; n (%) | 62,762 (62.8%) | 17,482 (63.8%) | 92,504 (94.1%) | 17,907 (94.7%) | N/A | N/A | 155,266 (78.3%) | 35,389 (76.4%) | 0.05 |

| Lab result number-Triglyceride level (mg/dl) mean (only=c | | 9,846 | 5,753 | 987 | N/A | N/A | 42,578 | 10,833 | |
|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 193.49 (177.23) | 207.63 (200.82) | 197.08 (184.91) | 210.43 (212.46) | N/A | N/A | 193.98 (178.29) | 207.89 (201.92) | -0.07 |
| median (IQR) | 155.00 [110.00, 223.00] | 160.00 [113.00, 236.00] | 153.00 [106.50, 228.25] | 157.50 [109.00, 233.00] | N/A | N/A | 154.73 (178.29) | 159.77 (201.92) | -0.03 |
| Missing: n (%) | 63,078 (63.1%) | 17,548 (64.1%) | 92,592 (94.2%) | 17,925 (94.8%) | N/A | N/A | 155,670 (78.5%) | 35,473 (76.6%) | 0.05 |
| Lab result number- Hemoglobin mean (only >0 included) | 28,791 | 7,333 | 4,328 | 643 | N/A | N/A | 33,119 | 7,976 | |
| mean (sd) | 13.72 (1.56) | 14.15 (1.49) | 6,342.54 (215,464.58) | 1,919.68 (16,045.24) | N/A | N/A | 840.77 (77884.39) | 167.77 (4553.05) | 0.01 |
| median [IQR] | 13.70 [12.65, 14.80] | 14.10 [13.10, 15.20] | 13.90 [12.85, 15.00] | 14.00 [13.00, 15.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 71,112 (71.2%) | 20,061 (73.2%) | 94,017 (95.6%) | 18,269 (96.6%) | N/A | N/A | 165,129 (83.3%) | 38,330 (82.8%) | 0.01 |
| Lab result number- Serum sodium mean (only > 90 and < 15 | 42,353 | 11,249 | 6,243 | 1,027 | N/A | N/A | 48,596 | 12,276 | |
| mean (sd) | 139.42 (2.77) | 139.45 (2.68) | 138.82 (2.61) | 139.17 (2.53) | N/A | N/A | 139.34 (2.75) | 139.43 (2.67) | -0.03 |
| median [IQR] | 139.50 [138.00, 141.00] | 139.50 [138.00, 141.00] | 139.00 [137.00, 140.50] | 139.00 [137.50, 141.00] | N/A | N/A | 139.44 (2.75) | 139.46 (2.67) | -0.01 |
| Missing; n (%) | 57,550 (57.6%) | 16,145 (58.9%) | 92,102 (93.7%) | 17,885 (94.6%) | N/A | N/A | 149,652 (75.5%) | 34,030 (73.5%) | 0.05 |
| • 17 | | | | | | | | | |
| Lab result number- Albumin mean (only >0 and <=10 includes | 39,793 | 10,600 | 5,330 | 848 | N/A | N/A | 45,123 | 11,448 | |
| mean (sd) | 4.29 (0.32) | 4.32 (0.31) | 4.20 (0.38) | 4.10 (0.39) | N/A | N/A | 4.28 (0.33) | 4.30 (0.32) | -0.06 |
| median [IQR] | 4.30 [4.10, 4.50] | 4.30 [4.10, 4.50] | 4.20 [4.00, 4.45] | 4.00 [4.00, 4.30] | N/A | N/A | 4.29 (0.33) | 4.28 (0.32) | 0.03 |
| Missing, n (%) | 60,110 (60.2%) | 16,794 (61.3%) | 93,015 (94.6%) | 18,064 (95.5%) | N/A | N/A | 153,125 (77.2%) | 34,858 (75.3%) | 0.04 |
| | ,, | | ,() | ,, | | | ,() | ,, | |
| Lab result number- Glucose (fasting or random) mean (only | 42,469 | 11,283 | 6,343 | 1,054 | N/A | N/A | 48.812 | 12,337 | |
| mean (sd) | 178.34 (72.25) | 182.55 (71.67) | 181.56 (74.01) | 177.65 (69.16) | N/A | N/A | 178.76 (72.48) | 182.13 (71.46) | -0.05 |
| median (IQR) | 161.00 [129.00, 209.50] | 167.00 [132.50, 217.00] | 163.00 [130.50, 215.50] | 161.75 [129.00, 209.00] | N/A | N/A | 161.26 (72.48) | 166.55 (71.46) | -0.07 |
| Missing n (%) | 57,434 (57.5%) | 16,111 (58.8%) | 92,002 (93.6%) | 17,858 (94.4%) | N/A | N/A | 149,436 (75.4%) | 33,969 (73.4%) | 0.05 |
| wessing, re(re) | 37,434 [37.37] | 10,111 (30.0/6) | 32,002 (33.0/0) | 17,030 [34.4/9] | nya. | N/A | 143,430 [73,476] | 33,363 [/3.4/6] | 0.03 |
| Lab result number- Potassium mean (only 1-7 included) | 43,384 | 11,485 | 6,118 | 973 | N/A | N/A | 49,502 | 12,458 | |
| mean (sd) | 4.48 (0.43) | 4.47 (0.40) | 4.32 (0.46) | 4.16 (0.50) | N/A | N/A | 4.46 (0.43) | 4.45 (0.41) | 0.02 |
| | | | , , | | N/A | N/A | , , | · · | 0.17 |
| median [IQR] | 4.50 [4.20, 4.70] | 4.45 [4.20, 4.70] | 4.30 [4.00, 4.60] | 4.00 [4.00, 4.50] | | | 4.48 (0.43) | 4.41 (0.41) | |
| Missing n (%) | 56,519 (56.6%) | 15,909 (58.1%) | 92,227 (93.8%) | 17,939 (94.9%) | N/A | N/A | 148,746 (75.0%) | 33,848 (73.1%) | 0.04 |
| Comorbidity Scores | | | | | | | | | |
| CCI (180 days)-ICD9 and ICD10 v2 | | | | | | | | | |
| mean (sd) | 2.43 (1.80) | 2.25 (1.47) | 1.64 (1.30) | 1.67 (1.06) | 2.63 (1.89) | 2.46 (1.56) | 2.34 (1.74) | 2.11(1.38) | 0.15 |
| median [IQR] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 1.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 2.00 [1.00, 4.00] | 2.00 [1.00, 3.00] | 1.76 (1.74) | 2.00 (1.38) | -0.15 |
| Frailty Score: Qualitative Version 365 days as Categories, v1 | | | | | | | | | |
| 0; n (%) | 68,126 (68.2%) | 23,602 (86.2%) | 60,170 (61.2%) | 14,653 (77.5%) | 92,074 (45.3%) | 10,006 (76.1%) | 220,370 (54.9%) | 48,261 (81.2%) | -0.59 |
| 1 to 2; n (%) | 24,208 (24.2%) | 3,375 (12.3%) | 29,743 (30.2%) | 3,605 (19.1%) | 66,971 (32.9%) | 2,319 (17.6%) | 120,922 (30.1%) | 9,299 (15.6%) | 0.35 |
| 3 or more; n (%) | 7,569 (7.6%) | 417 (1.5%) | 8,432 (8.6%) | 654 (3.5%) | 44,249 (21.8%) | 831 (6.3%) | 60,250 (15.0%) | 1,902 (3.2%) | 0.42 |
| Frailty Score: Empirical Version 365 days as Categories, v3 | | | | | | | | | |
| <0.12908; n (%) | 28,978 (29.0%) | 9,111 (33.3%) | 32,840 (33.4%) | 6,951 (36.8%) | 26,735 (13.2%) | 2,162 (16.4%) | 88,553 (22.1%) | 18,224 (30.6%) | -0.19 |
| 0.12908 -0.1631167; n (%) | 33,399 (33.4%) | 9,641 (35.2%) | 36,156 (36.8%) | 7,300 (38.6%) | 55,651 (27.4%) | 4,179 (31.8%) | 125,206 (31.2%) | 21,120 (35.5%) | -0.09 |
| >=0.1631167; n (%) | 37,526 (37.6%) | 8,642 (31.5%) | 29,349 (29.8%) | 4,661 (24.6%) | 120,908 (59.5%) | 6,815 (51.8%) | 187,783 (46.8%) | 20,118 (33.8%) | 0.27 |
| Non-Frailty; n (%) | 57,586 (57.6%) | 16,315 (59.6%) | 50,767 (51.6%) | 10,157 (53.7%) | 10,528 (5.2%) | 611 (4.6%) | 118,881 (29.6%) | 27,083 (45.5%) | -0.33 |
| PVI | | | | | | . , | - 1 | | |
| Frailty Score (mean): Qualitative Version 365 days, v1 | | | | | | | | | |
| mean (sd) | 0.64 (1.29) | 0.21 (0.64) | 0.75 (1.28) | 0.37 (0.86) | 1.43 (1.93) | 0.48 (1.11) | 1.07 (1.64) | 0.32 (0.83) | 0.58 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 (0.00, 0.00) | 1.00 (0.00, 2.00) | 0.00 [0.00, 0.00] | 0.51 (1.64) | 0.00 (0.83) | 0.39 |
| Frailty Score (mean): Empirical Version 365 days, v2 | | | | | | | 1 | | |
| mean (sd) | 0.16 (0.05) | 0.15 (0.04) | 0.15 (0.04) | 0.14 (0.03) | 0.19 (0.06) | 0.17 (0.05) | 0.17 (0.05) | 0.15 (0.04) | 0.44 |
| median (IQR) | 0.15 [0.13, 0.18] | 0.14[0.12, 0.17] | 0.14 [0.12, 0.16] | 0.13 [0.12, 0.16] | | 0.17 [0.14, 0.20] | 0.16 (0.05) | 0.14 (0.04) | 0.44 |
| Healthcare Utilization | 0.13 (0.13, 0.10) | 0.27 [0.22, 0.27] | 0.21 (0.22, 0.20) | 0.13 [0.11, 0.10] | 0.27 (0.24, 0.22) | 0.27 [0.24, 0.25] | 0.20 (0.00) | 5.27(5.54) | |
| | 5.407/5.5%) | 1,088 (4.0%) | 2 250 /2 454 | 447 /2 294) | 12 442 (6 194) | AD2 (2 7%) | 24 207 (5 2%) | 4 007 (2 291) | 0.10 |
| Any hospitalization; n (%) | 5,497 (5.5%) | - 1 | 3,358 (3.4%) | 417 (2.2%) | 12,442 (6.1%) | 482 (3.7%) | 21,297 (5.3%) | 1,987 (3.3%) | 0.10 |
| Any hospitalization within prior 30 days; n (%) | 1,947 (1.9%) | 275 (1.0%) | 982 (1.0%) | 61 (0.3%) | 3,634 (1.8%) | 65 (0.5%) | 6,563 (1.6%) | 401 (0.7%) | |
| Any hospitalization during prior 31-180 days; n (%) | 3,821 (3.8%) | 845 (3.1%) | 2,452 (2.5%) | 362 (1.9%) | 9,387 (4.6%) | 424 (3.2%) | 15,660 (3.9%) | 1,631 (2.7%) | 0.07 |
| Endocrinologist Visit; n (%) | 9,696 (9.7%) | 6,083 (22.2%) | 8,916 (9.1%) | 4,696 (24.8%) | 24,295 (12.0%) | 3,503 (26.6%) | 42,907 (10.7%) | 14,282 (24.0%) | -0.36 |
| Endocrinologist Visit (30 days prior); n (%) | 6,358 (6.4%) | 4,656 (17.0%) | 5,990 (6.1%) | 3,590 (19.0%) | 15,500 (7.6%) | 2,720 (20.7%) | 27,848 (6.9%) | 10,966 (18.4%) | -0.35 |
| Endocrinologist Visit (31 to 180 days prior); n (%) | 6,361 (6.6%) | 4,086 (14.9%) | 5,999 (6.1%) | 3,222 (17.0%) | 17,451 (8.6%) | 2,594 (19.7%) | 30,011 (7.5%) | 9,902 (16.7%) | -0.28 |
| Internal medicine/family medicine visits; n (%) | 79,699 (79.8%) | 19,568 (71.4%) | 85,692 (87.1%) | 15,991 (84.6%) | 164,752 (81.0%) | 10,436 (79.3%) | 330,143 (82.2%) | 45,995 (77.4%) | 0.12 |
| Internal medicine/family medicine visits (30 days prior) v2; | 59,806 (59.9%) | 14,110 (51.5%) | 64,158 (65.2%) | 11,352 (60.0%) | 116,541 (57.3%) | 7,146 (54.3%) | 240,505 (59.9%) | 32,608 (54.8%) | 0.10 |
| Internal medicine/family medicine visits (31 to 180 days pr | | 16,887 (61.6%) | 69,171 (70.3%) | 13,393 (70.8%) | 142,940 (70.3%) | 9,188 (69.8%) | 280,621 (69.9%) | 39,468 (66.4%) | 0.08 |
| Cardiologist visit; n (%) | 23,368 (23.4%) | 6,777 (24.7%) | 14,980 (15.2%) | 3,006 (15.9%) | 60,430 (29.7%) | 4,227 (32.1%) | 98,778 (24.6%) | 14,010 (23.6%) | 0.02 |
| Number of Cardiologist visits (30 days prior); n (%) | 8,018 (8.0%) | 2,440 (8.9%) | 4,841 (4.9%) | 894 (4.7%) | 19,046 (9.4%) | 1,399 (10.6%) | 31,905 (7.9%) | 4,733 (8.0%) | 0.00 |

| Number of Cardiologist visits (31 to 180 days prior); n (%) | 19,586 (19.6%) | 5,663 (20.7%) | 12,542 (12.8%) | 2,550 (13.5%) | 52,580 (25.9%) | 3,650 (27.7%) | 84,708 (21.1%) | 11,863 (20.0%) | 0.03 |
|---|---|---|---|---|---|---|---|---|---|
| Bectrocardiogram v2; n (%) | 26,602 (26.6%) | 7,163 (26.1%) | 22,603 (23.0%) | 4,033 (21.3%) | 61,061 (30.0%) | 4,106 (31.2%) | 110,266 (27.5%) | 15,302 (25.7%) | 0.04 |
| Use of glucose test strips; n (%) | 3,648 (3.7%) | 852 (3.1%) | 3,332 (3.4%) | 754 (4.0%) | 6,468 (3.2%) | 414 (3.1%) | 13,448 (3.3%) | 2,020 (3.4%) | -0.01 |
| Dialysis; n (%) | 26 (0.0%) | 1 (0.0%) | 10 (0.0%) | 0 (0.0%) | • | | - | | |
| Naive new user v8 Copy; n (%) | 13,650 (13.7%) | 1,877 (6.9%) | 13,152 (13.4%) | 1,106 (5.8%) | 24,032 (11.8%) | 647 (4.9%) | 50,834 (12.7%) | 3,630 (6.1%) | 0.23 |
| Nantidiabetic drugs at index date v3 Copy | | | | | | | | | |
| mean (sd) | 2.26 (0.83) | 2.34 (0.93) | 2.28 (0.82) | 2.39 (0.96) | 2.23 (0.83) | 2.44 (0.93) | 2.25 (0.83) | 2.38 (0.94) | -0.15 |
| median (IQR) | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 (0.83) | 2.00 (0.94) | 0.00 |
| number of different/distinct medication prescriptions | | | | | | | | | |
| mean (sd) | 9.99 (4.61) | 10.50 (4.73) | 8.93 (4.09) | 9.97 (4.24) | 9.91 (4.25) | 10.60 (4.22) | 9.69 (4.30) | 10.35 (4.47) | -0.15 |
| median (IQR) | 9.00 [7.00, 12.00] | 10.00 [7.00, 13.00] | 8.00 [6.00, 11.00] | 9.00 [7.00, 12.00] | 9.00 [7.00, 12.00] | 10.00 [8.00, 13.00] | 8.76 (4.30) | 9.68 (4.47) | -0.21 |
| Number of Hospitalizations | | | | | | | \ <i>\</i> | \ / | |
| mean (sd) | 0.07 (0.30) | 0.05 (0.24) | 0.04 (0.21) | 0.02 (0.16) | 0.07 (0.32) | 0.04 (0.23) | 0.06 (0.29) | 0.04 (0.22) | 0.08 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | | 0.00 (0.29) | 0.00 (0.22) | 0.00 |
| Number of hospital days | ,, | ,, | ,, | ,, | ,, | ,, | | | |
| mean (sd) | 0.37 (2.52) | 0.21 (1.44) | 0.19 (1.51) | 0.10 (0.90) | 0.45 (2.78) | 0.19 (1.28) | 0.37 (2.46) | 0.17 (1.26) | 0.10 |
| median (IQR) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | \ <i>\</i> | 0.00 (2.46) | 0.00 (1.26) | 0.00 |
| Number of Emergency Department (ED) visits v3 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00(2.10) | 0.00(2.20) | 0.00 |
| mean (sd) | 0.38 (1.19) | 0.30 (1.09) | 0.07 (0.75) | 0.05 (0.57) | 0.43(1.21) | 0.30 (0.93) | 0.33 (1.11) | 0.22 (0.92) | 0.11 |
| | | · · | \ , , | | · · · | | \ <i>\</i> | \ 1 | 0.00 |
| median (IQR) Number of Office visits | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (1.11) | 0.00 (0.92) | 0.00 |
| mean (sd) | 4.40 (3.47) | 4.68 (3.48) | 3.93 (3.12) | 4.16 (3.11) | 4.87 (3.70) | 5.39 (3.66) | 4.52 (3.51) | 4.67 (3.41) | -0.04 |
| median (IQR) | 4.00 [2.00, 6.00] | 4.00 [2.00, 6.00] | 3.00 [2.00, 5.00] | 3.00 [2.00, 5.00] | 4.00 [2.00, 7.00] | 5.00 [3.00, 7.00] | 3.76 (3.51) | 3.90 (3.41) | -0.04 |
| Number of Endocrinologist visits | | | | | | | | | |
| mean (sd) | 0.44 (2.07) | 1.13 (3.39) | 0.41 (2.05) | 1.25 (3.46) | 0.63 (2.84) | 1.59 (4.88) | 0.53 (2.49) | 1.27 (3.79) | -0.23 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 (2.49) | 0.00 (3.79) | 0.00 |
| Number of internal medicine/family medicine visits | | | | | | | | | |
| mean (sd) | 8.66 (12.52) | 7.06 (10.58) | 6.43 (7.97) | 6.12 (7.44) | 6.99 (9.20) | 6.58 (8.74) | 7.27 (9.87) | 6.65 (9.28) | 0.06 |
| median [IQR] | 5.00 [1.00, 11.00] | 4.00 [0.00, 9.00] | 4.00 [2.00, 8.00] | 4.00 [2.00, 8.00] | 4.00 [1.00, 9.00] | 4.00 [1.00, 9.00] | 4.25 (9.87) | 4.00 (9.28) | 0.03 |
| Number of Cardiologist visits | | | | | | | | | |
| mean (sd) | 1.05 (3.12) | 1.18 (3.46) | 0.59 (2.18) | 0.60 (2.16) | 1.39 (3.76) | 1.50 (3.89) | 1.11 (3.28) | 1.07 (3.22) | 0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (3.28) | 0.00 (3.22) | 0.00 |
| Number electrocardiograms received v2 | | | | | | | | | |
| mean (sd) | 0.49 (1.20) | 0.47 (1.16) | 0.37 (0.88) | 0.33 (0.83) | 0.56(1.18) | 0.55 (1.12) | 0.50 (1.12) | 0.44 (1.06) | 0.06 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (1.12) | 0.00 (1.06) | 0.00 |
| Number of HbA1c tests ordered | | | | | | | . , | , , | |
| mean (sd) | 1.29 (0.88) | 1.37 (0.88) | 1.09 (0.85) | 1.33 (0.82) | 1.41 (0.85) | 1.57 (0.81) | 1.30 (0.86) | 1.40 (0.85) | -0.12 |
| median (IQR) | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | | 1.00 (0.86) | 1.22 (0.85) | -0.26 |
| Number of glucose tests ordered | | | | | | | | | |
| mean (sd) | 0.55 (3.54) | 0.46 (1.58) | 0.34 (1.10) | 0.43 (1.22) | 0.42 (1.02) | 0.48 (1.08) | 0.43 (1.99) | 0.45 (1.37) | -0.01 |
| median (IQR) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | | 0.00 (1.99) | 0.00 (1.37) | 0.00 |
| Number of lipid tests ordered | | | | | | | () | () | |
| mean (sd) | 0.97 (0.91) | 1.01 (0.94) | 0.89 (1.17) | 1.05 (1.16) | 0.98 (0.81) | 1.07 (0.83) | 0.96 (0.93) | 1.04 (0.99) | -0.08 |
| median [IQR] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | | 1.00 [1.00, 2.00] | 1.00 (0.93) | 1.00 (0.99) | 0.00 |
| mesian pupi<br>Number of creatinine tests ordered | 2.00 [0.00, 2.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 2.00 (0.00, 2.00) | 1.00 (0.00, 1.00) | 2.00 [2.00, 2.00] | 1.00 (0.93) | 2.00 (0.33) | 0.00 |
| mean (sd) | 0.04 (0.26) | 0.04 (0.25) | 0.03 (0.23) | 0.04 (0.25) | 0.06 (0.32) | 0.07 (0.34) | 0.05 (0.29) | 0.05 (0.27) | 0.00 |
| mean (sa)<br>median (lQR) | | 0.04 (0.25) | 0.03 (0.23) | 0.04 (0.25) | | | | | 0.00 |
| Number of BUN tests ordered | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.29) | 0.00 (0.27) | 0.00 |
| | 0.02 (0.20) | 0.02 (0.17) | 0.02 (0.18) | 0.02 (0.17) | 0.04(0.26) | 0.04 (0.26) | 0.03 (0.33) | 0.02 (0.19) | 0.05 |
| mean (sd) | | | | | | | 0.03 (0.23) | | |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.23) | 0.00 (0.19) | 0.00 |
| Number of tests for microal burninuma | | | | | | | | | |
| meen (sd) | 0.81 (1.17) | 0.87 (1.18) | 0.64 (1.03) | 0.81 (1.12) | 0.48 (0.70) | 0.56 (0.71) | 0.60 (0.92) | 0.78 (1.07) | -0.18 |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (0.92) | 0.00 (1.07) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd digit level Co | | | | | | | | | |
| mean (sd) | 6.92 (7.38) | 8.25 (6.87) | 2.91 (3.94) | 3.91 (3.75) | 6.39 (7.39) | 8.79 (7.04) | 5.67 (6.71) | 6.99 (6.10) | -0.21 |
| median [IQR] | 5.00 [0.00, 10.00] | 7.00 [4.00, 11.00] | 2.00 [0.00, 5.00] | 4.00 [0.00, 6.00] | 5.00 [0.00, 10.00] | 7.00 [4.00, 12.00] | 4.27 (6.71) | 6.05 (6.10) | -0.28 |
| Use of thiazide; n (%) | 11,963 (12.0%) | 3,080 (11.2%) | 10,371 (10.5%) | 1,926 (10.2%) | 27,843 (13.7%) | 1,804 (13.7%) | 50,177 (12.5%) | 6,810 (11.5%) | 0.03 |
| Use of beta blockers; n (%) | 36,576 (36.6%) | 9,851 (36.0%) | 30,224 (30.7%) | 5,661 (29.9%) | 96,233 (47.3%) | 6,419 (48.8%) | 163,033 (40.6%) | 21,931 (36.9%) | 0.08 |
| Use of calcium channel blockers; n (%) | 30,078 (30.1%) | 7,288 (26.6%) | 26,215 (26.7%) | 4,370 (23.1%) | 69,690 (34.3%) | 4,001 (30.4%) | 125,983 (31.4%) | 15,659 (26.3%) | 0.11 |

| | Unmatched | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| · · | Optu | m | Market | ican | Medicare | | | POOLED | |
| • | Орго | Exposure - Empaginican | | Exposure - Empagimozin | THE GIVE | Exposure - | | Exposure - Empaginiozin | |
| Variable | Reference-DPP4i v2 | v3 | Reference-DPP4iv2 | v3 | Reference-DPP4i v2 | | Reference-DPP4iv2 | v3 | St. Diff. |
| Number of patients | 99,903 | 27,394 | 98,345 | 18,912 | 203,294 | 13,156 | 401,542 | 59,462 | |
| Age | | | | | | | | | |
| mean (sd) | 64.93 (11.69) | 60.53 (10.62) | 58.66 (11.12) | 55.47 (8.77) | 74.08 (6.94) | 71.46 (5.19) | 68.03 (9.42) | 61.34 (9.08) | 0.72 |
| median [IQR] | 66.00 [37.00, 73.00] | 61.00 [53.00, 68.00] | 58.00 [52.00, 64.00] | 56.00 [50.00, 61.00] | 73.00 [68.00, 78.00] 0 | .00 [68.00, 74.00] | 67.58 (9.42) | 61.40 (9.08) | 0.67 |
| Age categories without zero category | | | | | | | | | |
| 18 - 54; n (%) | 19,490 (19.5%) | 7,748 (28.3%) | 33,966 (34.5%) | 7,944 (42.0%) | 0 (0.0%) | 0 (0.0%) | 53,456 (13.3%) | 15,692 (26.4%) | -0.33 |
| 55 -64; n (%) | 23,551 (23.6%) | 8,844 (32.3%) | 41,612 (42.3%) | 9,123 (48.2%) | 1,132 (0.6%) | 43 (0.3%) | 66,295 (16.5%) | 18,010 (30.3%) | -0.33<br>0.18 |
| 65 - 74; n (%)<br>>=75; n (%) | 36,281 (36.3%)<br>20,581 (20.6%) | 8,539 (31.2%)<br>2,263 (8.3%) | 13,769 (14.0%)<br>8,998 (9.1%) | 1,483 (7.8%)<br>362 (1.9%) | 119,235 (58.7%)<br>82,927 (40.8%) | 9,986 (75.9%)<br>3,127 (23.8%) | 169,285 (42.2%)<br>112,506 (28.0%) | 20,008 (33.6%)<br>5,752 (9.7%) | 0.18 |
| Gender without zero category-United | 20,361 (20.6/6) | 2,203 (0.3/9) | 0,330 [3.1/6] | 302 (1.3/6) | 02,327 [40.070] | 3,127 (23.0/9) | 112,300 (20.0/6) | 3,732 (3.770) | 0.46 |
| Males; n (%) | 53,340 (53.4%) | 16,618 (60.7%) | 57,603 (58.6%) | 11,785 (62.3%) | 92,595 (45.5%) | 7,494 (57.0%) | 203,538 (50.7%) | 35,897 (60.4%) | -0.20 |
| Females; n (%) | 46,563 (46.6%) | 10,776 (39.3%) | 40,742 (41.4%) | 7,127 (37.7%) | 110,699 (54.5%) | 5,662 (43.0%) | 198,004 (49.3%) | 23,565 (39.6%) | 0.20 |
| Race | | | | | | | | | |
| White; n (%) | N/A | N/A | N/A | N/A | 151,073 (74.3%) | 10,799 (82.1%) | 151,073 (74.3%) | 10,799 (82.1%) | -0.19 |
| Black; n (%) | N/A | N/A | N/A | N/A | 22,905 (11.3%) | 916 (7.0%) | 22,905 (11.3%) | 916 (7.0%) | 0.15 |
| Asian; n (%) | N/A | N/A | N/A | N/A | 9,749 (4.8%) | 387 (2.9%) | 9,749 (4.8%) | 387 (2.9%) | 0.10 |
| Hispanic; n (%) | N/A | N/A | N/A | N/A | 9,554 (4.7%) | 333 (2.5%) | 9,554 (4.7%) | 333 (2.5%) | 0.12 |
| North American Native; n (%) | N/A | N/A | N/A | N/A | 1,385 (0.7%) | 58 (0.4%) | 1,385 (0.7%) | 58 (0.4%) | 0.04 |
| Other/Unknown; n (%) | N/A | N/A | N/A | N/A | 8,628 (4.2%) | 663 (5.0%) | 8,628 (4.2%) | 663 (5.0%) | -0.04 |
| Region without zero category-United v3 (lumping missing | &other category with West) | | | | | | | | |
| Northeast; n (%) | 10,960 (11.0%) | 2,334 (8.5%) | 17,603 (17.9%) | 2,575 (13.6%) | 38,218 (18.8%) | 2,505 (19.0%) | 66,781 (16.6%) | 7,414 (12.5%) | 0.12 |
| South; n (%) | 52,164 (52.2%) | 15,303 (55.9%) | 20,254 (20.6%) | 3,296 (17.4%) | 86,895 (42.7%) | 5,524 (42.0%) | 159,313 (39.7%) | 24,123 (40.6%) | -0.02 |
| Midwest; n (%) | 18,103 (18.1%) | 5,373 (19.6%) | 50,370 (51.2%) | 11,006 (38.2%) | 42,468 (20.9%) | 2,506 (19.0%) | 110,941 (27.6%) | 18,885 (31.8%) | -0.09 |
| West; n (%) | 18,676 (18.7%) | 4,384 (16.0%) | 9,489 (9.6%) | 1,978 (10.5%) | 35,713 (17.6%) | 2,621 (19.9%) | 63,878 (15.9%) | 8,983 (15.1%) | 0.02 |
| Unknown+missing; n (%) | N/A | N/A | 629 (0.6%) | 57 (0.3%) | N/A | N/A | 629 (0.6%) | 57 (0.3%) | 0.04 |
| CV Covariates | | | | | | | | | |
| Ischemicheart disease; n (%)<br>Acute MI; n (%) | 18,990 (19.0%)<br>931 (0.9%) | 5,885 (21.5%)<br>344 (1.3%) | 12,693 (12.9%)<br>372 (0.4%) | 2,535 (13.4%)<br>104 (0.5%) | 54,534 (26.8%)<br>1,288 (0.6%) | 4,200 (31.9%)<br>89 (0.7%) | 86,217 (21.5%)<br>2,591 (0.6%) | 12,620 (21.2%)<br>537 (0.9%) | 0.01<br>-0.03 |
| ACS/unstable angina; n (%) | 702 (0.7%) | 231 (0.8%) | 300 (0.5%) | 107 (0.6%) | 1,499 (0.7%) | 118 (0.9%) | 2,701 (0.7%) | 456 (0.8%) | -0.01 |
| Old MI; n (%) | 2,549 (2.6%) | 819 (3.0%) | 906 (0.9%) | 191 (1.0%) | 5,824 (2.9%) | 466 (3.5%) | 9,279 (2.3%) | 1,476 (2.5%) | -0.01 |
| Stable angina; n (%) | 3,164 (3.2%) | 1,100 (4.0%) | 1,545 (1.6%) | 382 (2.0%) | 6,343 (3.1%) | 626 (4.8%) | 11,052 (2.8%) | 2,108 (3.5%) | -0.04 |
| Coronary atherosclerosis and other forms of chronic ischer | 17,701 (17.7%) | 5,558 (20.3%) | 11,987 (12.2%) | 2,406 (12.7%) | 52,219 (25.7%) | 4,074 (31.0%) | 81,907 (20.4%) | 12,038 (20.2%) | 0.00 |
| Other atherosclerosis with ICD10 v2 Copy; n (%) | 501 (0.5%) | 106 (0.4%) | 451 (0.5%) | 57 (0.3%) | 2,443 (1.2%) | 86 (0.7%) | 3,395 (0.8%) | 249 (0.4%) | 0.05 |
| Previous cardiac procedure (CABG or PTCA or Stent) v4; n (5 | 407 (0.4%) | 189 (0.7%) | 212 (0.2%) | 52 (0.3%) | 461 (0.2%) | 55 (0.4%) | 1,080 (0.3%) | 296 (0.5%) | -0.03 |
| History of CABG or PTCA; n (%) | 4,493 (4.5%) | 1,679 (6.1%) | 1,629 (1.7%) | 369 (2.0%) | 13,342 (6.6%) | 1,156 (8.8%) | 19,464 (4.8%) | 3,204 (5.4%) | -0.03 |
| Anystroke; n (%) | 4,963 (5.0%) | 1,153 (4.2%) | 2,035 (2.1%) | 273 (1.4%) | 10,123 (5.0%) | 391 (4.3%) | 17,121 (4.3%) | 2,017 (3.4%) | 0.05 |
| | 4,000 (0.0.4) | 2,222(1.2.4) | 2,000 [2.2.4] | 2.0 (2) | 20,223 (3.0.4) | 552() | | 4,444 | |
| Ischemic stroke (wand w/o mention of cerebral infarction) | 4,899 (4.9%) | 1,140 (4.2%) | 2,000 (2.0%) | 271 (1.4%) | 9,999 (4.9%) | 385 (4.4%) | 16,898 (4.2%) | 1,996 (3.4%) | 0.04 |
| Hemorrhagic stroke; n (%) | 163 (0.2%) | 23 (0.1%) | 48 (0.0%) | 4 (0.0%) | | | | | |
| TIA; n (%) | 1,176 (1.2%) | 266 (1.0%) | 465 (0.5%) | 68 (0.4%) | 1,913 (0.9%) | 98 (0.7%) | 3,554 (0.9%) | 432 (0.7%) | 0.02 |
| Other cerebrovascular disease; n (%) | 1,704 (1.7%) | 322 (1.2%) | 670 (0.7%) | 86 (0.5%) | 3,962 (1.9%) | 236 (1.8%) | 6,336 (1.6%) | 644 (1.1%) | 0.04 |
| Late effects of cerebrovascular disease; n (%) | 1,554 (1.6%) | 233 (0.9%) | 423 (0.4%) | 34 (0.2%) | 3,186 (1.6%) | 107 (0.8%) | 5,163 (1.3%) | 374 (0.6%) | 0.07 |
| Cerebrovascular procedure; n (%)<br>Heart failure (CHF); n (%) | 70 (0.1%)<br>6,419 (6.4%) | 28 (0.1%)<br>1,435 (5.2%) | 15 (0.0%)<br>2,935 (3.0%) | 4 (0.0%)<br>399 (2.1%) | 18,631 (9.2%) | 951 (7.2%) | 27 005 /7 0%) | 2,785 (4.7%) | 0.10 |
| Heart failure (CHF); ft (76) | 6,419 (6.4%) | 1,453 (3.2%) | 2,933 (3.0%) | 399 (2.176) | 18,631 (9.276) | 931 (7.2%) | 27,985 (7.0%) | 2,783 [4.776] | 0.10 |
| Peripheral Vascular Disease (PVD) or PVD Surgery v2; n (%) | 6,638 (6.6%) | 1,465 (5.3%) | 3,369 (3.4%) | 497 (2.6%) | 20,972 (10.3%) | 1,195 (9.1%) | 30,979 (7.7%) | 3,157 (5.3%) | 0.10 |
| Atrial fibrillation; n (%) | 5,807 (5.8%) | 1,313 (4.8%) | 3,583 (3.6%) | 474 (2.5%) | 20,723 (10.2%) | 1,268 (9.6%) | 30,113 (7.5%) | 3,055 (5.1%) | 0.10 |
| Other cardiac dysrhythmia; n (%) | 8,278 (8.3%) | 2,142 (7.8%) | 4,579 (4.7%) | 793 (4.2%) | 24,622 (12.1%) | 1,806 (13.7%) | 37,479 (9.3%) | 4,741 (8.0%) | 0.05 |
| Cardiac conduction disorders; n (%) | 2,246 (2.2%) | 580 (2.1%) | 1,171 (1.2%) | 192 (1.0%) | 6,903 (3.4%) | 459 (3.5%) | 10,320 (2.6%) | 1,231 (2.1%) | 0.03 |
| Other CVD; n (%) | 8,797 (8.8%) | 2,259 (8.2%) | 5,483 (5.6%) | 817 (4.3%) | 25,637 (12.6%) | 1,671 (12.7%) | 39,917 (9.9%) | 4,747 (8.0%) | 0.07 |
| Diabetes-related complications | p to -== | | | | | | | !* ' | |
| Diabetic retinopathy; n (%) | 6,367 (6.4%) | 2,196 (8.0%) | 3,371 (3.4%) | 764 (4.0%) | 14,304 (7.0%) | 1,298 (9.9%) | 24,042 (6.0%) | 4,258 (7.2%) | -0.05 |
| Diabetes with other ophthalmic manifestations; n (%) | 904 (0.9%) | 230 (0.8%) | 1,868 (1.9%) | 305 (1.6%) | 4,906 (2.4%) | 267 (2.0%) | 7,678 (1.9%) | 802 (1.3%) | 0.05 |
| Retinal detachment, vitreous hemorrhage, vitrectomy; n (7 | 415 (0.4%) | 135 (0.5%) | 328 (0.3%) | 76 (0.4%) | 780 (0.4%) | 80 (0.6%) | 1,523 (0.4%) | 291 (0.5%) | -0.01 |
| Retinal laser coagulation therapy; n (%) | 560 (0.6%) | 158 (0.6%) | 504 (0.5%) | 115 (0.6%) | 1,220 (0.6%) | 74 (0.6%) | 2,284 (0.6%) | 347 (0.6%) | 0.00 |
| Occurrence of Diabetic Neuropathy v2 Copy; n (%) | 19,198 (19.2%) | 5,771 (21.1%) | 10,496 (10.7%) | 2,631 (13.9%) | 39,771 (19.6%) | 3,284 (25.0%) | 69,465 (17.3%) | 11,686 (19.7%) | -0.06 |

| Occurrence of diabetic nephropathy V3 with ICD10 Copy; r | 15,429 (15.4%) | 3,259 (11.9%) | 6,218 (6.3%) | 1,309 (6.9%) | 22,695 (11.2%) | 1,478 (11.2%) | 44,342 (11.0%) | 6,046 (10.2%) | 0.03 |
|---|---|---|---|---|---|---|---|---|---|
| Hypoglycemia v2; n (%) | 1,757 (1.8%) | 141 (0.5%) | 1,705 (1.7%) | 183 (1.0%) | 4,423 (2.2%) | 107 (0.8%) | 7,885 (2.0%) | 431 (0.7%) | 0.11 |
| Hyperglycemia; n (%) | 4,186 (4.2%) | 1,098 (4.0%) | 3,136 (3.2%) | 518 (2.7%) | 8,064 (4.0%) | 466 (3.5%) | 15,386 (3.8%) | 2,082 (3.5%) | 0.02 |
| 11 01 - 17 | | | | | | | | | |
| Disorders of fluid electrolyte and acid-base balance; n (%) | 6,080 (6.1%) | 1,099 (4.0%) | 3,203 (3.3%) | 434 (2.3%) | 12,731 (6.3%) | 479 (3.6%) | 22,014 (5.5%) | 2,012 (3.4%) | 0.10 |
| Diabetic ketoacidosis: n (%) | 385 (0.4%) | 76 (0.3%) | 309 (0.3%) | 47 (0.2%) | 668 (0.3%) | 22 (0.2%) | 1,362 (0.3%) | 145 (0.2%) | 0.02 |
| | | | | | | | 4 | | |
| Hyperosmolar hyperglycemic nonketotic syndrome (HONK | 589 (0.6%) | 166 (0.6%) | 468 (0.5%) | 92 (0.5%) | 1,077 (0.5%) | 80 (0.6%) | 2,134 (0.5%) | 338 (0.6%) | -0.01 |
| · | () | | 100 | 55 (5.5.4) | 2,011 (0.014) | | -,, | | |
| Diabetes with peripheral circulatory disorders with ICD-10 | 7,150 (7.2%) | 1,909 (7.0%) | 2,798 (2.8%) | 630 (3.3%) | 15,464 (7.6%) | 1,122 (8.5%) | 25,412 (6.3%) | 3,661 (6.2%) | 0.00 |
| Diabetic Foot; n (%) | 1,967 (2.0%) | 591 (2.2%) | 1,422 (1.4%) | 320 (1.7%) | 4,932 (2.4%) | 286 (2.2%) | 8,321 (2.1%) | 1,197 (2.0%) | 0.01 |
| | | | - 1 | · · · | | | | | 0.00 |
| Gangrenev2; n (%) | 235 (0.2%) | 63 (0.2%) | 144 (0.1%) | 28 (0.1%) | 380 (0.2%) | 33 (0.3%) | 759 (0.2%) | 124 (0.2%) | |
| Lower extremity amputation; n (%) | 644 (0.6%) | 207 (0.8%) | 256 (0.3%) | 66 (0.3%) | 1,155 (0.6%) | 81 (0.6%) | 2,055 (0.5%) | 354 (0.6%) | -0.01 |
| Osteomyelitis; n (%) | 491 (0.5%) | 155 (0.6%) | 361 (0.4%) | 78 (0.4%) | 936 (0.5%) | 34 (0.4%) | 1,788 (0.4%) | 287 (0.5%) | -0.01 |
| Skin infections v2; n (%) | 4,914 (4.9%) | 1,384 (5.1%) | 4,428 (4.5%) | 886 (4.7%) | 11,729 (5.8%) | 781 (5.9%) | 21,071 (5.2%) | 3,051 (5.1%) | 0.00 |
| Erectile dysfunction; n (%) | 2,938 (2.9%) | 1,188 (4.3%) | 2,680 (2.7%) | 585 (3.1%) | 4,367 (2.1%) | 501 (3.8%) | 9,985 (2.5%) | 2,274 (3.8%) | -0.07 |
| Diabetes with unspecified complication; n (%) | 5,922 (5.9%) | 1,946 (7.1%) | 4,818 (4.9%) | 1,306 (6.9%) | 11,396 (5.6%) | 953 (7.2%) | 22,136 (5.5%) | 4,205 (7.1%) | -0.07 |
| Diabetes mellitus without mention of complications; n (%) | 82,871 (83.0%) | 21,178 (77.3%) | 86,660 (88.1%) | 15,269 (80.7%) | 184,478 (90.7%) | 11,109 (84.4%) | 354,009 (88.2%) | 47,556 (80.0%) | 0.23 |
| Hypertension: 1 inpatient or 2 outpatient claims within 36 | 84,740 (84.8%) | 23,304 (85.1%) | 75,314 (76.6%) | 14,637 (77.4%) | 185,875 (91.4%) | 11,981 (91.1%) | 345,929 (86.2%) | 49,922 (84.0%) | 0.06 |
| Hyperlipidemia v2; n (%) | 70,468 (70.5%) | 19,569 (71.4%) | 65,929 (67.0%) | 13,478 (71.3%) | 154,166 (75.8%) | 10,169 (77.3%) | 290,563 (72.4%) | 43,216 (72.7%) | -0.01 |
| Edema; n (%) | 5,273 (5.3%) | 1,202 (4.4%) | 2,878 (2.9%) | 467 (2.5%) | 16,056 (7.9%) | 876 (6.7%) | 24,207 (6.0%) | 2,545 (4.3%) | 0.08 |
| Renal Dysfunction (non-diabetic) v2; n (%) | 19,382 (19.6%) | 3,179 (11.6%) | 8,494 (8.6%) | 958 (5.1%) | 42,497 (20.9%) | 1,822 (13.8%) | 70,573 (17.6%) | 5,959 (10.0%) | 0.22 |
| Occurrence of acute renal disease v2; n (%) | 2,581 (2.6%) | 332 (1.2%) | 1,243 (1.3%) | 80 (0.4%) | 5.423 (2.7%) | 130 (1.0%) | 9.247 (2.3%) | 542 (0.9%) | 0.11 |
| | | | | | -, | | -, | | |
| Occurrence of chronic renal insufficiency; n (%) | 16,369 (16.4%) | 2,354 (8.6%) | 6,265 (6.4%) | 657 (3.5%) | 36,061 (17.7%) | 1,453 (11.0%) | 58,695 (14.6%) | 4,464 (7.5%) | 0.23 |
| Chronic kidney disease v2; n (%) | 15,864 (15.9%) | 2,270 (8.3%) | 5,871 (6.0%) | 615 (3.3%) | 34,532 (17.0%) | 1,391 (10.6%) | 56,267 (14.0%) | 4,276 (7.2%) | 0.22 |
| CKD Stage 3-4; n (%) | 10,687 (10.7%) | 1,245 (4.5%) | 3,761 (3.8%) | 303 (1.6%) | 24,060 (11.8%) | 839 (6.4%) | 38,508 (9.6%) | 2,387 (4.0%) | 0.22 |
| Occurrence of hypertensive nephropathy; n (%) | 6,766 (6.8%) | 968 (3.5%) | 2,293 (2.3%) | 229 (1.2%) | 13,584 (6.7%) | 526 (4.0%) | 22,643 (5.6%) | 1,723 (2.9%) | 0.13 |
| Occurrence of miscellaneous renal insufficiency v2; n (%) | 4,400 (4.4%) | 874 (3.2%) | 2,417 (2.5%) | 271 (1.4%) | 11,162 (5.5%) | 523 (4.0%) | 17,979 (4.5%) | 1,668 (2.8%) | 0.09 |
| Glaucoma or cataracts v2; n (%) | 18,320 (18.3%) | 4,419 (16.1%) | 12,973 (13.2%) | 2,270 (12.0%) | 54,403 (26.8%) | 3,639 (27.7%) | 85,696 (21.3%) | 10,328 (17.4%) | 0.10 |
| Cellulitis or abscess of toe; n (%) | 1,284 (1.3%) | 391 (1.4%) | 849 (0.9%) | 225 (1.2%) | 2,592 (1.3%) | 237 (1.8%) | 4,725 (1.2%) | 853 (1.4%) | -0.02 |
| Footuicer; n (%) | 1,877 (1.9%) | 539 (2.0%) | 1,377 (1.4%) | 296 (1.6%) | 4.802 (2.4%) | 270 (2.1%) | 8.056 (2.0%) | 1,105 (1.9%) | 0.01 |
| Bladder stones; n (%) | 125 (0.1%) | 27 (0.1%) | 71 (0.1%) | 11 (0.1%) | 307 (0.2%) | 17 (0.1%) | 503 (0.1%) | 55 (0.1%) | 0.00 |
| Kidneystones; n (%) | 1,974 (2.0%) | 533 (1.9%) | 1,775 (1.8%) | 310 (1.6%) | 4,540 (2.2%) | 294 (2.2%) | 8,289 (2.1%) | 1,137 (1.9%) | 0.01 |
| 1 | | | | | | | | | |
| Urinary tract infections (UTIs); n (%) | 7,752 (7.8%) | 1,339 (4.9%) | 4,684 (4.8%) | 565 (3.0%) | 23,016 (11.3%) | 885 (6.7%) | 35,452 (8.8%) | 2,789 (4.7%) | 0.16 |
| Dipstick urinelysis; n (%) | 34,548 (34.6%) | 8,269 (30.2%) | 29,300 (29.8%) | 5,259 (27.8%) | 76,034 (37.4%) | 4,496 (34.2%) | 139,882 (34.8%) | 18,024 (30.3%) | 0.10 |
| Non-dipstick urinalysis; n (%) | 43,363 (43.4%) | 12,648 (46.2%) | 36,411 (37.0%) | 8,432 (44.6%) | 84,136 (41.4%) | 6,319 (48.0%) | 163,910 (40.8%) | 27,399 (46.1%) | -0.11 |
| Urine function test; n (%) | 1,897 (1.9%) | 418 (1.5%) | 1,625 (1.7%) | 200 (1.1%) | 6,250 (3.1%) | 434 (3.3%) | 9,772 (2.4%) | 1,052 (1.8%) | 0.04 |
| Cytology; n (%) | 360 (0.6%) | 117 (0.4%) | 522 (0.5%) | 60 (0.3%) | 1,497 (0.7%) | 67 (0.5%) | 2,579 (0.6%) | 244 (0.4%) | 0.03 |
| Cystoscopy; n (%) | 843 (0.8%) | 204 (0.7%) | 726 (0.7%) | 103 (0.5%) | 2,199 (1.1%) | 129 (1.0%) | 3,768 (0.9%) | 436 (0.7%) | 0.02 |
| Other Covariates | 1 | 1 | 1 | 1 | | | | ( ) | |
| Liver disease; n (%) | 3,416 (3.4%) | 1,355 (4.9%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 3,416 (0.9%) | 1,355 (2.3%) | -0.11 |
| Osteoarthritis; n (%) | 14,159 (14.2%) | 3,503 (12.8%) | 8,944 (9.1%) | 1,459 (7.7%) | 41,716 (20.5%) | 2,523 (19.2%) | 64,819 (16.1%) | 7,485 (12.6%) | 0.10 |
| Carcara tra rea, in proj | 24,255 (24.274) | 3,505 (12.074) | 0,544 (5.254) | 2,455 (1.114) | 42,720 (20.579) | 2,23(23,23) | 04,025 (20.254) | 7,405 (12.074) | 0.20 |
| Other arthritis, arthropathies and musculoskeletal pain; n | 33,077 (33.1%) | 8,620 (31.5%) | 26,598 (27.0%) | 4,912 (26.0%) | 82,377 (40.5%) | 4,956 (37.7%) | 142,052 (35.4%) | 18,488 (31.1%) | 0.09 |
| Dorsopathies; n (%) | 20,631 (20.7%) | 3,739 (21.0%) | 15,907 (16.2%) | 3,084 (16.3%) | 48,687 (23.9%) | 3,203 (24.3%) | 85,225 (21.2%) | 12,046 (20.3%) | 0.02 |
| Fractures; n (%) | 2,412 (2.4%) | 501 (1.8%) | 1,716 (1.7%) | 279 (1.5%) | 6,339 (3.1%) | 342 (2.6%) | 10,467 (2.6%) | 1,122 (1.9%) | 0.05 |
| Fallsv2; n (%) | 3,187 (3.2%) | 522 (1.9%) | 965 (1.0%) | 123 (0.7%) | 7,872 (3.9%) | 346 (2.6%) | 12,024 (3.0%) | 991 (1.7%) | 0.09 |
| Osteoporosis; n (%) | 4,316 (4.3%) | 634 (2.3%) | 1,543 (1.6%) | 149 (0.8%) | 15,070 (7.4%) | 631 (4.8%) | 20,929 (5.2%) | 1,414 (2.4%) | 0.15 |
| Hyperthyroidism; n (%) | 588 (0.6%) | 179 (0.7%) | 466 (0.5%) | 85 (0.4%) | 1,690 (0.8%) | 99 (0.8%) | 2,744 (0.7%) | 363 (0.6%) | 0.01 |
| Hypothyroidism v2; n (%) | 13,829 (13.8%) | 3,532 (12.9%) | 10,304 (10.5%) | 2,178 (11.5%) | 21,523 (10.6%) | 946 (7.2%) | 45,656 (11.4%) | 6,636 (11.2%) | 0.01 |
| Other disorders of thyroid gland V2; n (%) | 3,455 (3.5%) | 1,215 (4.4%) | 2,934 (3.0%) | 902 (4.8%) | 7,712 (3.8%) | 667 (5.1%) | 14,101 (3.5%) | 2,784 (4.7%) | -0.06 |
| Depression; n (%) | 7,320 (7.3%) | 1,821 (6.6%) | 5,335 (5.4%) | 914 (4.8%) | 17,919 (8.8%) | 902 (6.9%) | 30,574 (7.6%) | 3,637 (6.1%) | 0.06 |
| Anxiety; n (%) | 7,953 (8.0%) | 2,396 (8.7%) | 5,309 (5.4%) | 1,125 (5.9%) | 15,687 (7.7%) | 995 (7.6%) | 28,949 (7.2%) | 4,516 (7.6%) | -0.02 |
| Sleep Disorder; n (%) | 3,987 (4.0%) | 673 (2.5%) | 5,785 (5.9%) | 766 (4.1%) | 11,002 (5.4%) | 418 (3.2%) | 20,774 (5.2%) | 1,857 (3.1%) | 0.11 |
| Dementia: n (%) | 3,796 (3.8%) | 361 (1.3%) | 1,343 (1.4%) | 91 (0.5%) | 14,445 (7.1%) | 369 (2.8%) | 19,584 (4.9%) | 821 (1.4%) | 0.11 |
| - 17 | | | | | | ١ ، | | \ \ / | 0.20 |
| Delirium; n (%) | 1,038 (1.0%) | 110 (0.4%) | 410 (0.4%) | 31 (0.2%) | 2,997 (1.5%) | 80 (0.6%) | 4,445 (1.1%) | 221 (0.4%) | |
| Psychosis; n (%) | 1,115 (1.1%) | 171 (0.6%) | 403 (0.4%) | 36 (0.2%) | 3,561 (1.8%) | 67 (0.5%) | 5,079 (1.3%) | 274 (0.5%) | 0.08 |
| Obesity; n (%) | 17,344 (17.6%) | 7,711 (28.1%) | 6,568 (6.7%) | 1,684 (8.9%) | 10,068 (5.0%) | 806 (6.1%) | 34,180 (8.5%) | 10,201 (17.2%) | -0.26 |
| Overweight; n (%) | 7,117 (7.1%) | 2,123 (7.7%) | 3,068 (3.1%) | 700 (3.7%) | 8,443 (4.2%) | 650 (4.9%) | 18,628 (4.6%) | 3,473 (5.8%) | -0.05 |
| Smoking; n (%) | 10,562 (10.6%) | 3,243 (11.8%) | 4,864 (4.9%) | 882 (4.7%) | 21,088 (10.4%) | 1,434 (10.9%) | 36,514 (9.1%) | 5,559 (9.3%) | -0.01 |
| Alcohol abuse or dependence; n (%) | 685 (0.7%) | 199 (0.7%) | o (o.a%) | 0 (0.0%) | ò (0.0%) | ò (0.0%) | #VALUE! | 199 (0.3%) | #VALUE! |
| Drug abuse or dependence; n (%) | 1,133 (1.1%) | 359 (1.3%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 1,133 (0.3%) | 359 (0.6%) | -0.04 |
| COPD; n (%) | 6,952 (7.0%) | 1,485 (5.4%) | 3,056 (3.1%) | 386 (2.0%) | 17,808 (8.8%) | 895 (6.8%) | 27,816 (6.9%) | 2,766 (4.7%) | 0.09 |
| | -,(-,) | -, () | -,() | | | | | | |

| Asthma; n (%) | 4,622 (4.6%) | 1,225 (4.5%) | 3,363 (3.4%) | 592 (3.1%) | 9,980 (4.9%) | 656 (5.0%) | 17,965 (4.5%) | 2,473 (4.2%) | 0.01 |
|---|---|---|---|---|---|---|---|---|---|
| Obstructive sleep apnes; n (%) | 7,880 (7.9%) | 3,326 (12.1%) | 7,903 (8.0%) | 2,046 (10.8%) | 10,766 (5.3%) | 1,274 (9.7%) | 26,549 (6.6%) | 6,646 (11.2%) | -0.16 |
| Pneumonia; n (%) | 1,745 (1.7%) | 319 (1.2%) | 1,136 (1.2%) | 158 (0.8%) | 4,422 (2.2%) | 214 (1.6%) | 7,303 (1.8%) | 691 (1.2%) | 0.05 |
| Imaging; n (%) | 73 (0.1%) | 17 (0.1%) | 17 (0.0%) | 4 (0.0%) | | ** | | | •• |
| Diabetes Medications | | | | | | | | | |
| DM Medications - AGIs; n (%) | 499 (0.5%) | 97 (0.4%) | 310 (0.3%) | 64 (0.3%) | 1,243 (0.6%) | 58 (0.4%) | 2,052 (0.5%) | 219 (0.4%) | 0.01 |
| DM Medications - Glitazones; n (%) | 7,594 (7.6%) | 2,318 (8.5%) | 6,881 (7.0%) | 1,520 (8.0%) | 14,722 (7.2%) | 1,253 (9.5%) | 29,197 (7.3%) | 5,091 (8.6%) | -0.05 |
| DM Medications - GLP-1 RA; n (%) | 4,184 (4.2%) | 5,850 (21.4%) | 4,354 (4.4%) | 4,829 (25.5%) | 5,290 (2.6%) | 2,529 (19.2%) | 13,828 (3.4%) | 13,208 (22.2%) | -0.59 |
| DM Medications - Insulin; n (%) | 17,835 (17.9%) | 7,838 (28.6%) | 14,817 (15.1%) | 5,867 (31.0%) | 39,115 (19.2%) | 4,548 (34.6%) | 71,767 (17.9%) | 18,253 (30.7%) | -0.30 |
| DM Medications - Meglitinides; n (%) | 1,041 (1.0%) | 212 (0.8%) | 1,089 (1.1%) | 171 (0.9%) | 3,580 (1.8%) | 247 (1.9%) | 5,710 (1.4%) | 630 (1.1%) | 0.03 |
| DM Medications - Metformin; n (%) | 74,681 (74.8%) | 20,362 (74.3%) | 79,574 (80.9%) | 14,355 (75.9%) | 142,034 (69.9%) | 9,591 (72.9%) | 296,289 (73.8%) | 44,308 (74.5%) | -0.02 |
| Concomitant initiation or current use of 2nd Generation S | 33,222 (33.3%) | 7,632 (27.9%) | 29,037 (29.5%) | 4,720 (25.0%) | 73,210 (36.0%) | 4,236 (32.2%) | 135,469 (33.7%) | 16,588 (27.9%) | 0.13 |
| Concomitant initiation or current use of AGIs; n (%) | 359 (0.4%) | 65 (0.2%) | 216 (0.2%) | 39 (0.2%) | 888 (0.4%) | 35 (0.3%) | 1,463 (0.4%) | 139 (0.2%) | 0.04 |
| Concomitant initiation or current use of Glitazones; n (%) | 6,052 (6.1%) | 1,790 (6.5%) | 5,547 (5.6%) | 1,221 (6.5%) | 11,634 (5.7%) | 990 (7.5%) | 23,233 (5.8%) | 4,001 (6.7%) | -0.04 |
| Concomitant initiation or current use of GLP-1 RA; n (%) | 2,392 (2.4%) | 4,382 (16.0%) | 2,527 (2.6%) | 3,730 (19.7%) | 2,849 (1.4%) | 1,906 (14.5%) | 7,768 (1.9%) | 10,018 (16.8%) | -0.53 |
| Concomitant initiation or current use of Insulin; n (%) | 13,381 (13.4%) | 5,986 (21.9%) | 11,021 (11.2%) | 4,466 (23.6%) | 29,957 (14.7%) | 3,603 (27.4%) | 54,359 (13.5%) | 14,055 (23.6%) | -0.26 |
| Concomitant initiation or current use of Meglitinides; n (% | 773 (0.8%) | 145 (0.5%) | 768 (0.8%) | 117 (0.6%) | 2,607 (1.3%) | 170 (1.3%) | 4,148 (1.0%) | 432 (0.7%) | 0.03 |
| Concomitant initiation or current use of Metformin; n (%) | 64,669 (64.7%) | 16,361 (60.3%) | 70,407 (71.6%) | 11,825 (62.5%) | 122,594 (60.3%) | 8,039 (61.1%) | 257,670 (64.2%) | 36,425 (61.3%) | 0.06 |
| Past use of 2nd Generation SUs Copy; n (%) | 7,266 (7.3%) | 2,028 (7.4%) | 6,956 (7.1%) | 1,253 (6.6%) | 14,813 (7.3%) | 902 (6.9%) | 29,035 (7.2%) | 4,183 (7.0%) | 0.01 |
| Past use of AGIs Copy; n (%) | 140 (0.1%) | 32 (0.1%) | 94 (0.1%) | 25 (0.1%) | 355 (0.2%) | 23 (0.2%) | 589 (0.1%) | 80 (0.1%) | 0.00 |
| Past use of Glitazones Copy; n (%) | 1,542 (1.5%) | 528 (1.9%) | 1,334 (1.4%) | 299 (1.6%) | 3,088 (1.5%) | 263 (2.0%) | 5,964 (1.5%) | 1,090 (1.8%) | -0.02 |
| Past use of GLP-1 RA Copy; n (%) | 1,977 (2.0%) | 1,701 (6.2%) | 2,007 (2.0%) | 1,253 (6.6%) | 2,441 (1.2%) | 623 (4.7%) | 6,425 (1.6%) | 3,577 (6.0%) | -0.23 |
| | | | | | | | | | -0.12 |
| Past use of Insulin Copy; n (%) | 4,434 (4.5%) | 1,852 (6.8%) | 3,797 (3.9%) | 1,401 (7.4%) | 9,160 (4.5%) | 945 (7.2%) | 17,411 (4.3%) | 4,198 (7.1%) | |
| Past use of Meglitinides Copy; n (%) | 268 (0.3%) | 67 (0.2%) | 321 (0.3%) | 54 (0.3%) | 973 (0.5%) | 77 (0.6%) | 1,562 (0.4%) | 198 (0.3%) | 0.02 |
| Past use of metformin (final) Copy; n (%) | 10,012 (10.0%) | 3,801 (13.9%) | 9,167 (9.3%) | 2,530 (13.4%) | 19,440 (9.6%) | 1,552 (11.8%) | 38,619 (9.6%) | 7,883 (13.3%) | -0.12 |
| Other Medications | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 52,616 (52.7%) | 14,800 (54.0%) | 52,849 (53.7%) | 10,492 (55.5%) | 96,076 (47.3%) | 6,205 (47.2%) | 201,541 (50.2%) | 31,497 (53.0%) | -0.06 |
| Use of ARBs; n (%) | 33,459 (33.5%) | 9,268 (33.8%) | 32,714 (33.3%) | 6,489 (34.3%) | 69,748 (34.3%) | 4,833 (36.7%) | 135,921 (33.8%) | 20,590 (34.6%) | -0.02 |
| Use of Loop Diuretics - United; n (%) | 10,502 (10.5%) | 2,316 (8.5%) | 6,912 (7.0%) | 1,075 (5.7%) | 33,131 (16.3%) | 1,744 (13.3%) | 30,343 (12.6%) | 5,135 (8.6%) | 0.13 |
| Use of other diuretics- United; n (%) | 2,623 (2.6%) | 833 (3.0%) | 2,133 (2.2%) | 453 (2.4%) | 6,785 (3.3%) | 483 (3.7%) | 11,541 (2.9%) | 1,769 (3.0%) | -0.01 |
| Use of nitrates-United; n (%) | 4,760 (4.8%) | 1,425 (5.2%) | 3,232 (3.3%) | 624 (3.3%) | 14,468 (7.1%) | 976 (7.4%) | 22,460 (5.6%) | 3,025 (5.1%) | 0.02 |
| Use of other hypertension drugs; n (%) | 6,251 (6.3%) | 1,267 (4.6%) | 4,430 (4.5%) | 643 (3.4%) | 15,746 (7.7%) | 809 (6.1%) | 26,447 (6.6%) | 2,719 (4.6%) | 0.09 |
| Use of digoxin-United; n (%) | 1,351 (1.4%) | 278 (1.0%) | 1,001 (1.0%) | 112 (0.6%) | 5,685 (2.8%) | 306 (2.3%) | 8,037 (2.0%) | 696 (1.2%) | 0.06 |
| | 1,058 (1.1%) | 283 (1.0%) | 807 (0.8%) | 143 (0.8%) | 3,770 (1.9%) | 218 (1.7%) | 5,635 (1.4%) | 644 (1.1%) | 0.03 |
| Use of Anti-errhythmics; n (%) | | , , | | , , | | | | , , | |
| Use of COPD/asthma meds- United; n (%) | 14,067 (14.1%) | 3,637 (13.3%) | 12,756 (13.0%) | 2,412 (12.8%) | 32,384 (15.9%) | 2,112 (16.1%) | 59,207 (14.7%) | 8,161 (13.7%) | 0.03 |
| Use of statins; n (%) | 71,183 (71.3%) | 20,272 (74.0%) | 65,053 (66.1%) | 13,377 (70.7%) | 148,529 (73.1%) | 10,331 (78.5%) | 284,765 (70.9%) | 43,980 (74.0%) | -0.07 |
| Use of other lipid-lowering drugs; n (%) | 11,144 (11.2%) | 3,351 (12.2%) | 12,301 (12.5%) | 2,743 (14.5%) | 24,891 (12.2%) | 1,915 (14.6%) | 48,336 (12.0%) | 8,009 (13.5%) | -0.04 |
| Use of antiplatelet agents; n (%) | 12,026 (12.0%) | 3,756 (13.7%) | 10,435 (10.6%) | 2,047 (10.8%) | 30,403 (15.0%) | 2,275 (17.3%) | 52,864 (13.2%) | 8,078 (13.6%) | -0.01 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban, Apixal | 5,155 (5.2%) | 1,283 (4.7%) | 3,619 (3.7%) | 581 (3.1%) | 17,505 (8.6%) | 1,132 (8.6%) | 26,279 (6.5%) | 2,996 (5.0%) | 0.06 |
| Use of heparin and other low-molecular weight heparins; n | 198 (0.2%) | 43 (0.2%) | 9 (0.0%) | 1 (0.0%) | 420 (0.2%) | 21 (0.2%) | 627 (0.2%) | 065 (0.1%) | 0.03 |
| Use of NSAIDs; n (%) | 16,220 (16.2%) | 4,317 (16.5%) | 16,087 (16.4%) | 3,178 (16.8%) | 32,311 (15.9%) | 1,975 (15.0%) | 64,618 (16.1%) | 9,670 (16.3%) | -0.01 |
| Use of oral corticosteroids; n (%) | 10,445 (10.5%) | 2,832 (10.3%) | 9,420 (9.6%) | 1,722 (9.1%) | 23,684 (11.7%) | 1,501 (11.4%) | 43,549 (10.8%) | 6,055 (10.2%) | 0.02 |
| Use of bisphosphonate (United); n (%) | 2,212 (2.2%) | 322 (1.2%) | 803 (0.8%) | 70 (0.4%) | 6,829 (3.4%) | 252 (1.9%) | 9,844 (2.5%) | 644 (1.1%) | 0.11 |
| Use of opioids-United; n (%) | 20,346 (20.4%) | 5,472 (20.0%) | 18,620 (18.9%) | 3,581 (18.9%) | 42,529 (20.9%) | 2,588 (19.7%) | 81,495 (20.3%) | 11,641 (19.6%) | 0.02 |
| Use of antidepressants; n (%) | 22,602 (22.6%) | 6,573 (24.0%) | 19,480 (19.8%) | 4,303 (22.8%) | 48,867 (24.0%) | 3,160 (24.0%) | 90,949 (22.6%) | 14,036 (23.6%) | -0.02 |
| Use of antipsychotics; n (%) | 2,384 (2.6%) | 556 (2.0%) | 1,381 (1.4%) | 263 (1.4%) | 6,338 (3.1%) | 258 (2.0%) | 10,303 (2.6%) | 1,077 (1.8%) | 0.05 |
| Use of anticonvulsants; n (%) | 16,330 (16.3%) | 4,552 (16.6%) | 10,690 (10.9%) | 2,193 (11.6%) | 34,272 (16.9%) | 2,157 (16.4%) | 61,292 (15.3%) | 8,902 (15.0%) | 0.01 |
| | | | | | 34,272 (10.376) | 2,137 (10.4/6) | 01,252 (13.3/6) | 0,502 (15.076) | 0.01 |
| Use of lithium-United; n (%) | 147 (0.1%) | 39 (0.1%) | 115 (0.1%) | 29 (0.2%) | | 4 222 (2 25) | an entre de afri | | |
| Use of Benzos-United; n (%) | 9,376 (9.4%) | 2,472 (9.0%) | 7,846 (8.0%) | 1,587 (8.4%) | 21,369 (10.5%) | 1,277 (9.7%) | 38,591 (9.6%) | 5,336 (9.0%) | 0.02 |
| Use of anxiolytics/hypnotics-United; n (%) | 4,899 (4.9%) | 1,421 (5.2%) | 5,117 (5.2%) | 1,058 (5.6%) | 10,049 (4.9%) | 683 (5.2%) | 20,065 (5.0%) | 3,162 (5.3%) | -0.01 |
| Use of dementia meds-United; n (%) | 2,332 (2.3%) | 208 (0.8%) | 1,003 (1.0%) | 51 (0.3%) | 10,424 (5.1%) | 272 (2.1%) | 13,759 (3.4%) | 531 (0.9%) | 0.17 |
| Use of antiparkinsonian meds- United; n (%) | 2,112 (2.1%) | 562 (2.1%) | 1,514 (1.5%) | 265 (1.4%) | 6,081 (3.0%) | 335 (2.5%) | 9,707 (2.4%) | 1,162 (2.0%) | 0.03 |
| Any use of pramtintide; n (%) | 2 (0.0%) | 9 (0.0%) | 9 (0.0%) | 23 (0.1%) | | | | | ** |
| Any use of 1st generation sulfonyluress; n (%) | 2 (0.0%) | 1 (0.0%) | 10 (0.0%) | 1 (0.0%) | | | | | ** |
| Entresto (sacubitril/valsartan); n (%) | 158 (0.2%) | 122 (0.4%) | 52 (0.1%) | 22 (0.1%) | 158 (0.1%) | 43 (0.3%) | 368 (0.1%) | 187 (0.3%) | 0.00 |
| Initiation as monotherapy v4 Copy; n (%) | 85,916 (86.0%) | 25,773 (94.1%) | 84,176 (85.6%) | 17,936 (94.8%) | 184,924 (91.0%) | 12,565 (95.5%) | 355,016 (88.4%) | 36,274 (94.6%) | -0.22 |
| Labs | | | | | ( | | 198,248 | 46,306 | |
| Lab values- HbA1c (%) v3; n (%) | 43,141 (43.2%) | 11,298 (41.2%) | 6,423 (6.5%) | 1,049 (5.5%) | N/A | N/A | 49,564 (25.0%) | 12,347 (26.7%) | -0.04 |
| Lab values- HbA1c (%) (within 3 months) v3; n (%) | 34,616 (34.6%) | 9,068 (33.1%) | 5,174 (5.3%) | 858 (4.5%) | N/A | N/A | 39,790 (20.1%) | 9,926 (21.4%) | -0.03 |
| | 21,020 (34.079) | 2,000 (23.279) | 2,2.4 (3.3%) | 536 [4.576] | II/A | Total Control | 25,150 [20.270] | 2,220 (22.470) | 0.03 |

| Lab values- HbA1c (%) (within 6 months) v3; n (%) | 43,141 (43.2%) | 11,298 (41.2%) | 6,423 (6.5%) | 1,049 (5.5%) | N/A | N/A | 49,564 (25.0%) | 12,347 (26.7%) | -0.04 |
|---|---|---|---|---|---|---|---|---|---|
| Lab values- BNP; n (%) | 749 (0.7%) | 156 (0.6%) | 74 (0.1%) | 5 (0.0%) | N/A | N/A | 823 (0.4%) | 161 (0.3%) | 0.02 |
| | | | | | N/A | N/A | | | 0.02 |
| Lab values- BNP (within 3 months); n (%) | 463 (0.5%) | 98 (0.4%) | 53 (0.1%) | 1 (0.0%) | | | 516 (0.3%) | 099 (0.2%) | |
| Lab values- BNP (within 6 months); n (%) | 749 (0.7%) | 156 (0.6%) | 74 (0.1%) | 5 (0.0%) | N/A | N/A | 823 (0.4%) | 161 (0.3%) | 0.02 |
| Lab values- BUN (mg/di); n (%) | 42,226 (42.3%) | 10,947 (40.0%) | 6,201 (6.3%) | 967 (5.1%) | N/A | N/A | 48,427 (24.4%) | 11,914 (25.7%) | -0.03 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 33,174 (33.2%) | 8,603 (31.4%) | 4,838 (4.9%) | 783 (4.1%) | N/A | N/A | 38,012 (19.2%) | 9,386 (20.3%) | -0.03 |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 42,226 (42.3%) | 10,947 (40.0%) | 6,201 (6.3%) | 967 (5.1%) | N/A | N/A | 48,427 (24.4%) | 11,914 (25.7%) | -0.03 |
| Lab values- Creatinine (mg/dl) v2; n (%) | 43,684 (43.7%) | 11,561 (42.2%) | 6,653 (6.8%) | 1,095 (5.8%) | N/A | N/A | 50,337 (25.4%) | 12,656 (27.3%) | -0.04 |
| cab values ci dacinine (ing/ui) vz, ii (xi) | 43,004 (43.776) | 11,361 (42.276) | 0,033 (0.8/9) | 1,050 (5.6.4) | N/A | IV. | 30,337 (23.4/6) | 12,030 (27.376) | 0.04 |
| Lab values- Creatinine (mg/dl) (within 3 months) v2; n (%) | 34,353 (34.4%) | 9,066 (33.1%) | 5,215 (5.3%) | 882 (4.7%) | N/A | N/A | 39,568 (20.0%) | 9,948 (21.5%) | -0.04 |
| cab values a cacinine (ingrai) (waliin s monais) vz., n (x) | 34,333 (34.4/8) | 3,000 (33.1/0) | اورو دا درود | 002 (4.770) | nya. | IVA | 33,366 (20.0/9) | 3,340 [21.3/9] | 0.04 |
| to the second se | 42 424 (42 28) | 44 864 (45 881) | a con la obil | 4 000 (0 00) | | *** | | 42 525 (22.25) | |
| Lab values- Creatinine (mg/dl) (within 6 months) v2; n (%) | 43,684 (43.7%) | 11,561 (42.2%) | 6,653 (6.8%) | 1,095 (5.8%) | N/A | N/A | 50,337 (25.4%) | 12,656 (27.3%) | -0.04 |
| Lab values- HDL level (mg/dl); n (%) | 36,599 (36.6%) | 9,688 (35.4%) | 5,867 (6.0%) | 1,004 (5.3%) | N/A | N/A | 42,466 (21.4%) | 10,692 (23.1%) | -0.04 |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 27,311 (27.3%) | 7,215 (26.3%) | 4,458 (4.5%) | 768 (4.1%) | N/A | N/A | 31,769 (16.0%) | 7,983 (17.2%) | -0.03 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 36,599 (36.6%) | 9,688 (35.4%) | 5,867 (6.0%) | 1,004 (5.3%) | N/A | N/A | 42,466 (21.4%) | 10,692 (23.1%) | -0.04 |
| Lab values-LDL level (mg/dl) v2; n (%) | 37,864 (37.9%) | 10,005 (36.5%) | 6,037 (6.1%) | 991 (5.2%) | N/A | N/A | 43,901 (22.1%) | 10,996 (23.7%) | -0.04 |
| 107-17 | | | | | | | | | |
| Lab values- LDL level (mg/dl) (within 3 months) v2; n (%) | 28,216 (28.2%) | 7,452 (27.2%) | 4,563 (4.6%) | 765 (4.0%) | N/A | N/A | 32,779 (16.5%) | 8,217 (17.7%) | -0.03 |
| | ,, | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | 3,555 (3,554) | | | | | -, () | |
| Lab values-LDL level (mg/dl) (within 6 months) v2; n (%) | 37,864 (37.9%) | 10,005 (36.5%) | 6,037 (6.1%) | 991 (5.2%) | N/A | N/A | 43,901 (22.1%) | 10,996 (23.7%) | -0.04 |
| | | | | | N/A | | | | 0.00 |
| Lab values- NT-proBNP; n (%) | 114 (0.1%) | 43 (0.2%) | 17 (0.0%) | 2 (0.0%) | | N/A | 131 (0.1%) | 45 (0.1%) | 0.00 |
| Lab values- NT-proBNP (within 3 months); n (%) | 66 (0.1%) | 27 (0.1%) | 12 (0.0%) | 2 (0.0%) | N/A | N/A | 78 (0.0%) | 29 (0.1%) | - |
| Lab values- NT-proBNP (within 6 months); n (%) | 114 (0.1%) | 43 (0.2%) | 17 (0.0%) | 2 (0.0%) | N/A | N/A | 131 (0.1%) | 45 (0.1%) | - |
| Lab values-Total cholesterol (mg/dl) v2; n (%) | 37,177 (37.2%) | 9,915 (36.2%) | 5,903 (6.0%) | 1,018 (5.4%) | N/A | N/A | 43,080 (21.7%) | 10,933 (23.6%) | -0.05 |
| (0) | | | | | | | | | |
| Lab values-Total cholesterol (mg/dl) (within 3 months) v2; | 27,768 (27.8%) | 7,384 (27.0%) | 4,489 (4.6%) | 783 (4.1%) | N/A | N/A | 32,257 (16.3%) | 8,167 (17.6%) | -0.03 |
| and the state of t | 27,700 (27.0.4) | ,,201,21101 | 4,100 [1.0.4] | 100 (1.004) | - | 141 | 32,237 (20.374) | 0,207 (27.074) | |
| Lab values-Total cholesterol (mg/dl) (within 6 months) v2; | 37,177 (37.2%) | 9,915 (36.2%) | 5,903 (6.0%) | 1,018 (5.4%) | N/A | N/A | 43,080 (21.7%) | 10,933 (23.6%) | -0.05 |
| | | | | | | - | | | -0.05 |
| Lab values-Triglyceride level (mg/dl); n (%) | 36,829 (36.9%) | 9,848 (35.9%) | 5,814 (5.9%) | 1,000 (5.3%) | N/A | N/A | 42,643 (21.5%) | 10,848 (23.4%) | -0.05 |
| Lab values-Triglyceride level (mg/dl) (within 3 months); n (: | 27,527 (27.6%) | 7,338 (26.8%) | 4,418 (4.5%) | 771 (4.1%) | N/A | N/A | 31,945 (16.1%) | 8,109 (17.5%) | -0.04 |
| Lab values-Triglyceride level (mg/dl) (within 6 months); n (: | 36,829 (36.9%) | 9,848 (35.9%) | 5,814 (5.9%) | 1,000 (5.3%) | N/A | N/A | 42,643 (21.5%) | 10,848 (23.4%) | -0.05 |
| Lab result number- HbA1c (%) mean (only 2 to 20 included) | 42,905 | 11,242 | 6,311 | 1,018 | N/A | N/A | 49,216 | 12,260 | |
| mean (sd) | 8.36 (1.78) | 8.55 (1.75) | 8.53 (1.88) | 8.32 (1.79) | N/A | N/A | 8.38 (1.79) | 8.53(1.75) | -0.08 |
| median (IQR) | 8.00 [7.15, 9.25] | 8.20 [7.30, 9.55] | 8.05 [7.15, 9.50] | 8.00 [7.00, 9.00] | N/A | N/A | 8.01 (1.79) | 8.18(1.75) | -0.10 |
| | | | | | N/A | N/A | | | 0.10 |
| Missing n (%) | 56,998 (57.1%) | 16,152 (59.0%) | 92,034 (93.6%) | 17,894 (94.6%) | | | 149,032 (75.2%) | 34,046 (73.5%) | 0.04 |
| Lab result number- BNP mean v2 | 749 | 156 | 74 | 3 | N/A | N/A | 823 | 161 | |
| mean (sd) | 154.93 (290.29) | 146.64 (514.40) | 3,931.76 (32,532.43) | 32.60 (34.74) | N/A | N/A | 494.52 (9710.65) | 143.10 (509.52) | 0.05 |
| median [IQR] | 65.20 [25.55, 167.50] | 34.45 [14.55, 89.70] | 76.50 [29.75, 193.00] | 18.00 [13.50, 59.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 99,154 (99.3%) | 27,238 (99.4%) | 98,271 (99.9%) | 18,907 (100.0%) | N/A | N/A | 197,425 (99.6%) | 46,145 (99.7%) | -0.02 |
| Lab result number- BUN (mg/di) mean v2 | 42,226 | 10.947 | 6.201 | 967 | N/A | N/A | 48.427 | 11 914 | |
| meen (sd) | 17.98 (7.45) | 16.64 (5.62) | 1,795.05 (17,168.60) | 2,184.17 (18,571.33) | N/A | N/A | 245.53 (6143.29) | 192.57 (5288.81) | 0.01 |
| | 16.50 [13.00, 21.00] | 16.00 [13.00, 19.50] | 16.00 [13.00, 20.00] | 15.50 [13.00, 19.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| median [IQR] | | | | | | | | | #VALUE: |
| Missing n (%) | 57,677 (57.7%) | 16,447 (60.0%) | 92,144 (93.7%) | 17,945 (94.9%) | N/A | N/A | 149,821 (75.6%) | 34,392 (74.3%) | 0.03 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 to 15 | 43,333 | 11,484 | 5,645 | 711 | N/A | N/A | 48,978 | 12,195 | |
| mean (sd) | 1.01 (0.39) | 0.92 (0.24) | 0.98 (0.33) | 0.94 (0.20) | N/A | N/A | 1.01 (0.38) | 0.92 (0.24) | 0.28 |
| median [IQR] | 0.93 [0.78, 1.15] | 0.89 [0.75, 1.05] | 0.95 [0.79, 1.08] | 0.95 [0.81, 1.00] | N/A | N/A | 0.93 (0.38) | 0.89 (0.24) | 0.13 |
| Missing; n (%) | 56,570 (56.6%) | 15,910 (58.1%) | 92,700 (94.3%) | 18,201 (96.2%) | N/A | N/A | 149,270 (75.3%) | 34,111 (73.7%) | 0.04 |
| <del></del> | | ,,, | | | - | | | | |
| Lab result number- HDL level (mg/dl) mean (only =5000 in | 36,599 | 9.688 | 5,805 | 994 | N/A | N/A | 42.404 | 10,682 | |
| | 45.86 (13.58) | 44.26 (12.89) | 44.94 (13.83) | 47.81 (132.54) | N/A | N/A | 45.73 (13.61) | 44.59 (42.24) | 0.04 |
| mean (sd) | , , | , , | , , | , , | | | , , | , , | |
| median [IQR] | 44.00 [37.00, 53.00] | 42.00 [36.00, 51.00] | 43.00 [36.00, 52.00] | 42.00 [35.00, 50.00] | N/A | N/A | 43.86 (13.61) | 42.00 (42.24) | 0.06 |
| Missing: n (%) | 63,304 (63.4%) | 17,706 (64.6%) | 92,540 (94.1%) | 17,918 (94.7%) | N/A | N/A | 155,844 (78.6%) | 35,624 (76.9%) | 0.04 |
| Lab result number-LDL level (mg/dl) mean (only =:5000 in | 36,994 | 9,856 | 5,343 | 919 | N/A | N/A | 42,337 | 10,775 | |
| mean (sd) | 85.89 (39.91) | 81.77 (40.57) | 90.89 (42.17) | 84.41 (40.86) | N/A | N/A | 86.52 (40.20) | 82.00 (40.60) | 0.11 |
| median (IQR) | 83.50 [62.00, 108.75] | 80.50 [58.00, 105.00] | 89.00 [67.00, 116.00] | 84.00 [61.00, 109.00] | N/A | N/A | 84.19 (40.20) | 80.80 (40.60) | 0.08 |
| Missing: n (%) | 62,909 (63.0%) | 17,538 (64.0%) | 93,002 (94.6%) | 17,993 (95.1%) | N/A | N/A | 155,911 (78.6%) | 35,531 (76.7%) | 0.05 |
| | UZ,303 (03.076) | 27,330 04,070 | 23,002 (34.0/0) | 27,333 [33.170] | N/A | N/A | 222,311 (70.0/6) | 22,331 [10.770] | 0.03 |
| International Principles of the International Control of the International | | | | | and a | *** | 42 982 | | |
| Lab result number-Total cholesterol (mg/dl) mean (only =< | 37,141 | 9,912 | 5,841 | 1,005 | N/A | N/A | | 10,917 | |
| mean (sd) | 173.84 (47.32) | 170.49 (47.05) | 179.36 (49.26) | 171.92 (49.48) | N/A | N/A | 174.59 (47.59) | 170.62 (47.28) | 0.08 |
| median (IQR) | 167.50 [143.00, 198.00] | 165.00 [139.00, 195.00] | 174.00 [148.00, 205.00] | 165.50 [140.25, 196.00] | N/A | N/A | 168.38 (47.59) | 165.05 (47.28) | 0.07 |
| Missing; n (%) | 62,762 (62.8%) | 17,482 (63.8%) | 92,504 (94.1%) | 17,907 (94.7%) | N/A | N/A | 155,266 (78.3%) | 35,389 (76.4%) | 0.05 |

| Lab result number-Triglyceride level (mg/dl) mean (only=c | | 9,846 | 5,753 | 987 | N/A | N/A | 42,578 | 10,833 | |
|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 193.49 (177.23) | 207.63 (200.82) | 197.08 (184.91) | 210.43 (212.46) | N/A | N/A | 193.98 (178.29) | 207.89 (201.92) | -0.07 |
| median (IQR) | 155.00 [110.00, 223.00] | 160.00 [113.00, 236.00] | 153.00 [106.50, 228.25] | 157.50 [109.00, 233.00] | N/A | N/A | 154.73 (178.29) | 159.77 (201.92) | -0.03 |
| Missing: n (%) | 63,078 (63.1%) | 17,548 (64.1%) | 92,592 (94.2%) | 17,925 (94.8%) | N/A | N/A | 155,670 (78.5%) | 35,473 (76.6%) | 0.05 |
| Lab result number- Hemoglobin mean (only >0 included) | 28,791 | 7,333 | 4,328 | 643 | N/A | N/A | 33,119 | 7,976 | |
| mean (sd) | 13.72 (1.56) | 14.15 (1.49) | 6,342.54 (215,464.58) | 1,919.68 (16,045.24) | N/A | N/A | 840.77 (77884.39) | 167.77 (4553.05) | 0.01 |
| median [IQR] | 13.70 [12.65, 14.80] | 14.10 [13.10, 15.20] | 13.90 [12.85, 15.00] | 14.00 [13.00, 15.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 71,112 (71.2%) | 20,061 (73.2%) | 94,017 (95.6%) | 18,269 (96.6%) | N/A | N/A | 165,129 (83.3%) | 38,330 (82.8%) | 0.01 |
| Lab result number- Serum sodium mean (only > 90 and < 15 | 42,353 | 11,249 | 6,243 | 1,027 | N/A | N/A | 48,596 | 12,276 | |
| mean (sd) | 139.42 (2.77) | 139.45 (2.68) | 138.82 (2.61) | 139.17 (2.53) | N/A | N/A | 139.34 (2.75) | 139.43 (2.67) | -0.03 |
| median [IQR] | 139.50 [138.00, 141.00] | 139.50 [138.00, 141.00] | 139.00 [137.00, 140.50] | 139.00 [137.50, 141.00] | N/A | N/A | 139.44 (2.75) | 139.46 (2.67) | -0.01 |
| Missing; n (%) | 57,550 (57.6%) | 16,145 (58.9%) | 92,102 (93.7%) | 17,885 (94.6%) | N/A | N/A | 149,652 (75.5%) | 34,030 (73.5%) | 0.05 |
| • 17 | | | | | | | | | |
| Lab result number- Albumin mean (only >0 and <=10 includes | 39,793 | 10,600 | 5,330 | 848 | N/A | N/A | 45,123 | 11,448 | |
| mean (sd) | 4.29 (0.32) | 4.32 (0.31) | 4.20 (0.38) | 4.10 (0.39) | N/A | N/A | 4.28 (0.33) | 4.30 (0.32) | -0.06 |
| median [IQR] | 4.30 [4.10, 4.50] | 4.30 [4.10, 4.50] | 4.20 [4.00, 4.45] | 4.00 [4.00, 4.30] | N/A | N/A | 4.29 (0.33) | 4.28 (0.32) | 0.03 |
| Missing, n (%) | 60,110 (60.2%) | 16,794 (61.3%) | 93,015 (94.6%) | 18,064 (95.5%) | N/A | N/A | 153,125 (77.2%) | 34,858 (75.3%) | 0.04 |
| | ,, | | ,() | ,, | | | ,() | ,, | |
| Lab result number- Glucose (fasting or random) mean (only | 42,469 | 11,283 | 6,343 | 1,054 | N/A | N/A | 48.812 | 12,337 | |
| mean (sd) | 178.34 (72.25) | 182.55 (71.67) | 181.56 (74.01) | 177.65 (69.16) | N/A | N/A | 178.76 (72.48) | 182.13 (71.46) | -0.05 |
| median (IQR) | 161.00 [129.00, 209.50] | 167.00 [132.50, 217.00] | 163.00 [130.50, 215.50] | 161.75 [129.00, 209.00] | N/A | N/A | 161.26 (72.48) | 166.55 (71.46) | -0.07 |
| Missing n (%) | 57,434 (57.5%) | 16,111 (58.8%) | 92,002 (93.6%) | 17,858 (94.4%) | N/A | N/A | 149,436 (75.4%) | 33,969 (73.4%) | 0.05 |
| wessing, re(re) | 37,434 [37.37] | 10,111 (30.0/6) | 32,002 (33.0/0) | 17,030 [34.4/9] | nya. | N/A | 143,430 [73,476] | 33,363 [/3.4/6] | 0.03 |
| Lab result number- Potassium mean (only 1-7 included) | 43,384 | 11,485 | 6,118 | 973 | N/A | N/A | 49,502 | 12,458 | |
| mean (sd) | 4.48 (0.43) | 4.47 (0.40) | 4.32 (0.46) | 4.16 (0.50) | N/A | N/A | 4.46 (0.43) | 4.45 (0.41) | 0.02 |
| | | | , , | | N/A | N/A | , , | · · | 0.17 |
| median [IQR] | 4.50 [4.20, 4.70] | 4.45 [4.20, 4.70] | 4.30 [4.00, 4.60] | 4.00 [4.00, 4.50] | | | 4.48 (0.43) | 4.41 (0.41) | |
| Missing n (%) | 56,519 (56.6%) | 15,909 (58.1%) | 92,227 (93.8%) | 17,939 (94.9%) | N/A | N/A | 148,746 (75.0%) | 33,848 (73.1%) | 0.04 |
| Comorbidity Scores | | | | | | | | | |
| CCI (180 days)-ICD9 and ICD10 v2 | | | | | | | | | |
| mean (sd) | 2.43 (1.80) | 2.25 (1.47) | 1.64 (1.30) | 1.67 (1.06) | 2.63 (1.89) | 2.46 (1.56) | 2.34 (1.74) | 2.11(1.38) | 0.15 |
| median [IQR] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 1.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 2.00 [1.00, 4.00] | 2.00 [1.00, 3.00] | 1.76 (1.74) | 2.00 (1.38) | -0.15 |
| Frailty Score: Qualitative Version 365 days as Categories, v1 | | | | | | | | | |
| 0; n (%) | 68,126 (68.2%) | 23,602 (86.2%) | 60,170 (61.2%) | 14,653 (77.5%) | 92,074 (45.3%) | 10,006 (76.1%) | 220,370 (54.9%) | 48,261 (81.2%) | -0.59 |
| 1 to 2; n (%) | 24,208 (24.2%) | 3,375 (12.3%) | 29,743 (30.2%) | 3,605 (19.1%) | 66,971 (32.9%) | 2,319 (17.6%) | 120,922 (30.1%) | 9,299 (15.6%) | 0.35 |
| 3 or more; n (%) | 7,569 (7.6%) | 417 (1.5%) | 8,432 (8.6%) | 654 (3.5%) | 44,249 (21.8%) | 831 (6.3%) | 60,250 (15.0%) | 1,902 (3.2%) | 0.42 |
| Frailty Score: Empirical Version 365 days as Categories, v3 | | | | | | | | | |
| <0.12908; n (%) | 28,978 (29.0%) | 9,111 (33.3%) | 32,840 (33.4%) | 6,951 (36.8%) | 26,735 (13.2%) | 2,162 (16.4%) | 88,553 (22.1%) | 18,224 (30.6%) | -0.19 |
| 0.12908 -0.1631167; n (%) | 33,399 (33.4%) | 9,641 (35.2%) | 36,156 (36.8%) | 7,300 (38.6%) | 55,651 (27.4%) | 4,179 (31.8%) | 125,206 (31.2%) | 21,120 (35.5%) | -0.09 |
| >=0.1631167; n (%) | 37,526 (37.6%) | 8,642 (31.5%) | 29,349 (29.8%) | 4,661 (24.6%) | 120,908 (59.5%) | 6,815 (51.8%) | 187,783 (46.8%) | 20,118 (33.8%) | 0.27 |
| Non-Frailty; n (%) | 57,586 (57.6%) | 16,315 (59.6%) | 50,767 (51.6%) | 10,157 (53.7%) | 10,528 (5.2%) | 611 (4.6%) | 118,881 (29.6%) | 27,083 (45.5%) | -0.33 |
| PVI | | | | | | . , | - 1 | | |
| Frailty Score (mean): Qualitative Version 365 days, v1 | | | | | | | | | |
| mean (sd) | 0.64 (1.29) | 0.21 (0.64) | 0.75 (1.28) | 0.37 (0.86) | 1.43 (1.93) | 0.48 (1.11) | 1.07 (1.64) | 0.32 (0.83) | 0.58 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 (0.00, 0.00) | 1.00 (0.00, 2.00) | 0.00 [0.00, 0.00] | 0.51 (1.64) | 0.00 (0.83) | 0.39 |
| Frailty Score (mean): Empirical Version 365 days, v2 | | | | | | | 1 | | |
| mean (sd) | 0.16 (0.05) | 0.15 (0.04) | 0.15 (0.04) | 0.14 (0.03) | 0.19 (0.06) | 0.17 (0.05) | 0.17 (0.05) | 0.15 (0.04) | 0.44 |
| median (IQR) | 0.15 [0.13, 0.18] | 0.14[0.12, 0.17] | 0.14 [0.12, 0.16] | 0.13 [0.12, 0.16] | | 0.17 [0.14, 0.20] | 0.16 (0.05) | 0.14 (0.04) | 0.44 |
| Healthcare Utilization | 0.13 (0.13, 0.10) | 0.27 [0.22, 0.27] | 0.21 (0.22, 0.20) | 0.13 [0.11, 0.10] | 0.27 (0.24, 0.22) | 0.27 [0.24, 0.25] | 0.20 (0.00) | 5.27(5.54) | |
| | 5.407/5.5%) | 1,088 (4.0%) | 2 250 /2 454 | 447 /2 294) | 12 442 (6 194) | AD2 (2 7%) | 24 207 (5 2%) | 4 007 (2 291) | 0.10 |
| Any hospitalization; n (%) | 5,497 (5.5%) | - 1 | 3,358 (3.4%) | 417 (2.2%) | 12,442 (6.1%) | 482 (3.7%) | 21,297 (5.3%) | 1,987 (3.3%) | 0.10 |
| Any hospitalization within prior 30 days; n (%) | 1,947 (1.9%) | 275 (1.0%) | 982 (1.0%) | 61 (0.3%) | 3,634 (1.8%) | 65 (0.5%) | 6,563 (1.6%) | 401 (0.7%) | |
| Any hospitalization during prior 31-180 days; n (%) | 3,821 (3.8%) | 845 (3.1%) | 2,452 (2.5%) | 362 (1.9%) | 9,387 (4.6%) | 424 (3.2%) | 15,660 (3.9%) | 1,631 (2.7%) | 0.07 |
| Endocrinologist Visit; n (%) | 9,696 (9.7%) | 6,083 (22.2%) | 8,916 (9.1%) | 4,696 (24.8%) | 24,295 (12.0%) | 3,503 (26.6%) | 42,907 (10.7%) | 14,282 (24.0%) | -0.36 |
| Endocrinologist Visit (30 days prior); n (%) | 6,358 (6.4%) | 4,656 (17.0%) | 5,990 (6.1%) | 3,590 (19.0%) | 15,500 (7.6%) | 2,720 (20.7%) | 27,848 (6.9%) | 10,966 (18.4%) | -0.35 |
| Endocrinologist Visit (31 to 180 days prior); n (%) | 6,361 (6.6%) | 4,086 (14.9%) | 5,999 (6.1%) | 3,222 (17.0%) | 17,451 (8.6%) | 2,594 (19.7%) | 30,011 (7.5%) | 9,902 (16.7%) | -0.28 |
| Internal medicine/family medicine visits; n (%) | 79,699 (79.8%) | 19,568 (71.4%) | 85,692 (87.1%) | 15,991 (84.6%) | 164,752 (81.0%) | 10,436 (79.3%) | 330,143 (82.2%) | 45,995 (77.4%) | 0.12 |
| Internal medicine/family medicine visits (30 days prior) v2; | 59,806 (59.9%) | 14,110 (51.5%) | 64,158 (65.2%) | 11,352 (60.0%) | 116,541 (57.3%) | 7,146 (54.3%) | 240,505 (59.9%) | 32,608 (54.8%) | 0.10 |
| Internal medicine/family medicine visits (31 to 180 days pr | | 16,887 (61.6%) | 69,171 (70.3%) | 13,393 (70.8%) | 142,940 (70.3%) | 9,188 (69.8%) | 280,621 (69.9%) | 39,468 (66.4%) | 0.08 |
| Cardiologist visit; n (%) | 23,368 (23.4%) | 6,777 (24.7%) | 14,980 (15.2%) | 3,006 (15.9%) | 60,430 (29.7%) | 4,227 (32.1%) | 98,778 (24.6%) | 14,010 (23.6%) | 0.02 |
| Number of Cardiologist visits (30 days prior); n (%) | 8,018 (8.0%) | 2,440 (8.9%) | 4,841 (4.9%) | 894 (4.7%) | 19,046 (9.4%) | 1,399 (10.6%) | 31,905 (7.9%) | 4,733 (8.0%) | 0.00 |

| Number of Cardiologist visits (31 to 180 days prior); n (%) | 19,586 (19.6%) | 5,663 (20.7%) | 12,542 (12.8%) | 2,550 (13.5%) | 52,580 (25.9%) | 3,650 (27.7%) | 84,708 (21.1%) | 11,863 (20.0%) | 0.03 |
|---|---|---|---|---|---|---|---|---|---|
| Bectrocardiogram v2; n (%) | 26,602 (26.6%) | 7,163 (26.1%) | 22,603 (23.0%) | 4,033 (21.3%) | 61,061 (30.0%) | 4,106 (31.2%) | 110,266 (27.5%) | 15,302 (25.7%) | 0.04 |
| Use of glucose test strips; n (%) | 3,648 (3.7%) | 852 (3.1%) | 3,332 (3.4%) | 754 (4.0%) | 6,468 (3.2%) | 414 (3.1%) | 13,448 (3.3%) | 2,020 (3.4%) | -0.01 |
| Dialysis; n (%) | 26 (0.0%) | 1 (0.0%) | 10 (0.0%) | 0 (0.0%) | 24,032 (11.8%) | 647 (4.9%) | 50,834 (12.7%) | 3,630 (6.1%) | 0.23 |
| Naive new user v8 Copy; n (%)<br>Nantidiabetic drugs at index date v3 Copy | 13,650 (13.7%) | 1,877 (6.9%) | 13,152 (13.4%) | 1,106 (5.8%) | 24,032 (11.8%) | 647 [4.976] | 30,834 (12.7%) | 3,630 (6.176) | 0.23 |
| mean (sd) | 2.26 (0.83) | 2.34 (0.93) | 2.28 (0.82) | 2.39 (0.96) | 2.23 (0.83) | 2.44 (0.93) | 2.25 (0.83) | 2.38 (0.94) | -0.15 |
| median [IQR] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | | 2.00 [2.00, 3.00] | 2.00 (0.83) | 2.00 (0.94) | 0.00 |
| | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.50 [2.50, 5.50] | 2.50 (2.50, 3.50) | 2.00 (2.00, 3.00) | 2.00 [2.00, 3.00] | 2.50 (0.55) | 200 (0.54) | 0.00 |
| number of different/distinct medication prescriptions | | | | | | | | | |
| mean (sd) | 9.99 (4.61) | 10.50 (4.73) | 8.93 (4.09) | 9.97 (4.24) | 9.91 (4.25) | 10.60 (4.22) | 9.69 (4.30) | 10.35 (4.47) | -0.15 |
| median (IQR) | 9.00 [7.00, 12.00] | 10.00 [7.00, 13.00] | 8.00 [6.00, 11.00] | 9.00 [7.00, 12.00] | 9.00 [7.00, 12.00] | 10.00 [8.00, 13.00] | 8.76 (4.30) | 9.68 (4.47) | -0.21 |
| Number of Hospitalizations | | | | | | | | | |
| mean (sd) | 0.07 (0.30) | 0.05 (0.24) | 0.04 (0.21) | 0.02 (0.16) | 0.07 (0.32) | 0.04 (0.23) | 0.06 (0.29) | 0.04 (0.22) | 0.08 |
| median (IQR) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.29) | 0.00 (0.22) | 0.00 |
| Number of hospital days | | | | | | | | | |
| mean (sd) | 0.37 (2.52) | 0.21 (1.44) | 0.19 (1.51) | 0.10 (0.90) | 0.45 (2.78) | 0.19 (1.28) | 0.37 (2.46) | 0.17 (1.26) | 0.10 |
| median (IQR) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (2.46) | 0.00 (1.26) | 0.00 |
| Number of Emergency Department (ED) visits v3<br>mean (sd) | 0.38 (1.19) | 0.30 (1.09) | 0.07 (0.75) | 0.05 (0.57) | 0.43(1.21) | 0.30 (0.93) | 0.33 (1.11) | 0.22 (0.92) | 0.11 |
| median [IOR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | | 0.00 (1.11) | 0.00 (0.92) | 0.00 |
| median purp<br>Number of Office visits | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00[1.11] | 0.00 (0.92) | 0.00 |
| mean (sd) | 4.40 (3.47) | 4.68 (3.48) | 3.93 (3.12) | 4.16(3.11) | 4.87 (3.70) | 5.39 (3.66) | 4.52 (3.51) | 4.67 (3.41) | -0.04 |
| median [IQR] | 4.00 [2.00, 6.00] | 4.00 [2.00, 6.00] | 3.00 [2.00, 5.00] | 3.00 [2.00, 5.00] | | 5.00 [3.00, 7.00] | 3.76 (3.51) | 3.90 (3.41) | -0.04 |
| Number of Endocrinologist visits | | | | | | | | ( | |
| mean (sd) | 0.44 (2.07) | 1.13 (3.39) | 0.41 (2.05) | 1.25 (3.46) | 0.63 (2.84) | 1.59 (4.88) | 0.53 (2.49) | 1.27 (3.79) | -0.23 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 (2.49) | 0.00 (3.79) | 0.00 |
| Number of internal medicine/family medicine visits | | | | | | | | | |
| mean (sd) | 8.66 (12.52) | 7.06 (10.58) | 6.43 (7.97) | 6.12 (7.44) | 6.99 (9.20) | 6.58 (8.74) | 7.27 (9.87) | 6.65 (9.28) | 0.06 |
| median [IQR] | 5.00 [1.00, 11.00] | 4.00 [0.00, 9.00] | 4.00 [2.00, 8.00] | 4.00 [2.00, 8.00] | 4.00 [1.00, 9.00] | 4.00 [1.00, 9.00] | 4.25 (9.87) | 4.00 (9.28) | 0.03 |
| Number of Cardiologist visits | | | | | | | | | |
| mean (sd) | 1.05 (3.12) | 1.18 (3.46) | 0.59 (2.18) | 0.60 (2.16) | 1.39 (3.76) | 1.50 (3.89) | 1.11 (3.28) | 1.07 (3.22) | 0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (3.28) | 0.00 (3.22) | 0.00 |
| Number electrocardiograms received v2 | 0.49 (1.20) | 0.47 (1.16) | 0.37 (0.88) | 0.33 (0.83) | 0.56(1.18) | 0.55 (1.12) | 0.50 (1.12) | 0.44(1.06) | 0.06 |
| mean (sd)<br>median (IOR) | 0.49 (1.20) | 0.47 (1.16) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | | 0.00 (1.12) | 0.00 (1.06) | 0.00 |
| Number of HbA1c tests ordered | 0.00 (0.00, 2.00) | 0.00 [0.00, 2.00] | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 [0.00, 1.00] | 0.00 (0.00, 2.00) | 0.00 (2.22) | 0.00(2.00) | 0.00 |
| mean (sd) | 1.29 (0.88) | 1.37 (0.88) | 1.09 (0.85) | 1.33 (0.82) | 1.41 (0.85) | 1.57 (0.81) | 1.30 (0.86) | 1.40 (0.85) | -0.12 |
| median (IQR) | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 [1.00, 2.00] | | 2.00 [1.00, 2.00] | 1.00 (0.86) | 1.22 (0.85) | -0.26 |
| Number of glucose tests ordered | | | | | | | | | |
| mean (sd) | 0.55 (3.54) | 0.46 (1.58) | 0.34 (1.10) | 0.43 (1.22) | 0.42 (1.02) | 0.48 (1.08) | 0.43 (1.99) | 0.45 (1.37) | -0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 (1.99) | 0.00 (1.37) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | |
| meen (sd) | 0.97 (0.91) | 1.01 (0.94) | 0.89 (1.17) | 1.05 (1.16) | 0.98 (0.81) | 1.07 (0.83) | 0.96 (0.93) | 1.04 (0.99) | -0.08 |
| median [IQR] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 1.00 [1.00, 2.00] | 1.00 (0.93) | 1.00 (0.99) | 0.00 |
| Number of creatinine tests ordered | | | () | | | | | | |
| mean (sd)<br>median (IOR) | 0.04 (0.26)<br>0.00 (0.00, 0.00) | 0.04 (0.25)<br>0.00 [0.00, 0.00] | 0.03 (0.23)<br>0.00 (0.00, 0.00) | 0.04 (0.25)<br>0.00 (0.00, 0.00) | 0.06 (0.32)<br>0.00 (0.00, 0.00) | 0.07 (0.34)<br>0.00 [0.00, 0.00] | 0.05 (0.29) | 0.05 (0.27) | 0.00 |
| Number of BUN tests ordered | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.29) | 0.00 (0.27) | 0.00 |
| mean (sd) | 0.02 (0.20) | 0.02 (0.17) | 0.02 (0.18) | 0.02 (0.17) | 0.04 (0.26) | 0.04 (0.26) | 0.03 (0.23) | 0.02 (0.19) | 0.05 |
| median (IQR) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | | 0.00 [0.00, 0.00] | 0.00 (0.23) | 0.00 (0.19) | 0.00 |
| Number of tests for microal burninuria | | | | | | | | | |
| mean (sd) | 0.81 (1.17) | 0.87 (1.18) | 0.64 (1.03) | 0.81(1.12) | 0.48 (0.70) | 0.56 (0.71) | 0.60 (0.92) | 0.78 (1.07) | -0.18 |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (0.92) | 0.00 (1.07) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd digit level Co | | | | | _ | _ | | _ | |
| mean (sd) | 6.92 (7.38) | 8.25 (6.87) | 2.91 (3.94) | 3.91 (3.75) | 6.39 (7.39) | 8.79 (7.04) | 5.67 (6.71) | 6.99 (6.10) | -0.21 |
| median [IQR] | 5.00 [0.00, 10.00] | 7.00 [4.00, 11.00] | 2.00 [0.00, 5.00] | 4.00 [0.00, 6.00] | 5.00 [0.00, 10.00] | 7.00 [4.00, 12.00] | 4.27 (6.71) | 6.05 (6.10) | -0.28 |
| Use of thiazide; n (%) | 11,963 (12.0%) | 3,080 (11.2%) | 10,371 (10.5%) | 1,926 (10.2%) | 27,843 (13.7%) | 1,804 (13.7%) | 50,177 (12.5%) | 6,810 (11.5%) | 0.03 |
| Use of beta blockers; n (%) | 36,576 (36.6%) | 9,851 (36.0%) | 30,224 (30.7%) | 3,661 (29.9%) | 96,233 (47.3%) | 6,419 (48.8%) | 163,033 (40.6%) | 21,931 (36.9%) | 0.03 |
| Use of calcium channel blockers; n (%) | 30,078 (30.1%) | 7,288 (26.6%) | 26,215 (26.7%) | 4,370 (23.1%) | 69,690 (34.3%) | 4,001 (30.4%) | 125,983 (31.4%) | 15,659 (26.3%) | 0.11 |